CLINICAL TRIAL: NCT01942668
Title: A Phase 3 Study Safety and Efficacy Study of the Combination Estradiol and Progesterone to Treat Vasomotor Symptoms in Postmenopausal Women With an Intact Uterus
Brief Title: A Safety and Efficacy Study of the Combination Estradiol and Progesterone to Treat Vasomotor Symptoms
Acronym: REPLENISH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TherapeuticsMD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TXC12-05; REPLENISH Trial (Other: Sponsor)
Record Dates: First submitted 2013-09-05; First posted 2013-09-16 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-04

CONDITIONS: Menopause
Keywords: Vasomotor symptoms; Hot flashes; Endometrial protection
MeSH Terms: conditions — Hot Flashes | interventions — Estradiol; Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment 1 (Experimental): Combined Estradiol 1 mg / Progesterone 100 mg softgel capsule formulation and placebo taken orally once a day for twelve months.
  Interventions: Drug: Estradiol; Drug: Progesterone; Drug: Placebo
- Treatment 2 (Experimental): Combined Estradiol 0.5 mg / Progesterone 100 mg softgel capsule formulation and placebo taken orally once a day for twelve months.
  Interventions: Drug: Estradiol; Drug: Progesterone; Drug: Placebo
- Treatment 3 (Experimental): Combined Estradiol 0.5 mg / Progesterone 50 mg softgel capsule formulation and placebo, taken orally once a day for twelve months.
  Interventions: Drug: Estradiol; Drug: Progesterone; Drug: Placebo
- Treatment 4 (Experimental): Combined Estradiol 0.25 mg / Progesterone 50 mg softgel capsule formulation and placebo, taken orally once a day for twelve months.
  Interventions: Drug: Estradiol; Drug: Progesterone; Drug: Placebo
- Placebo (Placebo Comparator): Two Placebo softgel capsules taken orally once a day for twelve months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Estradiol
  Other Names: 17B-estradiol; Estrace
  Arms: Treatment 1; Treatment 2; Treatment 3; Treatment 4
Drug: Progesterone
  Other Names: Prometrium
  Arms: Treatment 1; Treatment 2; Treatment 3; Treatment 4
Drug: Placebo

SUMMARY:
This study will be a prospective, randomized, double-blind, placebo-controlled, parallel group, multicenter trial of postmenopausal subjects with an intact uterus.

DETAILED DESCRIPTION:
Postmenopausal subjects with an intact uterus who meet the study entry criteria will be randomized to one of five treatment arms (four active and one placebo) and followed for 12 months. During the Screening period all subjects will be provided with a diary to self-assess the frequency and severity of their vasomotor symptoms. Subjects experiencing a minimum daily frequency of ≥7 (or ≥50 per week) moderate to severe hot flushes will participate in a VMS Substudy during the first 12 weeks of treatment. The Substudy subjects will be stratified by treatment arm within the sites, and only Substudy subjects have the possibility of being randomized to placebo. Subjects who qualify for the study except for experiencing a minimum daily frequency of ≥7 (or ≥50 per week) moderate to severe hot flushes will be stratified within sites to one of the four active treatment arms and followed for 12 months, but will not participate in the VMS Substudy. (However, VMS information will be collected from all subjects during the first 12 weeks of treatment.) All Study Subjects: Postmenopausal women with an intact uterus who seek relief from hot flushes and meet all other inclusion/exclusion criteria are eligible for 12 months of study treatment.

VMS Substudy Subjects: A subset of All Study Subjects who have ≥7 per day or ≥50 per week moderate to severe hot flushes (as determined during Screening) are eligible for the 12-week VMS Substudy and for a total of 12 months of study treatment.

Clinical evaluations will be performed at the following time points:

* Screening Period (Week: - 8.5) (up to -60 Days)
* Visit 1 Randomization (Week 0) (Day 1)
* Visit 2 Interim (Week 4)
* Visit 3 Interim (Week 8)
* Visit 4 Interim (Week 12)
* Visit 5 Interim (Month 6)
* Visit 6 Interim (Month 9)
* Visit 7 End of Treatment (Month 12)

ELIGIBILITY:
Inclusion Criteria:

1. Be a female between the ages of 40 and 65 years (at the time of randomization) who is willing to participate in the study, as documented by signing the informed consent form.
2. Be a postmenopausal woman with an intact uterus and a Screening serum estradiol level of ≤50 pg/mL. Postmenopausal is defined herein as:

   1. ≥ 12 months of spontaneous amenorrhea, or
   2. at least 6 months of spontaneous amenorrhea with a Screening serum FSH level of >40 mIU/ml, or
   3. ≥ 6 weeks postsurgical bilateral oophorectomy.
3. Be seeking treatment or relief for vasomotor symptoms associated with menopause.
4. To participate in the VMS Substudy, a subject must also report ≥7 moderate to severe hot flushes per day, or ≥50 per week, at the baseline assessment during Screening (subjects whose hot flushes are less frequent may still participate as non-Substudy subjects.

   Note: A minimum of 14 consecutive days of complete hot flush diary data are required during the baseline assessment at Screening, and these consecutive days must occur within the last 14 days prior to the Randomization visit (not counting the Randomization visit day itself). The most recent 7 consecutive days of data prior to randomization (Day -7 to Day -1) will be used to determine the baseline number of mild, moderate and severe hot flushes for each subject.
5. Have a Body Mass Index (BMI) less than or equal to 34 kg/mP2P. (BMI values should be rounded to the nearest integer [e.g., 34.4 rounds down to 34, while 26.5 rounds up to 27]).
6. Be willing to abstain from using products (other than study medication) that contain estrogen, progestin, or progesterone throughout study participation.
7. Be judged by the principal or sub-investigator physician as being in otherwise generally good health based on a medical evaluation performed during the Screening period prior to the initial dose of study medication. The medical evaluation findings must include:

   1. a normal or non-clinically significant physical examination, including vital signs (sitting blood pressure, heart rate, respiratory rate and temperature). Sitting systolic blood pressure is ≤140 mmHg and diastolic blood pressure ≤90 mmHg at Screening. A subject may be taking up to two antihypertensive medications.
   2. a normal or non-clinically significant pelvic examination.
   3. a mammogram that shows no sign of significant disease (can be performed within previous 6 months prior to initial dose of study medication). Subjects must have a BI-RADS 1 or 2 to enroll in the study. An incomplete mammogram result, i.e. BI-RADS 0, is not acceptable. The site must obtain a copy of the official report for the subject's study file, and it must be verified that the mammogram itself is available if needed for additional assessment.
   4. a normal or non-clinically significant clinical breast examination. An acceptable breast examination is defined as no masses or other findings identified that are suspicious of malignancy.
   5. a normal Screening Papanicolaou ("Pap") smear. (Subjects with findings of atypical glandular cells [AGC], AGUS, ASCUS with high risk HPV type upon reflex testing, LSIL, ASC-H, HSIL, dysplastic cells, or malignant cells must be excluded from randomization.)
   6. an acceptable result from an evaluable Screening endometrial biopsy. The endometrial biopsy reports by the two central pathologists at Screening must each specify one of the following: proliferative endometrium; weakly proliferative endometrium; disordered proliferative pattern; secretory endometrium; endometrial tissue other (including benign, inactive or atrophic fragments of endometrial epithelium, glands, stroma, etc); endometrial tissue insufficient for diagnosis; no endometrium identified; or no tissue identified. However, at least one pathologist must identify sufficient tissue to evaluate the biopsy. Additionally, the endometrial biopsy reports by the two central pathologists of Other Findings at Screening must each specify one of the following: endometrial polyp not present; benign endometrial polyp; or polyp other. (See Exclusion criterion #27)
   7. a normal or non-clinically significant 12-lead ECG.

Exclusion Criteria:

* To participate in the study, a subject must NOT:

  1. Be currently hospitalized.
  2. Have a history of thrombosis of deep veins or arteries or a thromboembolic disorder.
  3. Have a history of coronary artery or cerebrovascular disease (e.g., myocardial infarction, angina, stroke, TIA).
  4. Have a history of a chronic liver or kidney dysfunction/disorder (e.g., Hepatitis C or chronic renal failure).
  5. Have a history of a malabsorption disorder (e.g., gastric bypass, Crohn's disease).
  6. Have a history of gallbladder dysfunction/disorders (e.g., cholangitis, cholecystitis), unless gallbladder has been removed.
  7. Have a history of diabetes, thyroid disease or any other endocrinological disease. (Subjects with diet-controlled diabetes or controlled hypothyroid disease at Screening are not excluded.)
  8. Have a history of estrogen-dependent neoplasia.
  9. Have a history of atypical ductal hyperplasia of the breast.
  10. Have a finding of clinically significant uterine fibroids at Screening.
  11. Have had a uterine ablation.
  12. Have a history of undiagnosed vaginal bleeding.
  13. Have any history of endometrial hyperplasia, melanoma, or uterine/endometrial, breast or ovarian cancer.
  14. Have any history of other malignancy within the last 5 years, with the exception of basal cell (excluded if within 1 year) or non-invasive squamous cell (excluded if within 1 year) carcinoma of the skin.
  15. Have a history of any other cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychological (e.g., bipolar disorder, schizophrenia, major depressive disorder), or musculoskeletal disease or disorder that is clinically significant in the opinion of the Principal Investigator or Medical Sub-Investigator.
  16. Have any of the following clinical laboratory values at Screening:

      1. fasting triglyceride of ≥300 mg/dL and/or total cholesterol of ≥300mg/dL
      2. positive laboratory finding for Factor V Leiden mutation
      3. AST or ALT ≥1.5 times the upper limit of normal (ULN)
      4. fasting glucose >125 mg/dL
  17. Be known to be pregnant or have a positive urine pregnancy test. (Note: A pregnancy test is not required for subjects who have had bilateral tubal ligation, bilateral oophorectomy, or are 55 years old or greater and have experienced cessation of menses for at least 1 year.)
  18. Have contraindication to estrogen and/or progestin therapy or allergy to the use of estradiol and/or progesterone or any components of the investigational drugs.
  19. Use 15 or more cigarettes per day or currently use any electronic cigarettes.
  20. Have a history of drug and/or alcohol abuse within one year of start of study.
  21. Have used, within 28 days prior to the initial dose of study medication at Visit 1, any medication known to induce or inhibit CYP3A4 enzyme activity that may affect estrogen and/or progestin drug metabolism. (See 48TUSection 4.3U48T)
  22. Have used, within 28 days prior to Screening, or plan to use during the study, any prescription or over-the-counter (OTC) medications (including herbal products, such as St. John's Wort) that would be expected to alter progesterone or estrogen activity or is being used to treat vasomotor symptoms. (See Section 4.3U48T)
  23. Have used estrogen alone or estrogen/progestin, SERM (selective estrogen receptor modulator), testosterone, or estrogen/testosterone for any of the following time periods:

      1. Vaginal nonsystemic hormonal products (rings, creams, gels) within 7 days prior to Screening, or vaginal systemic products (e.g., FemRing) within 28 days prior to Screening.
      2. Transdermal estrogen alone or estrogen/progestin products within 8 weeks prior to Screening.
      3. Oral estrogen and/or progestin and/or SERM therapy within 8 weeks prior to Screening.
      4. Progestational implants, estrogen or estrogen/progestational injectable drug therapy within 3 months prior to Screening.
      5. Estrogen pellet therapy or progestational injectable drug therapy within 6 months prior to Screening.
      6. Percutaneous estrogen lotions/gels within 8 weeks prior to Screening.
      7. Oral, topical, vaginal, patch, implantable or injectable androgen therapy within 8 weeks prior to Screening.
  24. Have used an intrauterine device (IUD) within the 12 weeks prior to Screening.
  25. For subjects in the VMS Substudy only: use of medication that may affect the outcome of the vasomotor symptom endpoints within 28 days prior to Screening (e.g. SSRIs [selective serotonin reuptake inhibitors], SNRIs [serotonin and norepinephrine reuptake inhibitors], aldomet, dopaminergic or antidopaminergic drugs, gabapentin, clonidine, or bellergal.)
  26. Have any reason which, in the opinion of the Principal Investigator or Medical Sub-Investigator, would prevent the subject from safely participating in the study or complying with protocol requirements.
  27. Have a Screening endometrial biopsy sample that is found by both primary pathologists to have endometrial tissue insufficient for diagnosis, no endometrium identified, or no tissue identified. (With the approval of the Medical Monitor, the Screening endometrial biopsy may be repeated once.)
  28. Endometrial polyps with atypical nuclei reported by at least 1 central pathologist.
  29. Have contraindication to any planned study assessments (e.g., endometrial biopsy).
  30. Have participated in another clinical trial within 30 days prior to Screening, have received an investigational drug within the three months prior to the initial dose of study medication, or be likely to participate in a clinical trial or receive another investigational medication during the study.
  31. Currently use marijuana.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1845 (Actual)
Dates: Start 2013-08-05 (Actual); Primary Completion 2016-10-28 (Actual); Study Completion 2016-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Mirkin, MD, Study Director — TherapeuticsMD
Locations (119):
- United States (119):
  - Simon Williamson Clinic, Birmingham, Alabama
  - Medical Affiliated Research Center, Huntsville, Alabama
  - Coastal Clinical Research, Mobile, Alabama
  - Mobile Ob-Gyn, P.C., Mobile, Alabama
  - Montgomery Women's Health, Montgomery, Alabama
  - Advanced Research Associates, Glendale, Arizona
  - Cactus Clinical Research, Mesa, Arizona
  - Precision Trials, Phoenix, Arizona
  - Radiant Research (Tucson), Tucson, Arizona
  - Visions Clinical Research Tucson, Tucson, Arizona
  - Health Star Research, LLC, Hot Springs, Arkansas
  - Sutter East Bay Medical Foundation, Berkeley, California
  - Grossmont Center for Clinical Research, La Mesa, California
  - Futura Research, Norwalk, California
  - Medical Center for Clinical Research, San Diego, California
  - Women's Health Care Research Corp., San Diego, California
  - Radiant Research, Inc., Santa Rosa, California
  - Diablo Clinical Research, Walnut Creek, California
  - Downtown Women's Healthcare, Denver, Colorado
  - Horizon's Clinical Research Center, Denver, Colorado
  - Red Rocks OB/Gyn, Lakewood, Colorado
  - Clinical Research Consulting, Milford, Connecticut
  - Coastal Connecticut Research, New London, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Nature Coast Clinical Research, Crystal River, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - Southeastern Integrated Medical, PL, d/b/a Florida Medical Research, Gainesville, Florida
  - UF College of Medicine-Jacksonville, Dept. of Obstetrics and Gynecology, Jacksonville, Florida
  - Suncoast Research, Margate, Florida
  - Accelovance, Melbourne, Florida
  - Suncoast Clinical Research, Inc, New Port Richey, Florida
  - Segal Institute, North Miami, Florida
  - Ideal Clinical Research, North Miami Beach, Florida
  - Compass Research, Orlando, Florida
  - Radiant Research (St. Petersburg), Pinellas Park, Florida
  - All Women's Healthcare of West Broward Discovery Clinical Research, Plantation, Florida
  - Comprehensive Clinical Trials, West Palm Beach, Florida
  - Radiant Research (Atlanta), Atlanta, Georgia
  - Women's Health Associates, Atlanta, Georgia
  - Soapstone Center for Clinical Research, Decatur, Georgia
  - Wake Research - Mount Vernon Clinical Research, Sandy Springs, Georgia
  - Fellows Research Alliance, Savannah, Georgia
  - Elite Clinical Trials, Blackfoot, Idaho
  - Advanced Clinical Research, Meridian, Idaho
  - Biofortis, Addison, Illinois
  - Women's Health Practice, Champaign, Illinois
  - Radiant Research (Chicago), Chicago, Illinois
  - The South Bend Clinic Granger, Granger, Indiana
  - Davis Clinic, Indianapolis, Indiana
  - Cypress Medical Research Center, LLC, Wichita, Kansas
  - Central Kentucky Research Associates, Lexington, Kentucky
  - Bluegrass Clinical Research, Louisville, Kentucky
  - Horizon Research Group, Eunice, Louisiana
  - Maryland Center for Sexual Health, Lutherville, Maryland
  - Quest Research Institute, Bingham Farms, Michigan
  - Female Pelvic Medicine & Urogynecology, Grand Rapids, Michigan
  - Beyer Research, Kalamazoo, Michigan
  - Saginaw Valley Medical Research Group, Saginaw, Michigan
  - Radiant Research (St. Louis), St Louis, Missouri
  - Billings Clinical Research, Billings, Montana
  - Montana Health, Billings, Montana
  - Women's Clinic of Lincoln, Lincoln, Nebraska
  - Affiliated Clinical Research INC, Las Vegas, Nevada
  - Affiliated Clinical Research, Las Vegas, Nevada
  - Lawrence OB-GYN Clinical Research, Lawrenceville, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Bosque Women's Care, Albuquerque, New Mexico
  - Southwest Clinical Research, Albuquerque, New Mexico
  - Columbia University, New York, New York
  - Suffolk OB/GYN, Port Jefferson, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - Women's Wellness Clinic, Durham, North Carolina
  - Carolina Medical Trials, High Point, North Carolina
  - Centre OBGYN, Raleigh, North Carolina
  - Wake County Research, Raleigh, North Carolina
  - Lyndhurst Clinical Research, Salem, North Carolina
  - Carolina Medical Trials, Winston-Salem, North Carolina
  - Hawthorne Research, Winston-Salem, North Carolina
  - Triad Ob-Gyn, Winston-Salem, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - Radiant Research (Akron), Akron, Ohio
  - University of Cincinnati Physicians Company, Cincinnati, Ohio
  - Rapid Medical Research, Cleveland, Ohio
  - Columbus Center for Women's Health Research, Columbus, Ohio
  - HWC Women's Research Center, Englewood, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Sunstone Medical Research, Medford, Oregon
  - The Clinical Trial Center, Jenkintown, Pennsylvania
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - Clinical Trials Research Services, LLC, Pittsburgh, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Fellows Research Group, Bluffton, South Carolina
  - Vista Clinical Research, Columbia, South Carolina
  - Upstate Pharmaceutical Research, Greenville, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Chattanooga Medical Research, Chattanooga, Tennessee
  - Volunteer Research Group/NOCCR, Knoxville, Tennessee
  - DiscoveResearch, Inc., Bryan, Texas
  - Advanced Research Associates, Corpus Christi, Texas
  - Research Across America, Dallas, Texas
  - Brownstone Clinical Trials, Fort Worth, Texas
  - Advances in Health, Houston, Texas
  - The Women's Hospital of Texas, Houston, Texas
  - TMC Life Research, Houston, Texas
  - Protenium Clinical Research, Hurst, Texas
  - MacArthur OB/GYN, Irving, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Stone Oak, LLC dba Discovery Clinical Trials, San Antonio, Texas
  - NECRSA, Schertz, Texas
  - PRO/ Salt Lake Women's Center, Draper, Utah
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Jean Brown Research, Salt Lake City, Utah
  - UVA/Midlife Health at North Ridge, Charlottesville, Virginia
  - Clinical Research Center Eastern Virginia Medical School, Norfolk, Virginia
  - Virginia Women's Center, Richmond, Virginia
  - National Clinical Research-Richmond, Inc, Richmond, Virginia
  - Tidewater Clinical Research, Virginia Beach, Virginia
  - Seattle Women's Health Research, Gynecology, Seattle, Washington
  - North Spokane Women's Health, Spokane, Washington

REFERENCES:
- [Background] Hilditch JR, Lewis J, Peter A, van Maris B, Ross A, Franssen E, Guyatt GH, Norton PG, Dunn E. A menopause-specific quality of life questionnaire: development and psychometric properties. Maturitas. 1996 Jul;24(3):161-75. doi: 10.1016/s0378-5122(96)82006-8. PMID 8844630
- [Background] Gerlinger C, Gude K, Hiemeyer F, Schmelter T, Schafers M. An empirically validated responder definition for the reduction of moderate to severe hot flushes in postmenopausal women. Menopause. 2012 Jul;19(7):799-803. doi: 10.1097/gme.0b013e31823de8ba. PMID 22228322
- [Background] Spritzer, K. L. & Hays, R. D. (2003, November). MOS Sleep Scale: A Manual for Use and Scoring, Version 1.0. Los Angeles, CA.
- [Background] Kurman RJ, Ellenson L H, and Ronnett B.M., ed. Blaustein's Pathology of the Female Genital Tract. 6th ed. New York, NY: Springer; 2011:305-452.
- [Background] Revicki D, Hays RD, Cella D, Sloan J. Recommended methods for determining responsiveness and minimally important differences for patient-reported outcomes. J Clin Epidemiol. 2008 Feb;61(2):102-9. doi: 10.1016/j.jclinepi.2007.03.012. Epub 2007 Aug 3. PMID 18177782
- [Background] Hays RD and Stewart AL. Sleep measures. In AL Stewart & JE Ware (eds), Measuring functioning and well-being: The Medical Outcomes Study approach (pp 235-259). Durham, NC: Duke University Press, 1992.
- [Derived] McClung MR, Kagan R, Graham S, Bernick B, Mirkin S, Constantine G. Effects of E2/P4 oral capsules on bone turnover in women with vasomotor symptoms. Menopause. 2022 Feb 14;29(3):304-308. doi: 10.1097/GME.0000000000001915. PMID 35213517
- [Derived] Constantine GD, Simon JA, Kaunitz AM, Pickar JH, Revicki DA, Graham S, Bernick B, Mirkin S. TX-001HR is associated with a clinically meaningful effect on severity of moderate to severe vasomotor symptoms in the REPLENISH trial. Menopause. 2020 Nov;27(11):1236-1241. doi: 10.1097/GME.0000000000001602. PMID 33110039
- [Derived] Black DR, Minkin MJ, Graham S, Bernick B, Mirkin S. Effects of combined 17beta-estradiol and progesterone on weight and blood pressure in postmenopausal women of the REPLENISH trial. Menopause. 2020 Sep 14;28(1):32-39. doi: 10.1097/GME.0000000000001659. PMID 32932401
- [Derived] Kaunitz AM, Bitner D, Constantine GD, Bernick B, Graham S, Mirkin S. 17beta-estradiol/progesterone in a single, oral, softgel capsule (TX-001HR) significantly increased the number of vasomotor symptom-free days in the REPLENISH trial. Menopause. 2020 Dec;27(12):1382-1387. doi: 10.1097/GME.0000000000001615. PMID 32740481
- [Derived] Mirkin S, Goldstein SR, Archer DF, Pickar JH, Graham S, Bernick B. Endometrial safety and bleeding profile of a 17beta-estradiol/progesterone oral softgel capsule (TX-001HR). Menopause. 2020 Apr;27(4):410-417. doi: 10.1097/GME.0000000000001480. PMID 31913228
- [Derived] Lobo RA, Kaunitz AM, Santoro N, Bernick B, Graham S, Mirkin S. Metabolic and cardiovascular effects of TX-001HR in menopausal women with vasomotor symptoms. Climacteric. 2019 Dec;22(6):610-616. doi: 10.1080/13697137.2019.1640197. Epub 2019 Jul 31. PMID 31364889
- [Derived] Mirkin S, Graham S, Revicki DA, Bender RH, Bernick B, Constantine GD. Relationship between vasomotor symptom improvements and quality of life and sleep outcomes in menopausal women treated with oral, combined 17beta-estradiol/progesterone. Menopause. 2019 Jan 9;26(6):637-642. doi: 10.1097/GME.0000000000001294. PMID 30601452
- [Derived] Kagan R, Constantine G, Kaunitz AM, Bernick B, Mirkin S. Improvement in sleep outcomes with a 17beta-estradiol-progesterone oral capsule (TX-001HR) for postmenopausal women. Menopause. 2018 Dec 21;26(6):622-628. doi: 10.1097/GME.0000000000001278. PMID 30586005
- [Derived] Lobo RA, Archer DF, Kagan R, Kaunitz AM, Constantine GD, Pickar JH, Graham S, Bernick B, Mirkin S. A 17beta-Estradiol-Progesterone Oral Capsule for Vasomotor Symptoms in Postmenopausal Women: A Randomized Controlled Trial. Obstet Gynecol. 2018 Jul;132(1):161-170. doi: 10.1097/AOG.0000000000002645. PMID 29889748
- [Derived] Mirkin S, Amadio JM, Bernick BA, Pickar JH, Archer DF. 17beta-Estradiol and natural progesterone for menopausal hormone therapy: REPLENISH phase 3 study design of a combination capsule and evidence review. Maturitas. 2015 May;81(1):28-35. doi: 10.1016/j.maturitas.2015.02.266. Epub 2015 Mar 9. PMID 25835751

RESULTS

PARTICIPANT FLOW:
Groups:
- Combined Estradiol 1 mg / Progesterone 100 mg: Combined Estradiol 1 mg / Progesterone 100 mg formulation and placebo softgel capsules taken orally once a day for twelve months.
- Combined Estradiol 0.5 mg / Progesterone 100 mg: Combined Estradiol 0.5 mg / Progesterone 100 mg formulation and placebo softgel capsules taken orally once a day for twelve months.
- Combined Estradiol 0.5 mg / Progesterone 50 mg: Combined Estradiol 0.5 mg / Progesterone 50 mg formulation and placebo softgel capsules taken orally once a day for twelve months.
- Combined Estradiol 0.25 mg / Progesterone 50 mg: Combined Estradiol 0.25 mg / Progesterone 50 mg formulation and placebo softgel capsules taken orally once a day for twelve months.
Period: Overall Study
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Started (Number of subjects started reflects total number of subjects randomized per arm.) | 418 | 426 | 422 | 427 | 152
Completed | 284 | 305 | 312 | 281 | 93
Not Completed | 134 | 121 | 110 | 146 | 59

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo | Total
Number analyzed (Participants) | 415 | 424 | 421 | 424 | 151 | 1835
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 415 | 424 | 421 | 424 | 151 | 1835
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (4.37) | 54.5 (4.52) | 54.9 (4.27) | 54.4 (4.04) | 54.5 (4.32) | 54.6 (4.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 415 | 424 | 421 | 424 | 151 | 1835
  Male | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 415 | 424 | 421 | 424 | 151 | 1835

OUTCOME MEASURES:

1. Primary Outcome: Co-Primary Efficacy Endpoint: Frequency of Moderate to Severe Vasomotor Symptoms (MITT-VMS)
Description: Mean change in frequency of moderate to severe vasomotor symptoms from Baseline to Week 4. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of moderate to severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of moderate to severe hot flushes for the subject week.
Time Frame: Baseline and Week 4
Population: Randomized to the VMS Substudy, taken one dose of IP, and had at least 5 days of VMS diary data for baseline measurement of freq. & severity of moderate to severe hot flushes, and had at least 4 days of VMS diary data for 1 on-treatment week of reporting freq. & severity of hot flushes following initiation of IP.
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 134 | 144 | 142 | 152 | 126
weekly hot flushes | -40.6 (30.59) | -35.1 (29.14) | -33.6 (30.64) | -38.9 (31.04) | -26.4 (27.05)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 4; Each co-primary endpt in each dose group tested at alpha=0.05;multiple dose groups vs. PBO comparisons are conducted using gatekeeping procedure; Mean Difference (Final Values) = -12.81, 95% CI 2-sided [-19.29 to -6.32], Standard Error of Mean 3.30 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.013, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 4; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.07, 95% CI 2-sided [-14.46 to -1.68], Standard Error of Mean 3.25 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.141, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 4; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.81, 95% CI 2-sided [-11.21 to 1.59], Standard Error of Mean 3.26 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 4; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -10.40, 95% CI 2-sided [-16.73 to -4.08], Standard Error of Mean 3.22 — Adjusted for baseline using MMRM

2. Primary Outcome: Co-Primary Efficacy Endpoint: Frequency of Moderate to Severe Vasomotor Symptoms (MITT-VMS)
Description: Mean change in frequency of moderate to severe vasomotor symptoms from Baseline to Week 12. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of moderate to severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of moderate to severe hot flushes for the subject week.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 129 | 124 | 135 | 115
weekly hot flushes | -55.1 (31.36) | -53.7 (31.93) | -50.2 (31.35) | -52.4 (33.90) | -40.2 (29.79)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -16.58, 95% CI 2-sided [-23.33 to -9.82], Standard Error of Mean 3.44 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -15.07, 95% CI 2-sided [-21.72 to -8.42], Standard Error of Mean 3.39 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -10.79, 95% CI 2-sided [-17.48 to -4.10], Standard Error of Mean 3.41 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -11.71, 95% CI 2-sided [-18.31 to -5.11], Standard Error of Mean 3.36 — Adjusted for baseline using MMRM

3. Primary Outcome: Co-Primary Efficacy Endpoint: Severity of Moderate to Severe Vasomotor Symptoms (MITT-VMS)
Description: Mean change in severity of moderate to severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 4. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score = (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of moderate to severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 134 | 144 | 142 | 152 | 126
scores on a scale | -0.48 (0.547) | -0.51 (0.563) | -0.40 (0.469) | -0.44 (0.514) | -0.34 (0.386)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.031, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 4; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.25 to -0.01], Standard Error of Mean 0.061 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.005, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 4; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.28 to -0.05], Standard Error of Mean 0.060 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.401, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 4; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.17 to 0.07], Standard Error of Mean 0.060 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.100, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 4; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.21 to 0.02], Standard Error of Mean 0.059 — Adjusted for baseline using MMRM

4. Primary Outcome: Co-Primary Efficacy Endpoint: Severity of Moderate to Severe Vasomotor Symptoms (MITT-VMS)
Description: Mean change in severity of moderate to severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 12. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score = (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of moderate to severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 129 | 124 | 135 | 115
scores on a scale | -1.12 (0.963) | -0.90 (0.783) | -0.76 (0.744) | -0.71 (0.806) | -0.56 (0.603)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-0.77 to -0.38], Standard Error of Mean 0.100 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.59 to -0.20], Standard Error of Mean 0.099 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.018, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.43 to -0.04], Standard Error of Mean 0.100 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.096, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.36 to 0.03], Standard Error of Mean 0.098 — Adjusted for baseline using MMRM

5. Primary Outcome: Primary Safety Endpoint: Endometrial Protection - Hyperplasia
Description: Endometrial biopsies centrally evaluated by 2 primary pathologists using criteria from Blaustein's Pathology text. Pathologists classified bx into 1 of following 3 categories: Cat.1: Non-endometrial malignancy/non-hyperplasia; Cat.2: Endometrial hyperplasia; Cat.3: Endometrial malignancy. Consensus reached when 2 primary pathologist agreed on any of above categories; if primary pathologists disagreed on presence of hyperplasia, result of 3rd pathologist was utilized and final decision regarding presence of hyperplasia was based on diagnosis of majority. If all 3 reads disparate, final diagnosis based on most severe dx. Incidence rate calculated as: I=A/B where I=incidence rate at M12 evaluation, A=all new subjects with biopsies positive for endometrial hyperplasia during study but post-Baseline, B=all subjects w/biopsies following M11 meeting criteria specified plus all subjects w/biopsies positive for endometrial hyperplasia by any pathologists before M11.
Time Frame: Baseline and Month 12
Population: Randomized subjects who had taken at least 1 capsule, had no major protocol violations, acceptable biopsy at baseline (evaluable tissue, no endometrial hyperplasia, polyp or cancer), had a biopsy at month 12 (on or after Study Day 326) or had a diagnosis of endometrial hyperplasia prior to month 12.
Measure: Count of Participants; unit: Participants
Groups:
- Combined Estradiol 1 mg / Progesterone 100 mg: Combined Estradiol 1 mg / Progesterone 100 mg formulation taken orally once a day for twelve months.
- Combined Estradiol 0.5 mg / Progesterone 100 mg: Combined Estradiol 0.5 mg / Progesterone 100 mg formulation taken orally once a day for twelve months.
- Combined Estradiol 0.5 mg / Progesterone 50 mg: Combined Estradiol 0.5 mg / Progesterone 50 mg formulation taken orally once a day for twelve months.
- Combined Estradiol 0.25 mg / Progesterone 50 mg: Combined Estradiol 0.25 mg / Progesterone 50 mg formulation taken orally once a day for twelve months.
- Placebo: Two Placebo capsules taken orally once a day for twelve months.
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 280 | 303 | 306 | 274 | 92
Participants | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg; Between group comparison is not intended. The purpose of the analysis is to calculate the incidence rate and the 95% CI of endometrial hyperplasia per FDA published guidance for Combined Estradiol 1 mg / Progesterone 100 mg; Test type: Other — Per FDA guidance hyperplasia proportion must be <=1% with an upper bound of the one-sided 95% confidence interval <=4%; Between group comparison was not performed; incidence rate = 0, 95% CI 1-sided [upper limit 1.06] — This calculation is based on a binomial distribution
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg; Between group comparison is not intended. The purpose of the analysis is to calculate the incidence rate and the 95% CI of endometrial hyperplasia per FDA published guidance for Combined Estradiol 0.5 mg / Progesterone 100 mg; Test type: Other — Per FDA guidance hyperplasia proportion must be <=1% with an upper bound of the one-sided 95% confidence interval <=4%; Between group comparison was not performed; incidence rate = 0, 95% CI 1-sided [upper limit 0.98] — This calculation is based on a binomial distribution
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg; Between group comparison is not intended. The purpose of the analysis is to calculate the incidence rate and the 95% CI of endometrial hyperplasia per FDA published guidance for Combined Estradiol 0.5 mg / Progesterone 50 mg; Test type: Other — Per FDA guidance hyperplasia proportion must be <=1% with an upper bound of the one-sided 95% confidence interval <=4%; Between group comparison was not performed; incidence rate = 0, 95% CI 1-sided [upper limit 0.97] — This calculation is based on a binomial distribution
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg; Between group comparison is not intended. The purpose of the analysis is to calculate the incidence rate and the 95% CI of endometrial hyperplasia per FDA published guidance for Combined Estradiol 0.25 mg / Progesterone 50 mg; Test type: Other — Per FDA guidance hyperplasia proportion must be <=1% with an upper bound of the one-sided 95% confidence interval <=4%; Between group comparison was not performed; incidence rate = 0, 95% CI 1-sided [upper limit 1.09] — This calculation is based on a binomial distribution
Statistical Analysis 5: Comparison: Placebo; Between group comparison is not intended. The purpose of the analysis is to calculate the incidence rate and the 95% CI of endometrial hyperplasia per FDA published guidance for Placebo; Test type: Other — Per FDA guidance hyperplasia proportion must be <=1% with an upper bound of the one-sided 95% confidence interval <=4%; Between group comparison was not performed; incidence rate = 0, 95% CI 1-sided [upper limit 3.20] — This calculation is based on a binomial distribution

6. Secondary Outcome: Endometrial Protection - Hyperplasia
Description: Endometrial biopsies centrally evaluated by 3 primary pathologists using criteria described in Blaustein's Pathology text. Pathologists classified biopsy into 1 of following 3 categories: Cat.1: Non-endometrial malignancy/non-hyperplasia; Cat.2: Endometrial hyperplasia; Cat.3: Endometrial malignancy. Consensus was reached when the 2 of 3 pathologist readers agreed on any of the above categories; if all three reads were disparate, the final diagnosis was based on the most severe diagnosis. Incidence rate calculated as: I=A/B where I=incidence rate at M12 evaluation, A=all new subjects with biopsies positive for endometrial hyperplasia during study but post-Baseline, B=all subjects with biopsies following M11 meeting the criteria specified plus all subjects with biopsies positive for endometrial hyperplasia by any of the pathologists before M11.
Time Frame: Baseline and Month 12
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 280 | 303 | 306 | 274 | 92
Participants | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg; [analysis description as in outcome 5, analysis 1]; Test type: Other — Per FDA guidance hyperplasia proportion must be <=1% with an upper bound of the one-sided 95% confidence interval <=4%; Between group comparison was not performed; incidence rate = 0, 95% CI 1-sided [upper limit 1.06] — This calculation is based on a binomial distribution
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg; [analysis description as in outcome 5, analysis 2]; Test type: Other — Per FDA guidance hyperplasia proportion must be <=1% with an upper bound of the one-sided 95% confidence interval <=4%; Between group comparison was not performed; incidence rate = 0, 95% CI 1-sided [upper limit 0.98] — This calculation is based on a binomial distribution
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg; [analysis description as in outcome 5, analysis 3]; Test type: Other — Per FDA guidance hyperplasia proportion must be <=1% with an upper bound of the one-sided 95% confidence interval <=4%; Between group comparison was not performed; incidence rate = 0, 95% CI 1-sided [upper limit 0.97] — This calculation is based on a binomial distribution
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg; [analysis description as in outcome 5, analysis 4]; Test type: Other — Per FDA guidance hyperplasia proportion must be <=1% with an upper bound of the one-sided 95% confidence interval <=4%; Between group comparison was not performed; incidence rate = 0, 95% CI 1-sided [upper limit 1.09] — This calculation is based on a binomial distribution
Statistical Analysis 5: Comparison: Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Other — Per FDA guidance hyperplasia proportion must be <=1% with an upper bound of the one-sided 95% confidence interval <=4%; Between group comparison was not performed; incidence rate = 0, 95% CI 1-sided [upper limit 3.20] — This calculation is based on a binomial distribution

7. Secondary Outcome: Frequency of Moderate to Severe Vasomotor Symptoms - Week 1 (MITT-VMS)
Description: Mean change in frequency of moderate to severe vasomotor symptoms from Baseline to Week 1. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of moderate to severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of moderate to severe hot flushes for the subject week.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 138 | 149 | 145 | 154 | 134
weekly hot flushes | -12.2 (20.10) | -11.5 (20.19) | -11.0 (20.94) | -16.3 (22.28) | -13.0 (21.25)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.588, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 1; Mean Difference (Final Values) = 1.36, 95% CI 2-sided [-3.57 to 6.30], Standard Error of Mean 2.51 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.601, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 1; Mean Difference (Final Values) = 1.29, 95% CI 2-sided [-3.56 to 6.15], Standard Error of Mean 2.47 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.202, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 1; Mean Difference (Final Values) = 3.17, 95% CI 2-sided [-1.71 to 8.06], Standard Error of Mean 2.49 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.431, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 1; Mean Difference (Final Values) = -1.93, 95% CI 2-sided [-6.76 to 2.89], Standard Error of Mean 2.46 — Adjusted for baseline using MMRM

8. Secondary Outcome: Frequency of Moderate to Severe Vasomotor Symptoms - Week 2 (MITT-VMS)
Description: Mean change in frequency of moderate to severe vasomotor symptoms from Baseline to Week 2. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of moderate to severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of moderate to severe hot flushes for the subject week.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 134 | 146 | 145 | 153 | 133
weekly hot flushes | -26.6 (27.67) | -21.2 (24.79) | -19.0 (28.32) | -25.4 (26.63) | -21.3 (24.75)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.154, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 2; Mean Difference (Final Values) = -4.35, 95% CI 2-sided [-10.34 to 1.64], Standard Error of Mean 3.05 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.956, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 2; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-6.06 to 5.73], Standard Error of Mean 3.00 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.240, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 2; Mean Difference (Final Values) = 3.54, 95% CI 2-sided [-2.37 to 9.46], Standard Error of Mean 3.01 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.353, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 2; Mean Difference (Final Values) = -2.77, 95% CI 2-sided [-8.62 to 3.08], Standard Error of Mean 2.98 — Adjusted for baseline using MMRM

9. Secondary Outcome: Frequency of Moderate to Severe Vasomotor Symptoms - Week 3 (MITT-VMS)
Description: Mean change in frequency of moderate to severe vasomotor symptoms from Baseline to Week 3. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of moderate to severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of moderate to severe hot flushes for the subject week.
Time Frame: Baseline and Week 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 136 | 144 | 144 | 153 | 131
weekly hot flushes | -34.3 (29.22) | -29.0 (26.73) | -28.1 (28.18) | -33.6 (27.76) | -25.1 (27.26)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.007, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 3; Mean Difference (Final Values) = -8.56, 95% CI 2-sided [-14.75 to -2.36], Standard Error of Mean 3.16 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.227, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 3; Mean Difference (Final Values) = -3.76, 95% CI 2-sided [-9.86 to 2.35], Standard Error of Mean 3.11 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.597, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 3; Mean Difference (Final Values) = -1.65, 95% CI 2-sided [-7.77 to 4.47], Standard Error of Mean 3.12 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.019, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 3; Mean Difference (Final Values) = -7.24, 95% CI 2-sided [-13.28 to -1.19], Standard Error of Mean 3.08 — Adjusted for baseline using MMRM

10. Secondary Outcome: Frequency of Moderate to Severe Vasomotor Symptoms - Week 4 (MITT-VMS)
Description: as for outcome 1
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 134 | 144 | 142 | 152 | 126
weekly hot flushes | -40.6 (30.59) | -35.1 (29.14) | -33.6 (30.64) | -38.9 (31.04) | -26.4 (27.05)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 4; Mean Difference (Final Values) = -12.81, 95% CI 2-sided [-19.29 to -6.32], Standard Error of Mean 3.30 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.013, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 4; Mean Difference (Final Values) = -8.07, 95% CI 2-sided [-14.46 to -1.68], Standard Error of Mean 3.25 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.141, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 4; Mean Difference (Final Values) = -4.81, 95% CI 2-sided [-11.21 to 1.59], Standard Error of Mean 3.26 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 4; Mean Difference (Final Values) = -10.40, 95% CI 2-sided [-16.73 to -4.08], Standard Error of Mean 3.22 — Adjusted for baseline using MMRM

11. Secondary Outcome: Frequency of Moderate to Severe Vasomotor Symptoms - Week 5 (MITT-VMS)
Description: Mean change in frequency of moderate to severe vasomotor symptoms from Baseline to Week 5. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of moderate to severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of moderate to severe hot flushes for the subject week.
Time Frame: Baseline and Week 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 131 | 143 | 139 | 147 | 124
weekly hot flushes | -45.9 (32.31) | -39.5 (28.53) | -37.1 (30.64) | -43.5 (33.31) | -31.6 (28.96)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 5; Mean Difference (Final Values) = -15.59, 95% CI 2-sided [-22.16 to -9.02], Standard Error of Mean 3.35 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.003, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 5; Mean Difference (Final Values) = -9.88, 95% CI 2-sided [-16.34 to -3.41], Standard Error of Mean 3.29 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.075, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 5; Mean Difference (Final Values) = -5.90, 95% CI 2-sided [-12.40 to 0.59], Standard Error of Mean 3.31 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 5; Mean Difference (Final Values) = -12.05, 95% CI 2-sided [-18.47 to -5.64], Standard Error of Mean 3.27 — Adjusted for baseline using MMRM

12. Secondary Outcome: Frequency of Moderate to Severe Vasomotor Symptoms - Week 6 (MITT-VMS)
Description: Mean change in frequency of moderate to severe vasomotor symptoms from Baseline to Week 6. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of moderate to severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of moderate to severe hot flushes for the subject week.
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 132 | 143 | 139 | 146 | 123
weekly hot flushes | -49.4 (32.76) | -41.7 (29.97) | -40.1 (33.62) | -45.5 (33.14) | -32.7 (28.53)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 6; Mean Difference (Final Values) = -17.87, 95% CI 2-sided [-24.57 to -11.05], Standard Error of Mean 3.44 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 6; Mean Difference (Final Values) = -11.35, 95% CI 2-sided [-18.00 to -4.70], Standard Error of Mean 3.39 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.022, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 6; Mean Difference (Final Values) = -7.82, 95% CI 2-sided [-14.50 to -1.14], Standard Error of Mean 3.40 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 6; Mean Difference (Final Values) = -12.51, 95% CI 2-sided [-19.11 to -5.91], Standard Error of Mean 3.36 — Adjusted for baseline using MMRM

13. Secondary Outcome: Frequency of Moderate to Severe Vasomotor Symptoms - Week 7 (MITT-VMS)
Description: Mean change in frequency of moderate to severe vasomotor symptoms from Baseline to Week 7. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of moderate to severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of moderate to severe hot flushes for the subject week.
Time Frame: Baseline and Week 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 130 | 142 | 139 | 147 | 120
weekly hot flushes | -51.5 (31.51) | -45.0 (30.73) | -43.8 (33.20) | -47.7 (32.18) | -33.4 (29.37)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 7; Mean Difference (Final Values) = -17.75, 95% CI 2-sided [-24.45 to -11.06], Standard Error of Mean 3.41 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 7; Mean Difference (Final Values) = -13.29, 95% CI 2-sided [-19.88 to -6.70], Standard Error of Mean 3.36 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.003, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 7; Mean Difference (Final Values) = -10.22, 95% CI 2-sided [-16.83 to -3.60], Standard Error of Mean 3.37 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 7; Mean Difference (Final Values) = -13.61, 95% CI 2-sided [-20.15 to -7.07], Standard Error of Mean 3.33 — Adjusted for baseline using MMRM

14. Secondary Outcome: Frequency of Moderate to Severe Vasomotor Symptoms - Week 8 (MITT-VMS)
Description: Mean change in frequency of moderate to severe vasomotor symptoms from Baseline to Week 8. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of moderate to severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of moderate to severe hot flushes for the subject week.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 129 | 140 | 137 | 147 | 120
weekly hot flushes | -52.3 (31.63) | -46.8 (30.64) | -45.4 (32.55) | -48.4 (32.82) | -36.0 (30.66)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 8; Mean Difference (Final Values) = -16.63, 95% CI 2-sided [-23.35 to -9.91], Standard Error of Mean 3.42 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 8; Mean Difference (Final Values) = -12.97, 95% CI 2-sided [-19.58 to -6.36], Standard Error of Mean 3.37 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.005, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 8; Mean Difference (Final Values) = -9.63, 95% CI 2-sided [-16.27 to -2.99], Standard Error of Mean 3.38 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 8; Mean Difference (Final Values) = -11.97, 95% CI 2-sided [-18.53 to -5.41], Standard Error of Mean 3.34 — Adjusted for baseline using MMRM

15. Secondary Outcome: Frequency of Moderate to Severe Vasomotor Symptoms - Week 9 (MITT-VMS)
Description: Mean change in frequency of moderate to severe vasomotor symptoms from Baseline to Week 9. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of moderate to severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of moderate to severe hot flushes for the subject week.
Time Frame: Baseline and Week 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 137 | 132 | 141 | 119
weekly hot flushes | -52.6 (32.57) | -50.5 (31.01) | -47.4 (30.13) | -50.1 (33.92) | -36.4 (29.09)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 9; Mean Difference (Final Values) = -17.12, 95% CI 2-sided [-23.79 to -10.44], Standard Error of Mean 3.40 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 9; Mean Difference (Final Values) = -15.58, 95% CI 2-sided [-22.15 to -9.01], Standard Error of Mean 3.34 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 9; Mean Difference (Final Values) = -11.05, 95% CI 2-sided [-17.65 to -4.44], Standard Error of Mean 3.36 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 9; Mean Difference (Final Values) = -13.02, 95% CI 2-sided [-19.54 to -6.50], Standard Error of Mean 3.32 — Adjusted for baseline using MMRM

16. Secondary Outcome: Frequency of Moderate to Severe Vasomotor Symptoms - Week 10 (MITT-VMS)
Description: Mean change in frequency of moderate to severe vasomotor symptoms from Baseline to Week 10. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of moderate to severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of moderate to severe hot flushes for the subject week.
Time Frame: Baseline and Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 126 | 133 | 129 | 140 | 118
weekly hot flushes | -53.2 (32.58) | -51.9 (32.79) | -49.0 (30.24) | -50.6 (33.36) | -37.1 (29.74)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 10; Mean Difference (Final Values) = -16.80, 95% CI 2-sided [-23.58 to -10.03], Standard Error of Mean 3.45 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 10; Mean Difference (Final Values) = -15.66, 95% CI 2-sided [-22.32 to -8.99], Standard Error of Mean 3.40 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 10; Mean Difference (Final Values) = -11.20, 95% CI 2-sided [-17.90 to -4.49], Standard Error of Mean 3.41 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 10; Mean Difference (Final Values) = -12.16, 95% CI 2-sided [-18.78 to -5.55], Standard Error of Mean 3.37 — Adjusted for baseline using MMRM

17. Secondary Outcome: Frequency of Moderate to Severe Vasomotor Symptoms - Week 11 (MITT-VMS)
Description: Mean change in frequency of moderate to severe vasomotor symptoms from Baseline to Week 11. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of moderate to severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of moderate to severe hot flushes for the subject week.
Time Frame: Baseline and Week 11
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 126 | 134 | 129 | 137 | 118
weekly hot flushes | -53.7 (32.21) | -52.0 (31.24) | -49.4 (30.71) | -50.9 (34.33) | -36.7 (30.32)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 11; Mean Difference (Final Values) = -18.11, 95% CI 2-sided [-24.92 to -11.29], Standard Error of Mean 3.47 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 11; Mean Difference (Final Values) = -16.45, 95% CI 2-sided [-23.17 to -9.74], Standard Error of Mean 3.42 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 11; Mean Difference (Final Values) = -12.41, 95% CI 2-sided [-19.15 to -5.66], Standard Error of Mean 3.44 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 11; Mean Difference (Final Values) = -13.60, 95% CI 2-sided [-20.26 to -6.93], Standard Error of Mean 3.39 — Adjusted for baseline using MMRM

18. Secondary Outcome: Frequency of Moderate to Severe Vasomotor Symptoms - Week 12 (MITT-VMS)
Description: as for outcome 2
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 129 | 124 | 135 | 115
weekly hot flushes | -55.1 (31.36) | -53.7 (31.93) | -50.2 (31.35) | -52.4 (33.90) | -40.2 (29.79)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -16.58, 95% CI 2-sided [-23.33 to -9.82], Standard Error of Mean 3.44 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -15.07, 95% CI 2-sided [-21.72 to -8.42], Standard Error of Mean 3.39 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -10.79, 95% CI 2-sided [-17.48 to -4.10], Standard Error of Mean 3.41 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -11.71, 95% CI 2-sided [-18.31 to -5.11], Standard Error of Mean 3.36 — Adjusted for baseline using MMRM

19. Secondary Outcome: Severity of Moderate to Severe Vasomotor Symptoms - Week 1 (MITT-VMS)
Description: Mean change in severity of moderate to severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 1. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score = (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of moderate to severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 138 | 149 | 145 | 154 | 134
scores on a scale | -0.24 (0.305) | -0.25 (0.270) | -0.23 (0.264) | -0.25 (0.327) | -0.25 (0.257)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.801, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 1; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.06 to 0.08], Standard Error of Mean 0.034 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.991, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 1; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.07 to 0.07], Standard Error of Mean 0.034 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.642, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 1; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.05 to 0.08], Standard Error of Mean 0.034 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.928, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 1; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.07 to 0.06], Standard Error of Mean 0.034 — Adjusted for baseline using MMRM

20. Secondary Outcome: Severity of Moderate to Severe Vasomotor Symptoms - Week 2 (MITT-VMS)
Description: Mean change in severity of moderate to severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 2. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score = (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of moderate to severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 134 | 146 | 145 | 153 | 133
scores on a scale | -0.34 (0.411) | -0.34 (0.390) | -0.27 (0.354) | -0.29 (0.314) | -0.28 (0.310)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.231, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 2; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.14 to 0.03], Standard Error of Mean 0.043 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.173, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 2; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.14 to 0.03], Standard Error of Mean 0.042 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.717, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 2; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.07 to 0.10], Standard Error of Mean 0.042 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.849, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 2; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.09 to 0.07], Standard Error of Mean 0.042 — Adjusted for baseline using MMRM

21. Secondary Outcome: Severity of Moderate to Severe Vasomotor Symptoms - Week 3 (MITT-VMS)
Description: Mean change in severity of moderate to severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 3. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score = (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of moderate to severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 136 | 144 | 144 | 153 | 131
scores on a scale | -0.43 (0.514) | -0.44 (0.437) | -0.32 (0.410) | -0.37 (0.424) | -0.32 (0.372)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.039, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 3; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.21 to -0.01], Standard Error of Mean 0.052 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.030, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 3; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.21 to -0.01], Standard Error of Mean 0.052 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.946, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 3; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.10 to 0.10], Standard Error of Mean 0.052 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.309, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 3; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.15 to 0.05], Standard Error of Mean 0.051 — Adjusted for baseline using MMRM

22. Secondary Outcome: Severity of Moderate to Severe Vasomotor Symptoms - Week 4 (MITT-VMS)
Description: as for outcome 3
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 134 | 144 | 142 | 152 | 126
scores on a scale | -0.48 (0.547) | -0.51 (0.563) | -0.40 (0.469) | -0.44 (0.514) | -0.34 (0.386)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.031, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 4; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.25 to -0.01], Standard Error of Mean 0.061 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.005, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 4; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.28 to -0.05], Standard Error of Mean 0.060 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.401, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 4; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.17 to 0.07], Standard Error of Mean 0.060 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.100, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 4; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.21 to 0.02], Standard Error of Mean 0.059 — Adjusted for baseline using MMRM

23. Secondary Outcome: Severity of Moderate to Severe Vasomotor Symptoms - Week 5 (MITT-VMS)
Description: Mean change in severity of moderate to severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 5. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score = (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of moderate to severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 131 | 143 | 139 | 147 | 124
scores on a scale | -0.64 (0.702) | -0.56 (0.558) | -0.44 (0.463) | -0.53 (0.610) | -0.42 (0.551)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 5; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.37 to -0.09], Standard Error of Mean 0.071 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.034, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 5; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.28 to -0.01], Standard Error of Mean 0.070 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.790, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 5; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.16 to 0.12], Standard Error of Mean 0.070 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.086, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 5; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.25 to 0.02], Standard Error of Mean 0.069 — Adjusted for baseline using MMRM

24. Secondary Outcome: Severity of Moderate to Severe Vasomotor Symptoms - Week 6 (MITT-VMS)
Description: Mean change in severity of moderate to severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 6. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score = (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of moderate to severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 132 | 143 | 139 | 146 | 123
scores on a scale | -0.80 (0.840) | -0.61 (0.640) | -0.54 (0.578) | -0.63 (0.763) | -0.45 (0.573)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 6; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.53 to -0.20], Standard Error of Mean 0.084 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.030, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 6; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.34 to -0.02], Standard Error of Mean 0.083 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.247, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 6; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.26 to 0.07], Standard Error of Mean 0.083 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.022, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 6; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.35 to -0.03], Standard Error of Mean 0.082 — Adjusted for baseline using MMRM

25. Secondary Outcome: Severity of Moderate to Severe Vasomotor Symptoms - Week 7 (MITT-VMS)
Description: Mean change in severity of moderate to severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 7. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score = (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of moderate to severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 130 | 142 | 139 | 147 | 120
scores on a scale | -0.81 (0.793) | -0.69 (0.694) | -0.63 (0.637) | -0.64 (0.764) | -0.44 (0.483)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 7; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.54 to -0.20], Standard Error of Mean 0.085 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 7; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.42 to -0.09], Standard Error of Mean 0.083 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.031, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 7; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.34 to -0.02], Standard Error of Mean 0.084 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.016, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 7; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.36 to -0.04], Standard Error of Mean 0.083 — Adjusted for baseline using MMRM

26. Secondary Outcome: Severity of Moderate to Severe Vasomotor Symptoms - Week 8 (MITT-VMS)
Description: Mean change in severity of moderate to severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 8. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score = (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of moderate to severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 129 | 140 | 137 | 147 | 120
scores on a scale | -0.88 (0.854) | -0.70 (0.642) | -0.65 (0.685) | -0.64 (0.745) | -0.51 (0.563)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 8; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-0.55 to -0.21], Standard Error of Mean 0.087 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.008, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 8; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.40 to -0.06], Standard Error of Mean 0.086 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.087, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 8; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.32 to 0.02], Standard Error of Mean 0.086 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.092, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 8; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.31 to 0.02], Standard Error of Mean 0.085 — Adjusted for baseline using MMRM

27. Secondary Outcome: Severity of Moderate to Severe Vasomotor Symptoms - Week 9 (MITT-VMS)
Description: Mean change in severity of moderate to severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 9. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score = (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of moderate to severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 137 | 132 | 141 | 119
scores on a scale | -0.96 (0.892) | -0.74 (0.699) | -0.73 (0.720) | -0.71 (0.772) | -0.48 (0.536)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 9; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-0.66 to -0.30], Standard Error of Mean 0.092 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 9; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.47 to -0.12], Standard Error of Mean 0.090 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.009, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 9; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.42 to -0.06], Standard Error of Mean 0.091 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.007, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 9; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.42 to -0.07], Standard Error of Mean 0.090 — Adjusted for baseline using MMRM

28. Secondary Outcome: Severity of Moderate to Severe Vasomotor Symptoms - Week 10 (MITT-VMS)
Description: Mean change in severity of moderate to severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 10. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score = (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of moderate to severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 126 | 133 | 129 | 140 | 118
scores on a scale | -1.05 (0.953) | -0.77 (0.727) | -0.78 (0.769) | -0.62 (0.739) | -0.53 (0.575)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 10; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-0.71 to -0.33], Standard Error of Mean 0.096 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.003, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 10; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.46 to -0.09], Standard Error of Mean 0.094 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.016, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 10; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.41 to -0.04], Standard Error of Mean 0.095 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.310, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 10; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.28 to 0.09], Standard Error of Mean 0.094 — Adjusted for baseline using MMRM

29. Secondary Outcome: Severity of Moderate to Severe Vasomotor Symptoms - Week 11 (MITT-VMS)
Description: Mean change in severity of moderate to severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 11. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score = (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of moderate to severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 11
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 126 | 134 | 129 | 137 | 118
scores on a scale | -1.04 (0.931) | -0.86 (0.777) | -0.78 (0.782) | -0.68 (0.767) | -0.54 (0.566)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 11; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-0.72 to -0.34], Standard Error of Mean 0.098 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 11; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.56 to -0.19], Standard Error of Mean 0.096 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.011, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 11; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.44 to -0.06], Standard Error of Mean 0.097 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.076, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 11; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.36 to 0.02], Standard Error of Mean 0.096 — Adjusted for baseline using MMRM

30. Secondary Outcome: Severity of Moderate to Severe Vasomotor Symptoms - Week 12 (MITT-VMS)
Description: as for outcome 4
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 129 | 124 | 135 | 115
scores on a scale | -1.12 (0.963) | -0.90 (0.783) | -0.76 (0.744) | -0.71 (0.806) | -0.56 (0.603)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-0.77 to -0.38], Standard Error of Mean 0.100 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.59 to -0.20], Standard Error of Mean 0.099 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.018, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.43 to -0.04], Standard Error of Mean 0.100 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.096, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.36 to 0.03], Standard Error of Mean 0.098 — Adjusted for baseline using MMRM

31. Secondary Outcome: Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 1 (MITT-VMS)
Description: Mean change in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 1. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of mild, moderate and severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of mild, moderate and severe hot flushes for the subject week.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 138 | 149 | 145 | 154 | 134
weekly hot flushes | -12.9 (22.12) | -12.4 (23.94) | -12.5 (24.62) | -17.7 (27.78) | -12.2 (23.76)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.865, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 1; Mean Difference (Final Values) = 0.49, 95% CI 2-sided [-5.16 to 6.14], Standard Error of Mean 2.88 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.847, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 1; Mean Difference (Final Values) = 0.55, 95% CI 2-sided [-5.01 to 6.10], Standard Error of Mean 2.83 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.463, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 1; Mean Difference (Final Values) = 2.09, 95% CI 2-sided [-3.50 to 7.68], Standard Error of Mean 2.85 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.207, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 1; Mean Difference (Final Values) = -3.55, 95% CI 2-sided [-9.07 to 1.97], Standard Error of Mean 2.81 — Adjusted for baseline using MMRM

32. Secondary Outcome: Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 2 (MITT-VMS)
Description: Mean change in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 2. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of mild, moderate and severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of mild, moderate and severe hot flushes for the subject week.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 134 | 146 | 145 | 153 | 133
weekly hot flushes | -28.2 (29.45) | -22.4 (30.53) | -21.8 (31.66) | -27.8 (32.35) | -21.7 (27.45)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.140, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 2; Mean Difference (Final Values) = -5.07, 95% CI 2-sided [-11.80 to 1.67], Standard Error of Mean 3.43 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.982, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 2; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-6.70 to 6.55], Standard Error of Mean 3.38 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.492, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 2; Mean Difference (Final Values) = 2.33, 95% CI 2-sided [-4.32 to 8.98], Standard Error of Mean 3.39 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.216, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 2; Mean Difference (Final Values) = -4.14, 95% CI 2-sided [-10.72 to 2.43], Standard Error of Mean 3.35 — Adjusted for baseline using MMRM

33. Secondary Outcome: Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 3 (MITT-VMS)
Description: Mean change in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 3. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of mild, moderate and severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of mild, moderate and severe hot flushes for the subject week.
Time Frame: Baseline and Week 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 136 | 144 | 144 | 153 | 131
weekly hot flushes | -37.4 (32.33) | -30.7 (32.00) | -31.3 (30.79) | -35.6 (33.52) | -25.8 (30.41)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.003, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 3; Mean Difference (Final Values) = -10.38, 95% CI 2-sided [-17.26 to -3.50], Standard Error of Mean 3.50 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.277, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 3; Mean Difference (Final Values) = -3.75, 95% CI 2-sided [-10.53 to 3.02], Standard Error of Mean 3.45 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.394, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 3; Mean Difference (Final Values) = -2.95, 95% CI 2-sided [-9.75 to 3.84], Standard Error of Mean 3.46 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.022, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 3; Mean Difference (Final Values) = -7.86, 95% CI 2-sided [-14.58 to -1.15], Standard Error of Mean 3.42 — Adjusted for baseline using MMRM

34. Secondary Outcome: Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 4 (MITT-VMS)
Description: Mean change in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 4. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of mild, moderate and severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of mild, moderate and severe hot flushes for the subject week.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 134 | 144 | 142 | 152 | 126
weekly hot flushes | -44.4 (34.53) | -37.7 (35.38) | -35.4 (34.58) | -41.5 (37.40) | -26.8 (30.52)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 4; Mean Difference (Final Values) = -15.32, 95% CI 2-sided [-22.75 to -7.89], Standard Error of Mean 3.78 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.017, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 4; Mean Difference (Final Values) = -8.92, 95% CI 2-sided [-16.24 to -1.60], Standard Error of Mean 3.73 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.223, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 4; Mean Difference (Final Values) = -4.56, 95% CI 2-sided [-11.90 to 2.78], Standard Error of Mean 3.74 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 4; Mean Difference (Final Values) = -11.32, 95% CI 2-sided [-18.57 to -4.07], Standard Error of Mean 3.69 — Adjusted for baseline using MMRM

35. Secondary Outcome: Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 5 (MITT-VMS)
Description: Mean change in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 5. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of mild, moderate and severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of mild, moderate and severe hot flushes for the subject week.
Time Frame: Baseline and Week 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 131 | 143 | 139 | 147 | 124
weekly hot flushes | -49.9 (33.86) | -42.3 (34.15) | -40.1 (32.52) | -46.8 (39.88) | -33.3 (33.49)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 5; Mean Difference (Final Values) = -17.47, 95% CI 2-sided [-24.65 to -10.28], Standard Error of Mean 3.66 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.005, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 5; Mean Difference (Final Values) = -10.26, 95% CI 2-sided [-17.33 to -3.18], Standard Error of Mean 3.60 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.087, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 5; Mean Difference (Final Values) = -6.21, 95% CI 2-sided [-13.31 to 0.89], Standard Error of Mean 3.62 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 5; Mean Difference (Final Values) = -12.66, 95% CI 2-sided [-19.68 to -5.65], Standard Error of Mean 3.57 — Adjusted for baseline using MMRM

36. Secondary Outcome: Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 6 (MITT-VMS)
Description: Mean change in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 6. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of mild, moderate and severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of mild, moderate and severe hot flushes for the subject week.
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 132 | 143 | 139 | 146 | 123
weekly hot flushes | -53.9 (35.34) | -44.9 (36.12) | -43.0 (34.84) | -49.4 (40.28) | -34.1 (33.32)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 6; Mean Difference (Final Values) = -20.32, 95% CI 2-sided [-27.77 to -12.87], Standard Error of Mean 3.80 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 6; Mean Difference (Final Values) = -12.61, 95% CI 2-sided [-19.95 to -5.28], Standard Error of Mean 3.73 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.027, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 6; Mean Difference (Final Values) = -8.33, 95% CI 2-sided [-15.70 to -0.96], Standard Error of Mean 3.75 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 6; Mean Difference (Final Values) = -13.85, 95% CI 2-sided [-21.13 to -6.58], Standard Error of Mean 3.71 — Adjusted for baseline using MMRM

37. Secondary Outcome: Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 7 (MITT-VMS)
Description: Mean change in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 7. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of mild, moderate and severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of mild, moderate and severe hot flushes for the subject week.
Time Frame: Baseline and Week 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 130 | 142 | 139 | 147 | 120
weekly hot flushes | -56.1 (34.55) | -48.8 (36.92) | -47.2 (34.39) | -51.5 (39.69) | -33.4 (33.71)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 7; Mean Difference (Final Values) = -21.45, 95% CI 2-sided [-28.87 to -14.04], Standard Error of Mean 3.78 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 7; Mean Difference (Final Values) = -16.10, 95% CI 2-sided [-23.39 to -8.80], Standard Error of Mean 3.71 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 7; Mean Difference (Final Values) = -12.01, 95% CI 2-sided [-19.34 to -4.68], Standard Error of Mean 3.73 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 7; Mean Difference (Final Values) = -15.73, 95% CI 2-sided [-22.97 to -8.49], Standard Error of Mean 3.69 — Adjusted for baseline using MMRM

38. Secondary Outcome: Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 8 (MITT-VMS)
Description: Mean change in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 8. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of mild, moderate and severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of mild, moderate and severe hot flushes for the subject week.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 129 | 140 | 137 | 147 | 120
weekly hot flushes | -57.1 (35.91) | -50.6 (37.73) | -49.5 (34.34) | -52.4 (40.65) | -36.9 (35.53)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 8; Mean Difference (Final Values) = -20.52, 95% CI 2-sided [-28.06 to -12.97], Standard Error of Mean 3.84 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 8; Mean Difference (Final Values) = -15.37, 95% CI 2-sided [-22.80 to -7.95], Standard Error of Mean 3.78 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.003, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 8; Mean Difference (Final Values) = -11.49, 95% CI 2-sided [-18.95 to -4.03], Standard Error of Mean 3.80 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 8; Mean Difference (Final Values) = -13.82, 95% CI 2-sided [-21.19 to -6.46], Standard Error of Mean 3.75 — Adjusted for baseline using MMRM

39. Secondary Outcome: Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 9 (MITT-VMS)
Description: Mean change in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 9. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of mild, moderate and severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of mild, moderate and severe hot flushes for the subject week.
Time Frame: Baseline and Week 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 137 | 132 | 141 | 119
weekly hot flushes | -57.6 (36.43) | -54.7 (38.76) | -52.8 (33.68) | -54.5 (41.89) | -38.3 (35.04)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 9; Mean Difference (Final Values) = -20.34, 95% CI 2-sided [-27.93 to -12.74], Standard Error of Mean 3.87 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 9; Mean Difference (Final Values) = -17.92, 95% CI 2-sided [-25.39 to -10.45], Standard Error of Mean 3.80 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 9; Mean Difference (Final Values) = -12.97, 95% CI 2-sided [-20.49 to -5.46], Standard Error of Mean 3.82 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 9; Mean Difference (Final Values) = -14.28, 95% CI 2-sided [-21.70 to -6.87], Standard Error of Mean 3.78 — Adjusted for baseline using MMRM

40. Secondary Outcome: Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 10 (MITT-VMS)
Description: Mean change in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 10. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of mild, moderate and severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of mild, moderate and severe hot flushes for the subject week.
Time Frame: Baseline and Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 126 | 133 | 129 | 140 | 118
weekly hot flushes | -58.5 (36.86) | -56.1 (39.97) | -53.7 (34.39) | -55.7 (41.55) | -38.3 (35.52)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 10; Mean Difference (Final Values) = -21.01, 95% CI 2-sided [-28.72 to -13.29], Standard Error of Mean 3.93 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 10; Mean Difference (Final Values) = -18.37, 95% CI 2-sided [-25.96 to -10.78], Standard Error of Mean 3.87 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 10; Mean Difference (Final Values) = -13.03, 95% CI 2-sided [-20.66 to -5.39], Standard Error of Mean 3.89 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 10; Mean Difference (Final Values) = -14.65, 95% CI 2-sided [-22.19 to -7.12], Standard Error of Mean 3.84 — Adjusted for baseline using MMRM

41. Secondary Outcome: Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 11 (MITT-VMS)
Description: Mean change in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 11. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of mild, moderate and severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of mild, moderate and severe hot flushes for the subject week.
Time Frame: Baseline and Week 11
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 126 | 134 | 129 | 137 | 118
weekly hot flushes | -58.8 (36.58) | -57.0 (38.81) | -54.2 (34.38) | -56.1 (42.45) | -38.4 (35.85)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 11; Mean Difference (Final Values) = -21.83, 95% CI 2-sided [-29.57 to -14.08], Standard Error of Mean 3.94 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 11; Mean Difference (Final Values) = -19.40, 95% CI 2-sided [-27.02 to -11.77], Standard Error of Mean 3.88 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 11; Mean Difference (Final Values) = -13.98, 95% CI 2-sided [-21.65 to -6.32], Standard Error of Mean 3.90 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 11; Mean Difference (Final Values) = -15.66, 95% CI 2-sided [-23.23 to -8.10], Standard Error of Mean 3.85 — Adjusted for baseline using MMRM

42. Secondary Outcome: Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 12 (MITT-VMS)
Description: Mean change in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 12. The baseline was the most recent 7 consecutive days of data prior to randomization. The weekly frequency of mild, moderate and severe hot flushes was calculated from the daily diary record using a forward counting process of 7 day intervals beginning with the baseline date. Weekly frequency equals total number of mild, moderate and severe hot flushes for the subject week.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 129 | 124 | 135 | 115
weekly hot flushes | -60.3 (36.42) | -58.8 (39.59) | -54.8 (34.94) | -57.0 (41.71) | -41.7 (36.35)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -20.61, 95% CI 2-sided [-28.32 to -12.89], Standard Error of Mean 3.93 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -18.24, 95% CI 2-sided [-25.84 to -10.65], Standard Error of Mean 3.87 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -12.62, 95% CI 2-sided [-20.26 to -4.98], Standard Error of Mean 3.89 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -13.97, 95% CI 2-sided [-21.51 to -6.43], Standard Error of Mean 3.84 — Adjusted for baseline using MMRM

43. Secondary Outcome: Severity of Mild, Moderate and Severe Vasomotor Symptoms - Week 1 (MITT-VMS)
Description: Mean change in severity of mild, moderate and severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 1. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score =(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 138 | 149 | 145 | 154 | 134
scores on a scale | -0.06 (0.211) | -0.05 (0.206) | -0.02 (0.197) | -0.08 (0.305) | -0.07 (0.200)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.676, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 1; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.04 to 0.07], Standard Error of Mean 0.027 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.436, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 1; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.03 to 0.07], Standard Error of Mean 0.027 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.106, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 1; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.01 to 0.10], Standard Error of Mean 0.027 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.752, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 1; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.06 to 0.04], Standard Error of Mean 0.027 — Adjusted for baseline using MMRM

44. Secondary Outcome: Severity of Mild, Moderate and Severe Vasomotor Symptoms - Week 2 (MITT-VMS)
Description: Mean change in severity of mild, moderate and severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 2. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score =(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 134 | 146 | 145 | 153 | 133
scores on a scale | -0.16 (0.349) | -0.14 (0.342) | -0.06 (0.309) | -0.12 (0.288) | -0.11 (0.275)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.193, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 2; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.12 to 0.02], Standard Error of Mean 0.038 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.319, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 2; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.11 to 0.04], Standard Error of Mean 0.037 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.239, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 2; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.03 to 0.12], Standard Error of Mean 0.037 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.720, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 2; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.09 to 0.06], Standard Error of Mean 0.037 — Adjusted for baseline using MMRM

45. Secondary Outcome: Severity of Mild, Moderate and Severe Vasomotor Symptoms - Week 3 (MITT-VMS)
Description: Mean change in severity of mild, moderate and severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 3. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score =(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 136 | 144 | 144 | 153 | 131
scores on a scale | -0.25 (0.480) | -0.24 (0.402) | -0.11 (0.379) | -0.20 (0.412) | -0.15 (0.350)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.030, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 3; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.20 to -0.01], Standard Error of Mean 0.049 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.060, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 3; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.19 to 0.00], Standard Error of Mean 0.048 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.506, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 3; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.06 to 0.13], Standard Error of Mean 0.048 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.232, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 3; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.15 to 0.04], Standard Error of Mean 0.048 — Adjusted for baseline using MMRM

46. Secondary Outcome: Severity of Mild, Moderate and Severe Vasomotor Symptoms - Week 4 (MITT-VMS)
Description: Mean change in severity of mild, moderate and severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 4. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score =(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 134 | 144 | 142 | 152 | 126
scores on a scale | -0.31 (0.527) | -0.31 (0.540) | -0.19 (0.434) | -0.27 (0.507) | -0.17 (0.368)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.027, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 4; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.24 to -0.01], Standard Error of Mean 0.058 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.011, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 4; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.26 to -0.03], Standard Error of Mean 0.057 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.710, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 4; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.13 to 0.09], Standard Error of Mean 0.057 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.072, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 4; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.21 to 0.01], Standard Error of Mean 0.057 — Adjusted for baseline using MMRM

47. Secondary Outcome: Severity of Mild, Moderate and Severe Vasomotor Symptoms - Week 5 (MITT-VMS)
Description: Mean change in severity of mild, moderate and severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 5. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score =(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 131 | 143 | 139 | 147 | 124
scores on a scale | -0.46 (0.680) | -0.37 (0.546) | -0.23 (0.441) | -0.36 (0.619) | -0.24 (0.524)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 5; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.36 to -0.09], Standard Error of Mean 0.069 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.062, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 5; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.26 to 0.01], Standard Error of Mean 0.068 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.886, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 5; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.12 to 0.14], Standard Error of Mean 0.068 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.067, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 5; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.26 to 0.01], Standard Error of Mean 0.067 — Adjusted for baseline using MMRM

48. Secondary Outcome: Severity of Mild, Moderate and Severe Vasomotor Symptoms - Week 6 (MITT-VMS)
Description: Mean change in severity of mild, moderate and severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 6. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score =(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 132 | 143 | 139 | 146 | 123
scores on a scale | -0.62 (0.835) | -0.42 (0.627) | -0.33 (0.588) | -0.46 (0.775) | -0.27 (0.548)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 6; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.53 to -0.20], Standard Error of Mean 0.084 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.053, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 6; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.32 to 0.00], Standard Error of Mean 0.082 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.413, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 6; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.23 to 0.09], Standard Error of Mean 0.083 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.018, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 6; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.35 to -0.03], Standard Error of Mean 0.082 — Adjusted for baseline using MMRM

49. Secondary Outcome: Severity of Mild, Moderate and Severe Vasomotor Symptoms - Week 7 (MITT-VMS)
Description: Mean change in severity of mild, moderate and severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 7. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score =(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 130 | 142 | 139 | 147 | 120
scores on a scale | -0.65 (0.798) | -0.50 (0.687) | -0.42 (0.660) | -0.47 (0.773) | -0.27 (0.469)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 7; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.54 to -0.20], Standard Error of Mean 0.085 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.006, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 7; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.40 to -0.07], Standard Error of Mean 0.083 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.072, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 7; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.32 to 0.01], Standard Error of Mean 0.084 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.014, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 7; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.37 to -0.04], Standard Error of Mean 0.083 — Adjusted for baseline using MMRM

50. Secondary Outcome: Severity of Mild, Moderate and Severe Vasomotor Symptoms - Week 8 (MITT-VMS)
Description: Mean change in severity of mild, moderate and severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 8. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score =(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 129 | 140 | 137 | 147 | 120
scores on a scale | -0.70 (0.858) | -0.51 (0.633) | -0.44 (0.701) | -0.47 (0.750) | -0.33 (0.545)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 8; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-0.55 to -0.21], Standard Error of Mean 0.087 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.016, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 8; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.37 to -0.04], Standard Error of Mean 0.085 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.169, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 8; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.29 to 0.05], Standard Error of Mean 0.086 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.081, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 8; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.31 to 0.02], Standard Error of Mean 0.085 — Adjusted for baseline using MMRM

51. Secondary Outcome: Severity of Mild, Moderate and Severe Vasomotor Symptoms - Week 9 (MITT-VMS)
Description: Mean change in severity of mild, moderate and severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 9. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score =(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 137 | 132 | 141 | 119
scores on a scale | -0.78 (0.909) | -0.55 (0.708) | -0.51 (0.735) | -0.54 (0.780) | -0.31 (0.515)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 9; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-0.66 to -0.30], Standard Error of Mean 0.092 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.003, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 9; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.45 to -0.10], Standard Error of Mean 0.091 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.022, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 9; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.39 to -0.03], Standard Error of Mean 0.091 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.006, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 9; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.43 to -0.07], Standard Error of Mean 0.090 — Adjusted for baseline using MMRM

52. Secondary Outcome: Severity of Mild, Moderate and Severe Vasomotor Symptoms - Week 10 (MITT-VMS)
Description: Mean change in severity of mild, moderate and severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 10. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score =(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 126 | 133 | 129 | 140 | 118
scores on a scale | -0.87 (0.970) | -0.58 (0.731) | -0.57 (0.785) | -0.45 (0.754) | -0.35 (0.557)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 10; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-0.71 to -0.33], Standard Error of Mean 0.096 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.007, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 10; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.44 to -0.07], Standard Error of Mean 0.095 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.038, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 10; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.39 to -0.01], Standard Error of Mean 0.095 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.283, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 10; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.29 to 0.08], Standard Error of Mean 0.094 — Adjusted for baseline using MMRM

53. Secondary Outcome: Severity of Mild, Moderate and Severe Vasomotor Symptoms - Week 11 (MITT-VMS)
Description: Mean change in severity of mild, moderate and severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 11. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score =(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 11
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 126 | 134 | 129 | 137 | 118
scores on a scale | -0.86 (0.950) | -0.67 (0.788) | -0.56 (0.800) | -0.50 (0.776) | -0.36 (0.543)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 11; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-0.72 to -0.34], Standard Error of Mean 0.099 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 11; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.54 to -0.16], Standard Error of Mean 0.097 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.027, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 11; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.41 to -0.02], Standard Error of Mean 0.098 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.071, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 11; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.36 to 0.01], Standard Error of Mean 0.096 — Adjusted for baseline using MMRM

54. Secondary Outcome: Severity of Mild, Moderate and Severe Vasomotor Symptoms - Week 12 (MITT-VMS)
Description: Mean change in severity of mild, moderate and severe vasomotor symptoms at Baseline to mild, moderate to severe vasomotor symptoms at Week 12. The baseline was the most recent 7 consecutive days of data prior to randomization. The severity score was derived as follows: mild = 1, moderate = 2, severe = 3. Baseline Weekly Severity Score =(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days). On Treatment Weekly Severity Score = [(number of mild hot flushes for 7 days) x 1 + (number of moderate hot flushes for 7 days) x 2 + (number of severe hot flushes for 7 days) x 3] / (total number of mild, moderate and severe hot flushes over 7 days).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 129 | 124 | 135 | 115
scores on a scale | -0.94 (0.986) | -0.71 (0.784) | -0.54 (0.761) | -0.54 (0.824) | -0.39 (0.585)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-0.77 to -0.37], Standard Error of Mean 0.101 — Adjusted for baseline using MMRM
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.57 to -0.18], Standard Error of Mean 0.100 — Adjusted for baseline using MMRM
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.039, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.40 to -0.01], Standard Error of Mean 0.100 — Adjusted for baseline using MMRM
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.088, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.36 to 0.03], Standard Error of Mean 0.099 — Adjusted for baseline using MMRM

55. Secondary Outcome: Reduction of Frequency of Moderate to Severe Vasomotor Symptoms - Week 1 (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of moderate to severe VMS from Baseline to Week 1.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 137 | 149 | 145 | 154 | 134
Participants
  >=50% Reduction | 15 | 17 | 15 | 25 | 16
  >=75% Reduction | 3 | 4 | 4 | 5 | 1
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.850, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 1
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.622, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 1
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 1.000, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 1
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.374, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 1
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.706, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 1
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.372, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 1
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.316, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 1
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.221, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 1

56. Secondary Outcome: Reduction of Frequency of Moderate to Severe Vasomotor Symptoms - Week 2 (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of moderate to severe vasomotor symptoms from Baseline to Week 2.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 133 | 146 | 145 | 153 | 133
Participants
  >=50% Reduction | 44 | 35 | 34 | 49 | 35
  >=75% Reduction | 21 | 12 | 15 | 20 | 6
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.283, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 2
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.004, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 2
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.680, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 2
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.232, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 2
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.677, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 2
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.073, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 2
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.301, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 2
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.013, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 2

57. Secondary Outcome: Reduction of Frequency of Moderate to Severe Vasomotor Symptoms - Week 3 (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of moderate to severe vasomotor symptoms from Baseline to Week 3.
Time Frame: Baseline and Week 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 135 | 144 | 144 | 153 | 131
Participants
  >=50% Reduction | 68 | 59 | 54 | 71 | 42
  >=75% Reduction | 38 | 24 | 21 | 29 | 15
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.003, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 3
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 3
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.135, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 3
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.231, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 3
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.377, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 3
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.478, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 3
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.015, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 3
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.100, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 3

58. Secondary Outcome: Reduction of Frequency of Moderate to Severe Vasomotor Symptoms - Week 4 (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of moderate to severe vasomotor symptoms from Baseline to Week 4.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 133 | 144 | 142 | 152 | 126
Participants
  >=50% Reduction | 82 | 70 | 74 | 81 | 41
  >=75% Reduction | 55 | 34 | 32 | 45 | 15
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 4
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 4
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.009, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 4
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.017, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 4
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 4
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.025, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 4
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 4
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 4

59. Secondary Outcome: Reduction of Frequency of Moderate to Severe Vasomotor Symptoms - Week 5 (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of moderate to severe vasomotor symptoms from Baseline to Week 5.
Time Frame: Baseline and Week 5
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 130 | 143 | 139 | 147 | 124
Participants
  >=50% Reduction | 93 | 80 | 74 | 90 | 55
  >=75% Reduction | 55 | 47 | 38 | 54 | 27
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 5
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 5
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.066, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 5
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.055, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 5
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.174, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 5
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.319, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 5
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.007, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 5
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.008, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 5

60. Secondary Outcome: Reduction of Frequency of Moderate to Severe Vasomotor Symptoms - Week 6 (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of moderate to severe vasomotor symptoms from Baseline to Week 6.
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 131 | 143 | 139 | 146 | 123
Participants
  >=50% Reduction | 98 | 85 | 82 | 95 | 55
  >=75% Reduction | 68 | 51 | 47 | 56 | 30
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 6
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 6
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.019, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 6
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.061, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 6
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.026, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 6
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.104, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 6
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 6
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.018, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 6

61. Secondary Outcome: Reduction of Frequency of Moderate to Severe Vasomotor Symptoms - Week 7 (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of moderate to severe vasomotor symptoms from Baseline to Week 7.
Time Frame: Baseline and Week 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 129 | 142 | 139 | 147 | 120
Participants
  >=50% Reduction | 96 | 93 | 88 | 101 | 58
  >=75% Reduction | 71 | 63 | 56 | 58 | 32
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 7
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 7
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.006, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 7
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.003, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 7
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.017, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 7
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.025, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 7
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 7
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.037, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 7

62. Secondary Outcome: Reduction of Frequency of Moderate to Severe Vasomotor Symptoms - Week 8 (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of moderate to severe vasomotor symptoms from Baseline to Week 8.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 129 | 140 | 137 | 147 | 120
Participants
  >=50% Reduction | 102 | 98 | 90 | 100 | 60
  >=75% Reduction | 78 | 64 | 59 | 62 | 37
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 8
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 8
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 8
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.016, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 8
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.012, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 8
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.053, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 8
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.004, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 8
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.074, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 8

63. Secondary Outcome: Reduction of Frequency of Moderate to Severe Vasomotor Symptoms - Week 9 (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of moderate to severe vasomotor symptoms from Baseline to Week 9.
Time Frame: Baseline and Week 9
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 137 | 132 | 141 | 119
Participants
  >=50% Reduction | 98 | 107 | 92 | 101 | 63
  >=75% Reduction | 72 | 73 | 63 | 63 | 35
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 9
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 9
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 9
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 9
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.009, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 9
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.004, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 9
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.002, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 9
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.015, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 9

64. Secondary Outcome: Reduction of Frequency of Moderate to Severe Vasomotor Symptoms - Week 10 (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of moderate to severe vasomotor symptoms from Baseline to Week 10.
Time Frame: Baseline and Week 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 126 | 133 | 129 | 140 | 118
Participants
  >=50% Reduction | 95 | 102 | 100 | 101 | 68
  >=75% Reduction | 78 | 69 | 62 | 64 | 37
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.004, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 10
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 10
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.002, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 10
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 10
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 10
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.009, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 10
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.018, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 10
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.021, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 10

65. Secondary Outcome: Reduction of Frequency of Moderate to Severe Vasomotor Symptoms - Week 11 (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of moderate to severe vasomotor symptoms from Baseline to Week 11.
Time Frame: Baseline and Week 11
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 126 | 134 | 129 | 137 | 118
Participants
  >=50% Reduction | 95 | 105 | 97 | 104 | 59
  >=75% Reduction | 79 | 74 | 65 | 68 | 34
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 11
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 11
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 11
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 11
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 11
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 11
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 11
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 11

66. Secondary Outcome: Reduction of Frequency of Moderate to Severe Vasomotor Symptoms - Week 12 (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of moderate to severe vasomotor symptoms from Baseline to Week 12.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 129 | 124 | 135 | 115
Participants
  >=50% Reduction | 98 | 104 | 94 | 99 | 67
  >=75% Reduction | 84 | 75 | 66 | 68 | 37
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.006, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.015, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.005, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12

67. Secondary Outcome: Reduction of Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 1 - (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 1.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 138 | 149 | 145 | 154 | 134
Participants
  >=50% Reduction | 14 | 10 | 12 | 19 | 10
  >=75% Reduction | 2 | 2 | 1 | 4 | 1
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.523, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 1
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 1.000, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 1
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.821, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 1
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 1.000, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 1
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.828, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 1
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 1.000, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 1
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.239, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 1
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.377, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 1

68. Secondary Outcome: Reduction of Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 2 - (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 2.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 134 | 146 | 145 | 153 | 133
Participants
  >=50% Reduction | 36 | 24 | 30 | 39 | 21
  >=75% Reduction | 15 | 7 | 9 | 17 | 4
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.036, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 2
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.015, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 2
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 1.000, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 2
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.546, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 2
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.352, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 2
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.261, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 2
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.058, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 2
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.011, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 2

69. Secondary Outcome: Reduction of Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 3 - (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 3.
Time Frame: Baseline and Week 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 136 | 144 | 144 | 153 | 131
Participants
  >=50% Reduction | 63 | 49 | 50 | 61 | 33
  >=75% Reduction | 33 | 14 | 15 | 22 | 6
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 3
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 3
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.115, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 3
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.110, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 3
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.089, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 3
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.074, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 3
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.011, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 3
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.008, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 3

70. Secondary Outcome: Reduction of Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 4 - (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 4.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 134 | 144 | 142 | 152 | 126
Participants
  >=50% Reduction | 80 | 62 | 65 | 73 | 35
  >=75% Reduction | 44 | 28 | 24 | 33 | 6
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 4
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 4
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.011, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 4
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 4
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.002, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 4
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.002, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 4
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 4
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 4

71. Secondary Outcome: Reduction of Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 5 - (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 5.
Time Frame: Baseline and Week 5
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 131 | 143 | 139 | 147 | 124
Participants
  >=50% Reduction | 86 | 72 | 69 | 82 | 47
  >=75% Reduction | 48 | 34 | 27 | 37 | 13
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 5
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 5
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.048, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 5
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.006, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 5
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.063, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 5
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.058, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 5
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.004, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 5
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.003, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 5

72. Secondary Outcome: Reduction of Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 6 - (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 6.
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 132 | 143 | 139 | 146 | 123
Participants
  >=50% Reduction | 92 | 78 | 76 | 83 | 52
  >=75% Reduction | 61 | 39 | 39 | 43 | 16
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 6
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 6
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.050, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 6
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.006, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 6
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.048, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 6
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.004, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 6
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.020, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 6
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 6

73. Secondary Outcome: Reduction of Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 7 - (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 7.
Time Frame: Baseline and Week 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 130 | 142 | 139 | 147 | 120
Participants
  >=50% Reduction | 93 | 87 | 81 | 95 | 49
  >=75% Reduction | 63 | 46 | 44 | 47 | 16
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 7
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 7
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 7
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 7
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.006, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 7
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 7
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 7
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 7

74. Secondary Outcome: Reduction of Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 8 - (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 8.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 129 | 140 | 137 | 147 | 120
Participants
  >=50% Reduction | 98 | 85 | 90 | 93 | 54
  >=75% Reduction | 64 | 53 | 45 | 51 | 20
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 8
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 8
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.013, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 8
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 8
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 8
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.004, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 8
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.003, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 8
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 8

75. Secondary Outcome: Reduction of Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 9 - (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 9.
Time Frame: Baseline and Week 9
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 137 | 132 | 141 | 119
Participants
  >=50% Reduction | 95 | 95 | 91 | 94 | 58
  >=75% Reduction | 69 | 63 | 54 | 56 | 22
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 9
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 9
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 9
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 9
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 9
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 9
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.004, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 9
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 9

76. Secondary Outcome: Reduction of Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 10 - (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 10.
Time Frame: Baseline and Week 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 126 | 133 | 129 | 140 | 118
Participants
  >=50% Reduction | 93 | 94 | 92 | 93 | 54
  >=75% Reduction | 73 | 60 | 57 | 57 | 23
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 10
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 10
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 10
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 10
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 10
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 10
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p = 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 10
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 10

77. Secondary Outcome: Reduction of Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 11 - (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 11.
Time Frame: Baseline and Week 11
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 126 | 134 | 129 | 137 | 118
Participants
  >=50% Reduction | 94 | 97 | 94 | 95 | 55
  >=75% Reduction | 71 | 64 | 52 | 62 | 26
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 11
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 11
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 11
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 11
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 11
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.003, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 11
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 11
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 11

78. Secondary Outcome: Reduction of Frequency of Mild, Moderate and Severe Vasomotor Symptoms - Week 12 - (MITT-VMS)
Description: Number of Subjects with >=50%, and separately, >=75% reduction in frequency of mild, moderate and severe vasomotor symptoms from Baseline to Week 12.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 129 | 124 | 135 | 115
Participants
  >=50% Reduction | 97 | 94 | 90 | 95 | 55
  >=75% Reduction | 73 | 64 | 50 | 58 | 32
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12
Statistical Analysis 4: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; >=75% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12
Statistical Analysis 5: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12
Statistical Analysis 6: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.056, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12
Statistical Analysis 7: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=50% Reduction; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12
Statistical Analysis 8: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; >=75% Reduction; Test type: Superiority; p = 0.017, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12

79. Secondary Outcome: Clinical Global Impression (CGI) - Week 4 (MITT-VMS)
Description: The number and percentage of subjects for each possible response to the CGI at Week 4. The CGI score is a seven point scale where subjects were asked to rate the total improvement, whether or not in her judgment it was due entirely to drug treatment, compared to her condition at admission to the study. Scale: Very much improved, Much improved, Minimally improved, No change, Minimally worse, Much worse, Very much worse. Results for the top two responses (Very Much Improved and Much Improved) and No Change or Worsening (Minimally worse, Much worse, Very much worse) were combined for each group and active treatment groups compare to placebo.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 136 | 141 | 144 | 148 | 125
Participants
  (Very) Much Improved | 86 | 71 | 72 | 75 | 41
  Minimally Improved | 37 | 49 | 49 | 51 | 49
  No Change or Worse | 13 | 21 | 23 | 22 | 35
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — P-value is derived from comparing % Very Much Improved+Much Improved between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 4
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.005, Fisher Exact — P-value is derived from comparing % Very Much Improved+Much Improved between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 4
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.007, Fisher Exact — P-value is derived from comparing % Very Much Improved+Much Improved between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 4
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.004, Fisher Exact — P-value is derived from comparing % Very Much Improved+Much Improved between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 4

80. Secondary Outcome: Mean Change in Frequency of Moderate to Severe VMS for the Respective CGI Category - Week 4 (MITT-VMS)
Description: Mean change in frequency of moderate to severe vasomotor symptoms from Baseline to Week 4 for the respective CGI category. The CGI score is a seven point scale where subjects were asked to rate the total improvement, whether or not in her judgment it was due entirely to drug treatment, compared to her condition at admission to the study. Scale: Very much improved, Much improved, Minimally improved, No change, Minimally worse, Much worse, Very much worse. Results for the top two responses (Very Much Improved and Much Improved) and No Change or Worsening (Minimally worse, Much worse, Very much worse) were combined for each group and active treatment groups compare to placebo.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 136 | 141 | 144 | 148 | 125
weekly hot flushes
  (Very) Much Improved | -52.5 (27.28) | -48.6 (28.87) | -46.2 (31.23) | -55.7 (25.69) | -47.0 (24.17)
  Minimally Improved | -24.1 (23.87) | -25.9 (21.43) | -29.2 (23.26) | -28.9 (26.08) | -26.8 (17.68)
  No Change or Worse | -6.5 (23.08) | -6.6 (16.39) | -2.7 (16.22) | -5.3 (21.97) | -5.3 (13.68)

81. Secondary Outcome: Clinical Global Impression (CGI) - Week 8 (MITT-VMS)
Description: The number and percentage of subjects for each possible response to the CGI at Week 8. The CGI score is a seven point scale where subjects were asked to rate the total improvement, whether or not in her judgment it was due entirely to drug treatment, compared to her condition at admission to the study. Scale: Very much improved, Much improved, Minimally improved, No change, Minimally worse, Much worse, Very much worse. Results for the top two responses (Very Much Improved and Much Improved) and No Change or Worsening (Minimally worse, Much worse, Very much worse) were combined for each group and active treatment groups compare to placebo.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 130 | 139 | 134 | 141 | 117
Participants
  (Very) Much Improved | 101 | 103 | 98 | 93 | 62
  Minimally Improved | 23 | 24 | 23 | 35 | 25
  No Change or Worse | 6 | 12 | 13 | 13 | 30
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — P-value is derived from comparing % Very Much Improved+Much Improved between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 8
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — P-value is derived from comparing % Very Much Improved+Much Improved between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 8
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.001, Fisher Exact — P-value is derived from comparing % Very Much Improved+Much Improved between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 8
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.002, Fisher Exact — P-value is derived from comparing % Very Much Improved+Much Improved between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 8

82. Secondary Outcome: Mean Change in Frequency of Moderate to Severe VMS for the Respective CGI Category - Week 8 (MITT-VMS)
Description: Mean change in frequency of moderate to severe vasomotor symptoms from Baseline to Week 8 for the respective CGI category. The CGI score is a seven point scale where subjects were asked to rate the total improvement, whether or not in her judgment it was due entirely to drug treatment, compared to her condition at admission to the study. Scale: Very much improved, Much improved, Minimally improved, No change, Minimally worse, Much worse, Very much worse. Results for the top two responses (Very Much Improved and Much Improved) and No Change or Worsening (Minimally worse, Much worse, Very much worse) were combined for each group and active treatment groups compare to placebo.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 130 | 139 | 134 | 141 | 117
weekly hot flushes
  (Very) Much Improved | -60.8 (28.49) | -55.1 (29.27) | -55.4 (29.06) | -57.8 (30.38) | -52.6 (24.62)
  Minimally Improved | -28.7 (18.93) | -27.3 (25.22) | -27.2 (22.79) | -36.8 (24.81) | -27.0 (13.54)
  No Change or Worse | -0.2 (28.80) | -15.2 (13.41) | -1.6 (19.93) | -7.4 (21.48) | -7.1 (21.46)

83. Secondary Outcome: Clinical Global Impression (CGI) - Week 12 (MITT-VMS)
Description: The number and percentage of subjects for each possible response to the CGI at Week 12. The CGI score is a seven point scale where subjects were asked to rate the total improvement, whether or not in her judgment it was due entirely to drug treatment, compared to her condition at admission to the study. Scale: Very much improved, Much improved, Minimally improved, No change, Minimally worse, Much worse, Very much worse. Results for the top two responses (Very Much Improved and Much Improved) and No Change or Worsening (Minimally worse, Much worse, Very much worse) were combined for each group and active treatment groups compare to placebo.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 123 | 133 | 131 | 139 | 116
Participants
  (Very) Much Improved | 101 | 97 | 102 | 101 | 62
  Minimally Improved | 17 | 29 | 22 | 24 | 26
  No Change or Worse | 5 | 7 | 7 | 14 | 28
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — P-value is derived from comparing % Very Much Improved+Much Improved between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — P-value is derived from comparing % Very Much Improved+Much Improved between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — P-value is derived from comparing % Very Much Improved+Much Improved between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.002, Fisher Exact — P-value is derived from comparing % Very Much Improved+Much Improved between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12

84. Secondary Outcome: Mean Change in Frequency of Moderate to Severe VMS for the Respective CGI Category - Week 12 (MITT-VMS)
Description: Mean change in frequency of moderate to severe vasomotor symptoms from Baseline to Week 12 for the respective CGI category. The CGI score is a seven point scale where subjects were asked to rate the total improvement, whether or not in her judgment it was due entirely to drug treatment, compared to her condition at admission to the study. Scale: Very much improved, Much improved, Minimally improved, No change, Minimally worse, Much worse, Very much worse. Results for the top two responses (Very Much Improved and Much Improved) and No Change or Worsening (Minimally worse, Much worse, Very much worse) were combined for each group and active treatment groups compare to placebo.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly hot flushes
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 123 | 133 | 131 | 139 | 116
weekly hot flushes
  (Very) Much Improved | -58.8 (30.71) | -60.0 (28.37) | -58.2 (29.42) | -59.9 (28.01) | -56.2 (26.50)
  Minimally Improved | -35.9 (24.78) | -34.9 (40.36) | -28.8 (21.99) | -40.6 (37.36) | -35.7 (19.55)
  No Change or Worse | -30.7 (32.89) | -38.8 (18.99) | -8.6 (18.42) | -8.3 (31.84) | -9.2 (16.77)

85. Secondary Outcome: Number of Subjects Without Bleeding for Consecutive Cycles
Description: No bleeding was defined as the absence of bleeding. Cumulative rates for no bleeding was defined as the percentage of women who reported consecutive cycles of no bleeding for a given cycle of time.
Time Frame: Cycle 1 to 13
Population: Subjects who received study drug for at least 1 complete 28-day cycle (at least 23 days in length); subjects who reported bleeding days during a partial cycle are also included.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 278 | 299 | 304 | 268 | 90
Participants | 204 | 251 | 263 | 239 | 82
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.000, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.122, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.280, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.692, Fisher Exact

86. Secondary Outcome: Number of Subjects Without Bleeding for Consecutive Cycles
Description: as for outcome 85
Time Frame: Cycle 2 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 278 | 299 | 304 | 268 | 90
Participants | 209 | 256 | 265 | 244 | 84
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.000, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.069, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.131, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.661, Fisher Exact

87. Secondary Outcome: Number of Subjects Without Bleeding for Consecutive Cycles
Description: as for outcome 85
Time Frame: Cycle 3 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 278 | 299 | 304 | 268 | 90
Participants | 214 | 258 | 267 | 246 | 85
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.000, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.040, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.082, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.495, Fisher Exact

88. Secondary Outcome: Number of Subjects Without Bleeding for Consecutive Cycles
Description: as for outcome 85
Time Frame: Cycle 4 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 278 | 299 | 304 | 268 | 90
Participants | 217 | 261 | 273 | 253 | 86
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.000, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.032, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.137, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.792, Fisher Exact

89. Secondary Outcome: Number of Subjects Without Bleeding for Consecutive Cycles
Description: as for outcome 85
Time Frame: Cycle 5 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 278 | 299 | 304 | 268 | 90
Participants | 224 | 265 | 278 | 253 | 86
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.000, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.067, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.260, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.792, Fisher Exact

90. Secondary Outcome: Number of Subjects Without Bleeding for Consecutive Cycles
Description: as for outcome 85
Time Frame: Cycle 6 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 278 | 299 | 304 | 268 | 90
Participants | 227 | 268 | 280 | 256 | 86
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.095, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.352, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 1.000, Fisher Exact

91. Secondary Outcome: Number of Subjects Without Bleeding for Consecutive Cycles
Description: as for outcome 85
Time Frame: Cycle 7 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 278 | 299 | 304 | 268 | 90
Participants | 237 | 271 | 282 | 256 | 87
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.002, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.075, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.225, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.769, Fisher Exact

92. Secondary Outcome: Number of Subjects Without Bleeding for Consecutive Cycles
Description: as for outcome 85
Time Frame: Cycle 8 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 278 | 299 | 304 | 268 | 90
Participants | 242 | 276 | 285 | 258 | 88
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.002, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.084, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.183, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.738, Fisher Exact

93. Secondary Outcome: Number of Subjects Without Bleeding for Consecutive Cycles
Description: as for outcome 85
Time Frame: Cycle 9 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 278 | 299 | 304 | 268 | 90
Participants | 245 | 279 | 288 | 259 | 88
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.006, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.125, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.386, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.737, Fisher Exact

94. Secondary Outcome: Number of Subjects Without Bleeding for Consecutive Cycles
Description: as for outcome 85
Time Frame: Cycle 10 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 278 | 299 | 304 | 268 | 90
Participants | 248 | 281 | 292 | 261 | 88
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.009, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.183, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.745, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 1.000, Fisher Exact

95. Secondary Outcome: Number of Subjects Without Bleeding for Consecutive Cycles
Description: as for outcome 85
Time Frame: Cycle 11 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 276 | 297 | 302 | 266 | 90
Participants | 251 | 284 | 294 | 261 | 88
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.035, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.536, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 1.000, Fisher Exact

96. Secondary Outcome: Number of Subjects Without Bleeding for Consecutive Cycles
Description: as for outcome 85
Time Frame: Cycle 12 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 276 | 297 | 302 | 265 | 90
Participants | 260 | 284 | 295 | 260 | 88
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.261, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.536, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 1.000, Fisher Exact

97. Secondary Outcome: Number of Subjects Without Bleeding for Consecutive Cycles
Description: as for outcome 85
Time Frame: The 13th Cycle
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 276 | 294 | 302 | 264 | 90
Participants | 268 | 287 | 296 | 261 | 89
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.463, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.687, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 1.000, Fisher Exact

98. Secondary Outcome: Number of Subjects With Cumulative Amenorrhea From Cycle 1 to 13
Description: Cumulative amenorrhea is defined as the absence of bleeding or spotting for a cumulative period. Cumulative rates of amenorrhea were defined as the percentage of women who reported consecutive cycles of amenorrhea for a given cycle of time. Within each treatment arm, the percentage of subjects with cumulative amenorrhea from Cycle 1 to 13 was calculated and compared between active and placebo treatments.
Time Frame: Cycle 1 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 278 | 299 | 304 | 268 | 90
Participants | 156 | 202 | 207 | 196 | 71
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.048, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.049, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.328, Fisher Exact

99. Secondary Outcome: Number of Subjects With Cumulative Amenorrhea From Cycle 2 to 13
Description: Cumulative amenorrhea is defined as the absence of bleeding or spotting for a cumulative period. Cumulative rates of amenorrhea were defined as the percentage of women who reported consecutive cycles of amenorrhea for a given cycle of time. Within each treatment arm, the percentage of subjects with cumulative amenorrhea from Cycle 2 to 13 was calculated and compared between active and placebo treatments.
Time Frame: Cycle 2 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 278 | 299 | 304 | 268 | 90
Participants | 166 | 220 | 215 | 212 | 74
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.123, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.030, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.649, Fisher Exact

100. Secondary Outcome: Number of Subjects With Cumulative Amenorrhea From Cycle 3 to 13
Description: Cumulative amenorrhea is defined as the absence of bleeding or spotting for a cumulative period. Cumulative rates of amenorrhea were defined as the percentage of women who reported consecutive cycles of amenorrhea for a given cycle of time. Within each treatment arm, the percentage of subjects with cumulative amenorrhea from Cycle 3 to 13 was calculated and compared between active and placebo treatments.
Time Frame: Cycle 3 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 278 | 299 | 304 | 268 | 90
Participants | 174 | 227 | 225 | 218 | 77
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.059, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.023, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.426, Fisher Exact

101. Secondary Outcome: Number of Subjects With Cumulative Amenorrhea From Cycle 4 to 13
Description: Cumulative amenorrhea is defined as the absence of bleeding or spotting for a cumulative period. Cumulative rates of amenorrhea were defined as the percentage of women who reported consecutive cycles of amenorrhea for a given cycle of time. Within each treatment arm, the percentage of subjects with cumulative amenorrhea from Cycle 4 to 13 was calculated and compared between active and placebo treatments.
Time Frame: Cycle 4 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 278 | 299 | 304 | 268 | 90
Participants | 177 | 236 | 233 | 229 | 80
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.044, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.011, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.481, Fisher Exact

102. Secondary Outcome: Number of Subjects With Cumulative Amenorrhea From Cycle 5 to 13
Description: Cumulative amenorrhea is defined as the absence of bleeding or spotting for a cumulative period. Cumulative rates of amenorrhea were defined as the percentage of women who reported consecutive cycles of amenorrhea for a given cycle of time. Within each treatment arm, the percentage of subjects with cumulative amenorrhea from Cycle 5 to 13 was calculated and compared between active and placebo treatments.
Time Frame: Cycle 5 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 278 | 299 | 304 | 268 | 90
Participants | 183 | 244 | 240 | 234 | 80
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.110, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.045, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.853, Fisher Exact

103. Secondary Outcome: Number of Subjects With Cumulative Amenorrhea From Cycle 6 to 13
Description: Cumulative amenorrhea is defined as the absence of bleeding or spotting for a cumulative period. Cumulative rates of amenorrhea were defined as the percentage of women who reported consecutive cycles of amenorrhea for a given cycle of time. Within each treatment arm, the percentage of subjects with cumulative amenorrhea from Cycle 6 to 13 was calculated and compared between active and placebo treatments.
Time Frame: Cycle 6 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 278 | 299 | 304 | 268 | 90
Participants | 186 | 250 | 249 | 236 | 80
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.245, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.145, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 1.000, Fisher Exact

104. Secondary Outcome: Number of Subjects With Cumulative Amenorrhea From Cycle 7 to 13
Description: Cumulative amenorrhea is defined as the absence of bleeding or spotting for a cumulative period. Cumulative rates of amenorrhea were defined as the percentage of women who reported consecutive cycles of amenorrhea for a given cycle of time. Within each treatment arm, the percentage of subjects with cumulative amenorrhea from Cycle 7 to 13 was calculated and compared between active and placebo treatments.
Time Frame: Cycle 7 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 278 | 299 | 304 | 268 | 90
Participants | 200 | 253 | 255 | 238 | 82
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.163, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.091, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.693, Fisher Exact

105. Secondary Outcome: Number of Subjects With Cumulative Amenorrhea From Cycle 8 to 13
Description: Cumulative amenorrhea is defined as the absence of bleeding or spotting for a cumulative period. Cumulative rates of amenorrhea were defined as the percentage of women who reported consecutive cycles of amenorrhea for a given cycle of time. Within each treatment arm, the percentage of subjects with cumulative amenorrhea from Cycle 8 to 13 was calculated and compared between active and placebo treatments.
Time Frame: Cycle 8 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 278 | 299 | 304 | 268 | 90
Participants | 209 | 262 | 262 | 242 | 84
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.178, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.097, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.522, Fisher Exact

106. Secondary Outcome: Number of Subjects With Cumulative Amenorrhea From Cycle 9 to 13
Description: Cumulative amenorrhea is defined as the absence of bleeding or spotting for a cumulative period. Cumulative rates of amenorrhea were defined as the percentage of women who reported consecutive cycles of amenorrhea for a given cycle of time. Within each treatment arm, the percentage of subjects with cumulative amenorrhea from Cycle 9 to 13 was calculated and compared between active and placebo treatments.
Time Frame: Cycle 9 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 278 | 299 | 304 | 268 | 90
Participants | 214 | 267 | 266 | 246 | 84
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.315, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.181, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.821, Fisher Exact

107. Secondary Outcome: Number of Subjects With Cumulative Amenorrhea From Cycle 10 to 13
Description: Cumulative amenorrhea is defined as the absence of bleeding or spotting for a cumulative period. Cumulative rates of amenorrhea were defined as the percentage of women who reported consecutive cycles of amenorrhea for a given cycle of time. Within each treatment arm, the percentage of subjects with cumulative amenorrhea from Cycle 10 to 13 was calculated and compared between active and placebo treatments.
Time Frame: Cycle 10 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 278 | 299 | 304 | 268 | 90
Participants | 222 | 271 | 273 | 248 | 85
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.387, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.215, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.639, Fisher Exact

108. Secondary Outcome: Number of Subjects With Cumulative Amenorrhea From Cycle 11 to 13
Description: Cumulative amenorrhea is defined as the absence of bleeding or spotting for a cumulative period. Cumulative rates of amenorrhea were defined as the percentage of women who reported consecutive cycles of amenorrhea for a given cycle of time. Within each treatment arm, the percentage of subjects with cumulative amenorrhea from Cycle 11 to 13 was calculated and compared between active and placebo treatments.
Time Frame: Cycle 11 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 276 | 297 | 302 | 266 | 90
Participants | 231 | 275 | 277 | 249 | 85
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.008, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.643, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.501, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 1.000, Fisher Exact

109. Secondary Outcome: Number of Subjects With Cumulative Amenorrhea From Cycle 12 to 13
Description: Cumulative amenorrhea is defined as the absence of bleeding or spotting for a cumulative period. Cumulative rates of amenorrhea were defined as the percentage of women who reported consecutive cycles of amenorrhea for a given cycle of time. Within each treatment arm, the percentage of subjects with cumulative amenorrhea from Cycle 12 to 13 was calculated and compared between active and placebo treatments.
Time Frame: Cycle 12 to 13
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 276 | 297 | 302 | 265 | 90
Participants | 238 | 278 | 278 | 252 | 86
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.013, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.616, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.352, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 1.000, Fisher Exact

110. Secondary Outcome: Number of Subjects With Cumulative Amenorrhea From the 13th Cycle
Description: Cumulative amenorrhea is defined as the absence of bleeding or spotting for a cumulative period. Cumulative rates of amenorrhea were defined as the percentage of women who reported consecutive cycles of amenorrhea for a given cycle of time. Within each treatment arm, the percentage of subjects with cumulative amenorrhea from the 13th Cycle was calculated and compared between active and placebo treatments.
Time Frame: The 13th Cycle
Population: as for outcome 85
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 276 | 294 | 302 | 264 | 90
Participants | 249 | 282 | 283 | 254 | 88
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.023, Fisher Exact
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.535, Fisher Exact
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.183, Fisher Exact
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.738, Fisher Exact

111. Secondary Outcome: Subject Incidence With Spotting - Trimester 1 (Safety Pop.)
Description: Summary of subject incidence with spotting per trimester as recorded in a daily diary. A trimester is defined as every 90 days since Day 1.
Time Frame: Trimester 1
Population: Subjects who had taken at least one dose (2 capsules) of IP and had at least one bleeding/spotting diary entry for Trimester 1. Subjects who reported bleeding/spotting diary only for partial trimester are also included.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 312 | 329 | 334 | 307 | 103
Participants | 90 | 74 | 68 | 58 | 10
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo during Trimester 1
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.004, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo during Trimester 1
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.012, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo during Trimester 1
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.032, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo during Trimester 1

112. Secondary Outcome: Subject Incidence With Spotting - Trimester 2 (Safety Pop.)
Description: as for outcome 111
Time Frame: Trimester 2
Population: Subjects who had taken at least one dose (2 capsules) of IP and had at least one bleeding/spotting diary entry for Trimester 2. Subjects who reported bleeding/spotting diary only for partial trimester are also included.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 309 | 323 | 325 | 302 | 98
Participants | 76 | 40 | 48 | 24 | 4
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo during Trimester 2
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.022, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo during Trimester 2
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.004, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo during Trimester 2
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.256, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo during Trimester 2

113. Secondary Outcome: Subject Incidence With Spotting - Trimester 3 (Safety Pop.)
Description: as for outcome 111
Time Frame: Trimester 3
Population: Subjects who had taken at least one dose (2 capsules) of IP and had at least one bleeding/spotting diary entry for Trimester 3. Subjects who reported bleeding/spotting diary only for partial trimester are also included.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 298 | 311 | 320 | 288 | 97
Participants | 54 | 33 | 29 | 18 | 2
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo during Trimester 3
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.006, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo during Trimester 3
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.025, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo during Trimester 3
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.182, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo during Trimester 3

114. Secondary Outcome: Subject Incidence With Spotting - Trimester 4 (Safety Pop.)
Description: as for outcome 111
Time Frame: Trimester 4
Population: Subjects who had taken at least one dose (2 capsules) of IP and had at least one bleeding/spotting diary entry for Trimester 4. Subjects who reported bleeding/spotting diary only for partial trimester are also included.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 282 | 304 | 308 | 276 | 93
Participants | 47 | 21 | 27 | 18 | 4
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.002, Fisher Exact — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo during Trimester 4
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.469, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo during Trimester 4
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.188, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo during Trimester 4
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.613, Fisher Exact — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo during Trimester 4

115. Secondary Outcome: Number of Days With Spotting - Trimester 1 (Safety Pop.)
Description: Summary of the number of days with spotting per trimester as recorded in a daily diary. A trimester is defined as every 90 days since Day 1.
Time Frame: Trimester 1
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 312 | 329 | 334 | 307 | 103
Days | 3.0 (8.81) | 1.7 (6.05) | 1.3 (5.08) | 0.8 (2.29) | 0.6 (2.63)

116. Secondary Outcome: Number of Days With Spotting - Trimester 2 (Safety Pop.)
Description: as for outcome 115
Time Frame: Trimester 2
Population: as for outcome 112
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 309 | 323 | 325 | 302 | 98
Days | 2.9 (8.63) | 0.9 (3.85) | 1.5 (9.16) | 0.7 (4.30) | 0.1 (0.74)

117. Secondary Outcome: Number of Days With Spotting - Trimester 3 (Safety Pop.)
Description: as for outcome 115
Time Frame: Trimester 3
Population: as for outcome 113
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 298 | 311 | 320 | 288 | 97
Days | 2.5 (8.28) | 0.7 (2.55) | 0.9 (6.04) | 0.3 (1.90) | 0.0 (0.14)

118. Secondary Outcome: Number of Days With Spotting - Trimester 4 (Safety Pop.)
Description: as for outcome 115
Time Frame: Trimester 4
Population: as for outcome 114
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 282 | 304 | 308 | 276 | 93
Days | 1.9 (7.59) | 0.5 (3.36) | 0.8 (5.75) | 0.3 (1.17) | 0.1 (0.67)

119. Secondary Outcome: Subject Incidence With Bleeding - Trimester 1 (Safety Pop.)
Description: Summary of subject incidence with bleeding per trimester as recorded in a daily diary. A trimester is defined as every 90 days since Day 1.
Time Frame: Trimester 1
Population: as for outcome 111
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 312 | 329 | 334 | 307 | 103
Participants | 48 | 29 | 25 | 24 | 4
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.002, Fisher Exact — [p-value comment as in outcome 111, analysis 1]
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.135, Fisher Exact — [p-value comment as in outcome 111, analysis 2]
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.260, Fisher Exact — [p-value comment as in outcome 111, analysis 3]
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.257, Fisher Exact — [p-value comment as in outcome 111, analysis 4]

120. Secondary Outcome: Subject Incidence With Bleeding - Trimester 2 (Safety Pop.)
Description: as for outcome 119
Time Frame: Trimester 2
Population: as for outcome 112
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 309 | 323 | 325 | 302 | 98
Participants | 45 | 23 | 19 | 5 | 2
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — [p-value comment as in outcome 112, analysis 1]
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.085, Fisher Exact — [p-value comment as in outcome 112, analysis 2]
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.184, Fisher Exact — [p-value comment as in outcome 112, analysis 3]
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.681, Fisher Exact — [p-value comment as in outcome 112, analysis 4]

121. Secondary Outcome: Subject Incidence With Bleeding - Trimester 3 (Safety Pop.)
Description: as for outcome 119
Time Frame: Trimester 3
Population: as for outcome 113
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 298 | 311 | 320 | 288 | 97
Participants | 25 | 21 | 16 | 7 | 1
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.008, Fisher Exact — [p-value comment as in outcome 113, analysis 1]
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.036, Fisher Exact — [p-value comment as in outcome 113, analysis 2]
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.138, Fisher Exact — [p-value comment as in outcome 113, analysis 3]
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.685, Fisher Exact — [p-value comment as in outcome 113, analysis 4]

122. Secondary Outcome: Subject Incidence With Bleeding - Trimester 4 (Safety Pop.)
Description: as for outcome 119
Time Frame: Trimester 4
Population: as for outcome 114
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 282 | 304 | 308 | 276 | 93
Participants | 27 | 16 | 9 | 5 | 2
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.023, Fisher Exact — [p-value comment as in outcome 114, analysis 1]
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.265, Fisher Exact — [p-value comment as in outcome 114, analysis 2]
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 114, analysis 3]
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 1.000, Fisher Exact — [p-value comment as in outcome 114, analysis 4]

123. Secondary Outcome: Number of Days With Bleeding - Trimester 1 (Safety Pop.)
Description: Summary of the number of days with bleeding per trimester as recorded in a daily diary. A trimester is defined as every 90 days since Day 1.
Time Frame: Trimester 1
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 312 | 329 | 334 | 307 | 103
Days | 1.2 (5.22) | 0.5 (2.21) | 0.5 (2.24) | 0.4 (1.79) | 0.2 (1.01)

124. Secondary Outcome: Number of Days With Bleeding - Trimester 2 (Safety Pop.)
Description: as for outcome 123
Time Frame: Trimester 2
Population: as for outcome 112
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 309 | 323 | 325 | 302 | 98
Days | 0.9 (3.22) | 0.4 (1.85) | 0.4 (2.02) | 0.2 (1.77) | 0.1 (0.42)

125. Secondary Outcome: Number of Days With Bleeding - Trimester 3 (Safety Pop.)
Description: as for outcome 123
Time Frame: Trimester 3
Population: as for outcome 113
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 298 | 311 | 320 | 288 | 97
Days | 0.5 (2.32) | 0.5 (2.29) | 0.2 (1.43) | 0.1 (0.67) | 0.0 (0.10)

126. Secondary Outcome: Number of Days With Bleeding - Trimester 4 (Safety Pop.)
Description: as for outcome 123
Time Frame: Trimester 4
Population: as for outcome 114
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 282 | 304 | 308 | 276 | 93
Days | 0.8 (3.48) | 0.4 (2.06) | 0.2 (1.20) | 0.0 (0.26) | 0.1 (0.43)

127. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Vasomotor Domain Score - Week 12 (MITT-VMS)
Description: Changes in Vasomotor Domain Score from Baseline to Week 12. The MENQOL is self-administered questionnaire which assessed changes in quality of life over a one-month period. It is composed of 29 questions indicating if subject experienced the problem (Yes/No) and if Yes, rating scale ranged from 0=Not bothered at all to 6=Extremely bothered. For analysis, the original scores were converted to the analysis score ranging from 1-8 where No=1, 0=2, 1=3...and 6=8. The scale contains four domains: vasomotor, psychosocial, physical and sexual. Each domain is scored separately. Vasomotor domain score is mean of = Q1,Q2, Q3, with 1 being "not at all bothered" and 8 being "extremely bothered".
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 135 | 132 | 142 | 116
Score on a Scale | -3.8 (1.98) | -3.3 (2.04) | -3.3 (1.97) | -3.2 (2.13) | -2.2 (1.83)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -1.65, 95% CI 2-sided [-2.13 to -1.17], Standard Error of Mean 0.246
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -1.31, 95% CI 2-sided [-1.79 to -0.84], Standard Error of Mean 0.242
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -1.17, 95% CI 2-sided [-1.64 to -0.69], Standard Error of Mean 0.242
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -1.04, 95% CI 2-sided [-1.51 to -0.58], Standard Error of Mean 0.238

128. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Vasomotor Domain Score - Month 6 (MITT-VMS)
Description: Changes in Vasomotor Domain Score from Baseline to Month 6. The MENQOL is self-administered questionnaire which assessed changes in quality of life over a one-month period. It is composed of 29 questions indicating if subject experienced the problem (Yes/No) and if Yes, rating scale ranged from 0=Not bothered at all to 6=Extremely bothered. For analysis, the original scores were converted to the analysis score ranging from 1-8 where No=1, 0=2, 1=3...and 6=8. The scale contains four domains: vasomotor, psychosocial, physical and sexual. Each domain is scored separately. Vasomotor domain score is mean of = Q1,Q2, Q3, with 1 being "not at all bothered" and 8 being "extremely bothered".
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 116 | 130 | 118 | 126 | 104
score on a scale | -4.3 (1.94) | -4.1 (1.99) | -4.0 (2.12) | -3.5 (1.95) | -3.0 (2.26)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -1.40, 95% CI 2-sided [-1.91 to -0.89], Standard Error of Mean 0.258
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -1.32, 95% CI 2-sided [-1.81 to -0.82], Standard Error of Mean 0.253
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -1.12, 95% CI 2-sided [-1.63 to -0.62], Standard Error of Mean 0.257
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.007, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-1.19 to -0.19], Standard Error of Mean 0.254

129. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Vasomotor Domain Score - Month 12 (MITT-VMS)
Description: Changes in Vasomotor Domain Score from Baseline to Month 12. The MENQOL is self-administered questionnaire which assessed changes in quality of life over a one-month period. It is composed of 29 questions indicating if subject experienced the problem (Yes/No) and if Yes, rating scale ranged from 0=Not bothered at all to 6=Extremely bothered. For analysis, the original scores were converted to the analysis score ranging from 1-8 where No=1, 0=2, 1=3...and 6=8. The scale contains four domains: vasomotor, psychosocial, physical and sexual. Each domain is scored separately. Vasomotor domain score is mean of = Q1,Q2, Q3, with 1 being "not at all bothered" and 8 being "extremely bothered".
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 97 | 118 | 104 | 104 | 93
score on a scale | -4.0 (2.15) | -4.1 (1.77) | -4.0 (2.11) | -3.4 (1.75) | -2.8 (2.26)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -1.20, 95% CI 2-sided [-1.75 to -0.66], Standard Error of Mean 0.276
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -1.46, 95% CI 2-sided [-1.98 to -0.94], Standard Error of Mean 0.265
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -1.23, 95% CI 2-sided [-1.76 to -0.69], Standard Error of Mean 0.272
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.008, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-1.26 to -0.19], Standard Error of Mean 0.272

130. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Psychosocial Domain Score - Week 12 (MITT-VMS)
Description: Changes in Psychosocial Domain Score from Baseline to Week 12. The MENQOL is self-administered questionnaire which assessed changes in quality of life over a one-month period. It is composed of 29 questions indicating if subject experienced the problem (Yes/No) and if Yes, rating scale ranged from 0=Not bothered at all to 6=Extremely bothered. For analysis, the original scores were converted to the analysis score ranging from 1-8 where No=1, 0=2, 1=3...and 6=8. The scale contains four domains: vasomotor, psychosocial, physical and sexual. Each domain is scored separately. Psychosocial domain score is mean of = Q4 to Q10, with 1 being "not at all bothered" and 8 being "extremely bothered".
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 135 | 131 | 142 | 116
score on a scale | -1.1 (1.42) | -0.9 (1.56) | -1.2 (1.69) | -1.1 (1.36) | -1.0 (1.66)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.284, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.49 to 0.14], Standard Error of Mean 0.161
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.732, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.36 to 0.26], Standard Error of Mean 0.158
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.437, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.44 to 0.19], Standard Error of Mean 0.159
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.439, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.43 to 0.19], Standard Error of Mean 0.156

131. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Psychosocial Domain Score - Month 6 (MITT-VMS)
Description: Changes in Psychosocial Domain Score from Baseline to Month 6. The MENQOL is self-administered questionnaire which assessed changes in quality of life over a one-month period. It is composed of 29 questions indicating if subject experienced the problem (Yes/No) and if Yes, rating scale ranged from 0=Not bothered at all to 6=Extremely bothered. For analysis, the original scores were converted to the analysis score ranging from 1-8 where No=1, 0=2, 1=3...and 6=8. The scale contains four domains: vasomotor, psychosocial, physical and sexual. Each domain is scored separately. Psychosocial domain score is mean of = Q4 to Q10, with 1 being "not at all bothered" and 8 being "extremely bothered".
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 116 | 130 | 118 | 126 | 104
score on a scale | -1.3 (1.64) | -1.1 (1.44) | -1.1 (1.76) | -1.0 (1.57) | -1.0 (1.61)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.040, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.68 to -0.02], Standard Error of Mean 0.169
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.066, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.63 to 0.02], Standard Error of Mean 0.165
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.469, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.45 to 0.21], Standard Error of Mean 0.168
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.616, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.41 to 0.24], Standard Error of Mean 0.166

132. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Psychosocial Domain Score - Month 12 (MITT-VMS)
Description: Changes in Psychosocial Domain Score from Baseline to Month 12. The MENQOL is self-administered questionnaire which assessed changes in quality of life over a one-month period. It is composed of 29 questions indicating if subject experienced the problem (Yes/No) and if Yes, rating scale ranged from 0=Not bothered at all to 6=Extremely bothered. For analysis, the original scores were converted to the analysis score ranging from 1-8 where No=1, 0=2, 1=3...and 6=8. The scale contains four domains: vasomotor, psychosocial, physical and sexual. Each domain is scored separately. Psychosocial domain score is mean of = Q4 to Q10, with 1 being "not at all bothered" and 8 being "extremely bothered".
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 97 | 118 | 104 | 104 | 93
score on a scale | -1.1 (1.51) | -1.3 (1.61) | -1.1 (1.84) | -1.0 (1.67) | -1.0 (1.61)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.250, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.57 to 0.15], Standard Error of Mean 0.183
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-0.88 to -0.20], Standard Error of Mean 0.175
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.796, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.40 to 0.31], Standard Error of Mean 0.179
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg; Test type: Superiority; p = 0.955, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.36 to 0.34], Standard Error of Mean 0.179

133. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Physical Domain Score - Week 12 (MITT-VMS)
Description: Changes in Physical Domain Score from Baseline to Week 12. The MENQOL is self-administered questionnaire which assessed changes in quality of life over a one-month period. It is composed of 29 questions indicating if subject experienced the problem (Yes/No) and if Yes, rating scale ranged from 0=Not bothered at all to 6=Extremely bothered. For analysis, the original scores were converted to the analysis score ranging from 1-8 where No=1, 0=2, 1=3...and 6=8. The scale contains four domains: vasomotor, psychosocial, physical and sexual. Each domain is scored separately. Physical domain score is mean of = Q11 to Q26, with 1 being "not at all bothered" and 8 being "extremely bothered".
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 135 | 131 | 142 | 116
score on a scale | -1.1 (1.30) | -1.0 (1.32) | -1.5 (1.50) | -1.0 (1.30) | -1.0 (1.38)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.474, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.38 to 0.18], Standard Error of Mean 0.143
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.378, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.40 to 0.15], Standard Error of Mean 0.140
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.018, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-0.61 to -0.06], Standard Error of Mean 0.141
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.730, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.32 to 0.22], Standard Error of Mean 0.138

134. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Physical Domain Score - Month 6 (MITT-VMS)
Description: Changes in Physical Domain Score from Baseline to Month 6. The MENQOL is self-administered questionnaire which assessed changes in quality of life over a one-month period. It is composed of 29 questions indicating if subject experienced the problem (Yes/No) and if Yes, rating scale ranged from 0=Not bothered at all to 6=Extremely bothered. For analysis, the original scores were converted to the analysis score ranging from 1-8 where No=1, 0=2, 1=3...and 6=8. The scale contains four domains: vasomotor, psychosocial, physical and sexual. Each domain is scored separately. Physical domain score is mean of = Q11 to Q26, with 1 being "not at all bothered" and 8 being "extremely bothered".
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 116 | 130 | 118 | 126 | 104
score on a scale | -1.2 (1.32) | -1.1 (1.37) | -1.5 (1.61) | -1.0 (1.28) | -1.1 (1.40)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.197, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.49 to 0.10], Standard Error of Mean 0.152
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.308, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.44 to 0.14], Standard Error of Mean 0.148
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.117, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.54 to 0.06], Standard Error of Mean 0.152
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.739, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.34 to 0.24], Standard Error of Mean 0.149

135. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Physical Domain Score - Month 12 (MITT-VMS)
Description: Changes in Physical Domain Score from Baseline to Month 12. The MENQOL is self-administered questionnaire which assessed changes in quality of life over a one-month period. It is composed of 29 questions indicating if subject experienced the problem (Yes/No) and if Yes, rating scale ranged from 0=Not bothered at all to 6=Extremely bothered. For analysis, the original scores were converted to the analysis score ranging from 1-8 where No=1, 0=2, 1=3...and 6=8. The scale contains four domains: vasomotor, psychosocial, physical and sexual. Each domain is scored separately. Physical domain score is mean of = Q11 to Q26, with 1 being "not at all bothered" and 8 being "extremely bothered".
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 97 | 118 | 104 | 104 | 93
score on a scale | -1.0 (1.57) | -1.2 (1.29) | -1.4 (1.60) | -1.1 (1.44) | -0.9 (1.39)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.635, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.42 to 0.26], Standard Error of Mean 0.171
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.010, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-0.75 to -0.10], Standard Error of Mean 0.164
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.092, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.62 to 0.05], Standard Error of Mean 0.169
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.243, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.53 to 0.13], Standard Error of Mean 0.168

136. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Sexual Domain Score - Week 12 (MITT-VMS)
Description: Changes in Sexual Domain Score from Baseline to Week 12. The MENQOL is self-administered questionnaire which assessed changes in quality of life over a one-month period. It is composed of 29 questions indicating if subject experienced the problem (Yes/No) and if Yes, rating scale ranged from 0=Not bothered at all to 6=Extremely bothered. For analysis, the original scores were converted to the analysis score ranging from 1-8 where No=1, 0=2, 1=3...and 6=8. The scale contains four domains: vasomotor, psychosocial, physical and sexual. Each domain is scored separately. Sexual domain score is mean of = Q27 to Q29, with 1 being "not at all bothered" and 8 being "extremely bothered".
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 135 | 130 | 141 | 116
score on a scale | -1.5 (2.03) | -1.1 (1.98) | -1.7 (2.04) | -1.4 (2.16) | -1.3 (2.22)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.049, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.83 to -0.00], Standard Error of Mean 0.210
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.773, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.34 to 0.46], Standard Error of Mean 0.206
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.081, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.77 to 0.05], Standard Error of Mean 0.208
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.625, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.50 to 0.30], Standard Error of Mean 0.204

137. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Sexual Domain Score - Month 6 (MITT-VMS)
Description: Changes in Sexual Domain Score from Baseline to Month 6. The MENQOL is self-administered questionnaire which assessed changes in quality of life over a one-month period. It is composed of 29 questions indicating if subject experienced the problem (Yes/No) and if Yes, rating scale ranged from 0=Not bothered at all to 6=Extremely bothered. For analysis, the original scores were converted to the analysis score ranging from 1-8 where No=1, 0=2, 1=3...and 6=8. The scale contains four domains: vasomotor, psychosocial, physical and sexual. Each domain is scored separately. Sexual domain score is mean of = Q27 to Q29, with 1 being "not at all bothered" and 8 being "extremely bothered".
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 115 | 130 | 118 | 125 | 104
score on a scale | -1.3 (2.18) | -1.2 (2.03) | -1.6 (2.12) | -1.4 (2.13) | -1.3 (1.93)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.221, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.70 to 0.16], Standard Error of Mean 0.221
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.992, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.42 to 0.42], Standard Error of Mean 0.214
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.181, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.72 to 0.14], Standard Error of Mean 0.219
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.846, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.47 to 0.38], Standard Error of Mean 0.216

138. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Sexual Domain Score - Month 12 (MITT-VMS)
Description: Changes in Sexual Domain Score from Baseline to Month 12. The MENQOL is self-administered questionnaire which assessed changes in quality of life over a one-month period. It is composed of 29 questions indicating if subject experienced the problem (Yes/No) and if Yes, rating scale ranged from 0=Not bothered at all to 6=Extremely bothered. For analysis, the original scores were converted to the analysis score ranging from 1-8 where No=1, 0=2, 1=3...and 6=8. The scale contains four domains: vasomotor, psychosocial, physical and sexual. Each domain is scored separately. Sexual domain score is mean of = Q27 to Q29, with 1 being "not at all bothered" and 8 being "extremely bothered".
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 96 | 118 | 103 | 104 | 93
score on a scale | -1.0 (2.44) | -1.5 (2.20) | -1.5 (2.26) | -1.4 (2.19) | -1.1 (2.29)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.421, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.71 to 0.30], Standard Error of Mean 0.257
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.044, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-0.97 to -0.01], Standard Error of Mean 0.244
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.093, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.92 to 0.07], Standard Error of Mean 0.252
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.247, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.79 to 0.20], Standard Error of Mean 0.252

139. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Overall Scores - Week 12 (MITT-VMS)
Description: Changes in Overall Scores from Baseline to Week 12. The MENQOL is self-administered questionnaire which assessed changes in quality of life over a one-month period. It is composed of 29 questions indicating if subject experienced the problem (Yes/No) and if Yes, rating scale ranged from 0=Not bothered at all to 6=Extremely bothered. The scale contains four domains: vasomotor, psychosocial, physical and sexual. For analysis, the original scores were converted to the analysis score ranging from 1-8 where No=1, 0=2, 1=3...and 6=8. The Overall Score is the mean of the 4 domain scores with 1 being "not at all bothered" and 8 being "extremely bothered".
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 135 | 132 | 142 | 116
score on a scale | -1.9 (1.20) | -1.6 (1.23) | -1.9 (1.41) | -1.7 (1.31) | -1.4 (1.36)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-0.87 to -0.29], Standard Error of Mean 0.145
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.016, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.62 to -0.06], Standard Error of Mean 0.143
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-0.76 to -0.20], Standard Error of Mean 0.143
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.023, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.60 to -0.05], Standard Error of Mean 0.141

140. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Overall Scores - Month 6 (MITT-VMS)
Description: Changes in Overall Scores from Baseline to Month 6. The MENQOL is self-administered questionnaire which assessed changes in quality of life over a one-month period. It is composed of 29 questions indicating if subject experienced the problem (Yes/No) and if Yes, rating scale ranged from 0=Not bothered at all to 6=Extremely bothered. The scale contains four domains: vasomotor, psychosocial, physical and sexual. For analysis, the original scores were converted to the analysis score ranging from 1-8 where No=1, 0=2, 1=3...and 6=8. The Overall Score is the mean of the 4 domain scores with 1 being "not at all bothered" and 8 being "extremely bothered".
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 116 | 130 | 118 | 126 | 104
score on a scale | -2.0 (1.22) | -1.8 (1.22) | -2.1 (1.50) | -1.7 (1.24) | -1.6 (1.31)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-0.84 to -0.25], Standard Error of Mean 0.150
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.004, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.71 to -0.13], Standard Error of Mean 0.146
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.003, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-0.73 to -0.14], Standard Error of Mean 0.149
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.179, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.49 to 0.09], Standard Error of Mean 0.147

141. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Overall Scores - Month 12 (MITT-VMS)
Description: Changes in Overall Scores from Baseline to Month 12. The MENQOL is self-administered questionnaire which assessed changes in quality of life over a one-month period. It is composed of 29 questions indicating if subject experienced the problem (Yes/No) and if Yes, rating scale ranged from 0=Not bothered at all to 6=Extremely bothered. The scale contains four domains: vasomotor, psychosocial, physical and sexual. For analysis, the original scores were converted to the analysis score ranging from 1-8 where No=1, 0=2, 1=3...and 6=8. The Overall Score is the mean of the 4 domain scores with 1 being "not at all bothered" and 8 being "extremely bothered".
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 97 | 118 | 104 | 104 | 93
score on a scale | -1.8 (1.45) | -2.0 (1.27) | -2.0 (1.50) | -1.7 (1.29) | -1.5 (1.50)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.012, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-0.76 to -0.10], Standard Error of Mean 0.169
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.73, 95% CI 2-sided [-1.05 to -0.41], Standard Error of Mean 0.162
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.004, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-0.81 to -0.16], Standard Error of Mean 0.166
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.070, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.63 to 0.03], Standard Error of Mean 0.166

142. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Sleep Scale - Total Sleep Score - Week 12 (MITT-VMS)
Description: Change from Baseline to Wk 12 in MOS Total Sleep Score as compared w/Placebo. MOS-Sleep Self Report Questionnaire is 12 items that measure 6 dimensions of sleep over past 4 wks. Q1 scored on scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 self-reported hrs of sleep per night. Q3-12 scored 1-6 where 1=All of the time to 6=None of the time. Total score includes items Q1, 3, 4, 5, 6, 7, 8, 9, & 12. Scoring method: Answers to Q3, 5, 6, 7, 8, 9 are reversed & rescaled to realign to be same direction and range (0 to 100 with 0="best possible" & 100="worst possible" as follows: MOS_n_new = (6-MOS_n_old) x 20. Answers to Q1, 4, & 12 are rescaled to 0-100 as follows: MOS_1_new =(MOS_1_old - 1) x 25; MOS_4_new =(MOS_4_old - 1) x 20; MOS_12_new=(MOS_12_old - 1) x 20. Total score= average of item scores; ranges =0 to 100, where higher score means worse outcome. If any of individual questions used to obtain total score is missing, total score will be set to missing value.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 122 | 134 | 131 | 136 | 111
score on a scale | -16.7 (16.99) | -13.1 (16.22) | -18.5 (19.41) | -14.6 (18.80) | -11.5 (19.67)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.033, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -4.39, 95% CI 2-sided [-8.44 to -0.35], Standard Error of Mean 2.059
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.207, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -2.54, 95% CI 2-sided [-6.50 to 1.41], Standard Error of Mean 2.015
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.024, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -4.60, 95% CI 2-sided [-8.58 to -0.61], Standard Error of Mean 2.030
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.207, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -2.53, 95% CI 2-sided [-6.47 to 1.41], Standard Error of Mean 2.007

143. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Sleep Scale - Total Sleep Score - Month 6 (MITT-VMS)
Description: Change from Baseline to Month 6 in MOS Total Sleep Score as compared w/Placebo. MOS-Sleep Self Report Questionnaire is 12 items that measure 6 dimensions of sleep over past 4 wks. Q1 scored on scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 self-reported hrs of sleep per night. Q3-12 scored 1-6 where 1=All of the time to 6=None of the time. Total score includes items Q1, 3, 4, 5, 6, 7, 8, 9, & 12. Scoring method: Answers to Q3, 5, 6, 7, 8, 9 are reversed & rescaled to realign to be same direction and range (0 to 100 with 0="best possible" & 100="worst possible" as follows: MOS_n_new = (6-MOS_n_old) x 20. Answers to Q1, 4, & 12 are rescaled to 0-100 as follows: MOS_1_new =(MOS_1_old - 1) x 25; MOS_4_new =(MOS_4_old - 1) x 20; MOS_12_new=(MOS_12_old - 1) x 20. Total score= average of item scores; ranges =0 to 100, where higher score means worse outcome. If any of individual questions used to obtain total score is missing, total score will be set to missing value.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 113 | 124 | 118 | 123 | 101
score on a scale | -17.8 (17.28) | -16.0 (16.60) | -19.8 (21.18) | -16.6 (19.01) | -11.7 (19.40)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.011, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.48, 95% CI 2-sided [-9.68 to -1.28], Standard Error of Mean 2.138
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.012, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.25, 95% CI 2-sided [-9.36 to -1.14], Standard Error of Mean 2.093
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.009, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.58, 95% CI 2-sided [-9.75 to -1.41], Standard Error of Mean 2.122
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.018, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -4.99, 95% CI 2-sided [-9.11 to -0.87], Standard Error of Mean 2.096

144. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Sleep Scale - Total Sleep Score - Month 12 (MITT-VMS)
Description: Change from Baseline to Month 12 in MOS Total Sleep Score as compared w/Placebo. MOS-Sleep Self Report Questionnaire is 12 items that measure 6 dimensions of sleep over past 4 wks. Q1 scored on scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 self-reported hrs of sleep per night. Q3-12 scored 1-6 where 1=All of the time to 6=None of the time. Total score includes items Q1, 3, 4, 5, 6, 7, 8, 9, & 12. Scoring method: Answers to Q3, 5, 6, 7, 8, 9 are reversed & rescaled to realign to be same direction and range (0 to 100 with 0="best possible" & 100="worst possible" as follows: MOS_n_new = (6-MOS_n_old) x 20. Answers to Q1, 4, & 12 are rescaled to 0-100 as follows: MOS_1_new =(MOS_1_old - 1) x 25; MOS_4_new =(MOS_4_old - 1) x 20; MOS_12_new=(MOS_12_old - 1) x 20. Total score= average of item scores; ranges =0 to 100, where higher score means worse outcome. If any of individual questions used to obtain total score is missing, total score will be set to missing value.
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 96 | 117 | 102 | 100 | 92
score on a scale | -14.9 (21.09) | -15.8 (17.72) | -20.6 (21.58) | -17.6 (18.81) | -10.3 (21.78)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.058, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -4.61, 95% CI 2-sided [-9.38 to 0.16], Standard Error of Mean 2.427
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -7.48, 95% CI 2-sided [-12.04 to -2.92], Standard Error of Mean 2.322
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -7.96, 95% CI 2-sided [-12.67 to -3.25], Standard Error of Mean 2.397
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.005, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -6.78, 95% CI 2-sided [-11.50 to -2.06], Standard Error of Mean 2.404

145. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Disturbance - Week 12 (MITT-VMS)
Description: Change from Baseline to Wk 12 in MOS Sleep Disturbance individual score as compared with Placebo. MOS-Sleep Self Report Questionnaire is 12 items that measure 6 dimensions of sleep over past 4 wks. Q1 scored on scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 self-reported hrs of sleep per night. Q3-12 scored 1-6 where 1=All of the time to 6=None of the time. Sleep disturbance includes items Q1, Q3, Q7, Q8. Scoring method: Answer to Q1 is rescaled to 0-100 as follows: MOS_1_new =(MOS_1_old - 1) x 25. Answers to Q3, 7, 8 are reversed & rescaled to realign to be same direction and range(0 to 100 with 0="best possible" & 100="worst possible" as follows: MOS_n_new = (6-MOS_n_old) x 20. Score is average of item scores; score range=0 to 100, where higher score means worse outcome.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 135 | 132 | 142 | 116
score on a scale | -22.3 (23.72) | -17.7 (24.75) | -23.6 (25.07) | -19.3 (26.31) | -15.1 (26.65)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.020, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -6.48, 95% CI 2-sided [-11.92 to -1.04], Standard Error of Mean 2.770
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.216, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -3.36, 95% CI 2-sided [-8.69 to 1.97], Standard Error of Mean 2.715
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.033, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -5.85, 95% CI 2-sided [-11.22 to -0.48], Standard Error of Mean 2.734
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.265, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -2.99, 95% CI 2-sided [-8.27 to 2.28], Standard Error of Mean 2.685

146. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Disturbance - Month 6 - (MITT-VMS)
Description: Change from Baseline to Month 6 in MOS Sleep Disturbance individual score as compared with Placebo. MOS-Sleep Self Report Questionnaire is 12 items that measure 6 dimensions of sleep over past 4 wks. Q1 scored on scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 self-reported hrs of sleep per night. Q3-12 scored 1-6 where 1=All of the time to 6=None of the time. Sleep disturbance includes items Q1, Q3, Q7, Q8. Scoring method: Answer to Q1 is rescaled to 0-100 as follows: MOS_1_new =(MOS_1_old - 1) x 25. Answers to Q3, 7, 8 are reversed & rescaled to realign to be same direction and range(0 to 100 with 0="best possible" & 100="worst possible" as follows: MOS_n_new = (6-MOS_n_old) x 20. Score is average of item scores; score range=0 to 100, where higher score means worse outcome.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 116 | 130 | 118 | 126 | 104
score on a scale | -23.5 (25.99) | -21.3 (24.42) | -26.9 (26.91) | -22.4 (26.76) | -15.4 (27.57)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.008, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -7.54, 95% CI 2-sided [-13.14 to -1.93], Standard Error of Mean 2.854
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.016, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -6.72, 95% CI 2-sided [-12.18 to -1.26], Standard Error of Mean 2.781
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -8.69, 95% CI 2-sided [-14.28 to -3.10], Standard Error of Mean 2.847
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.028, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -6.18, 95% CI 2-sided [-11.68 to -0.68], Standard Error of Mean 2.800

147. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Disturbance - Month 12 - (MITT-VMS)
Description: Change from Baseline to Month 12 in MOS Sleep Disturbance individual score as compared with Placebo. MOS-Sleep Self Report Questionnaire is 12 items that measure 6 dimensions of sleep over past 4 wks. Q1 scored on scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 self-reported hrs of sleep per night. Q3-12 scored 1-6 where 1=All of the time to 6=None of the time. Sleep disturbance includes items Q1, Q3, Q7, Q8. Scoring method: Answer to Q1 is rescaled to 0-100 as follows: MOS_1_new =(MOS_1_old - 1) x 25. Answers to Q3, 7, 8 are reversed & rescaled to realign to be same direction and range(0 to 100 with 0="best possible" & 100="worst possible" as follows: MOS_n_new = (6-MOS_n_old) x 20. Score is average of item scores; score range=0 to 100, where higher score means worse outcome.
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 97 | 118 | 104 | 104 | 93
score on a scale | -20.0 (28.25) | -22.3 (24.84) | -26.1 (27.21) | -26.1 (25.32) | -14.1 (28.67)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.040, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -6.56, 95% CI 2-sided [-12.80 to -0.31], Standard Error of Mean 3.180
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -10.02, 95% CI 2-sided [-15.99 to -4.04], Standard Error of Mean 3.040
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -9.96, 95% CI 2-sided [-16.11 to -3.81], Standard Error of Mean 3.129
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.029, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -6.85, 95% CI 2-sided [-12.99 to -0.70], Standard Error of Mean 3.127

148. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Snoring - Week 12 - (MITT-VMS)
Description: Change from Baseline to Wk 12 in MOS Snoring individual score as compared with Placebo. The MOS-Sleep Self Report Questionnaire is composed of 12 items that measure 6 dimensions of sleep over the past 4 weeks. Q1 is scored on a scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 is self-reported hours of sleep per night. Q3-Q12 are scored 1-6 ranging from 1=All of the time to 6=None of the time. Snoring item is Q10. Scoring method: Answer to Q10 is reversed & rescaled to 0 to 100 such that 0="best possible" & 100="worst possible". MOS_n_new <- (6-MOS_n_old) x 20. Score range=0 to 100, where higher score means worse outcome.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 121 | 135 | 130 | 141 | 116
score on a scale | -0.5 (23.73) | -3.6 (25.84) | -7.1 (28.49) | -5.7 (24.65) | -5.7 (25.13)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.294, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = 3.15, 95% CI 2-sided [-2.75 to 9.05], Standard Error of Mean 3.003
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.327, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = 2.86, 95% CI 2-sided [-2.87 to 8.60], Standard Error of Mean 2.922
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.637, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -1.39, 95% CI 2-sided [-7.18 to 4.39], Standard Error of Mean 2.947
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.952, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-5.51 to 5.86], Standard Error of Mean 2.893

149. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Snoring - Month 6 - (MITT-VMS)
Description: Change from Baseline to Month 6 in MOS Snoring individual score as compared with Placebo. The MOS-Sleep Self Report Questionnaire is composed of 12 items that measure 6 dimensions of sleep over the past 4 weeks. Q1 is scored on a scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 is self-reported hours of sleep per night. Q3-Q12 are scored 1-6 ranging from 1=All of the time to 6=None of the time. Snoring item is Q10. Scoring method: Answer to Q10 is reversed & rescaled to 0 to 100 such that 0="best possible" & 100="worst possible". MOS_n_new <- (6-MOS_n_old) x 20. Score range=0 to 100, where higher score means worse outcome.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 112 | 130 | 118 | 125 | 104
score on a scale | 0.7 (26.29) | -5.5 (26.24) | -8.8 (24.47) | -6.1 (30.29) | -3.5 (27.08)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.573, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = 1.82, 95% CI 2-sided [-4.51 to 8.14], Standard Error of Mean 3.219
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.769, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.91, 95% CI 2-sided [-7.01 to 5.19], Standard Error of Mean 3.107
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.047, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -6.33, 95% CI 2-sided [-12.56 to -0.09], Standard Error of Mean 3.176
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.409, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -2.59, 95% CI 2-sided [-8.74 to 3.56], Standard Error of Mean 3.133

150. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Snoring - Month 12 - (MITT-VMS)
Description: Change from Baseline to Month 12 in MOS Snoring individual score as compared with Placebo. The MOS-Sleep Self Report Questionnaire is composed of 12 items that measure 6 dimensions of sleep over the past 4 weeks. Q1 is scored on a scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 is self-reported hours of sleep per night. Q3-Q12 are scored 1-6 ranging from 1=All of the time to 6=None of the time. Snoring item is Q10. Scoring method: Answer to Q10 is reversed & rescaled to 0 to 100 such that 0="best possible" & 100="worst possible". MOS_n_new <- (6-MOS_n_old) x 20. Score range=0 to 100, where higher score means worse outcome.
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 95 | 118 | 104 | 103 | 93
score on a scale | -1.1 (28.04) | -10.5 (29.43) | -6.2 (27.03) | -8.0 (26.77) | -4.5 (26.23)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.579, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = 1.91, 95% CI 2-sided [-4.85 to 8.67], Standard Error of Mean 3.443
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.223, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -3.99, 95% CI 2-sided [-10.43 to 2.44], Standard Error of Mean 3.275
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.542, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -2.05, 95% CI 2-sided [-8.67 to 4.56], Standard Error of Mean 3.367
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.476, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -2.41, 95% CI 2-sided [-9.04 to 4.23], Standard Error of Mean 3.376

151. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Short of Breath or Headache - Week 12 - (MITT-VMS)
Description: Change from Baseline to Wk 12 in MOS Sleep Short of Breath or Headache(SOBHA) individual score as compared with Placebo. The MOS-Sleep Self Report Questionnaire is composed of 12 items that measure 6 dimensions of sleep over the past 4 weeks. Q1 is scored on a scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 is self-reported hours of sleep per night. Q3-Q12 are scored 1-6 ranging from 1=All of the time to 6=None of the time. SOBHA item is Q5. Scoring method: Answer to Q5 is reversed & rescaled to 0 to 100 such that 0="best possible" & 100="worst possible". MOS_n_new <- (6-MOS_n_old) x 20. Score range=0 to 100, where higher score means worse outcome.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 135 | 132 | 142 | 116
score on a scale | -7.7 (26.83) | -4.3 (22.18) | -12.3 (29.62) | -7.9 (27.67) | -3.6 (25.52)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.631, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -1.25, 95% CI 2-sided [-6.34 to 3.84], Standard Error of Mean 2.593
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.651, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = 1.15, 95% CI 2-sided [-3.84 to 6.14], Standard Error of Mean 2.540
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.813, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-5.67 to 4.45], Standard Error of Mean 2.578
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.869, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-5.35 to 4.52], Standard Error of Mean 2.515

152. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Short of Breath or Headache - Month 6 - (MITT-VMS)
Description: Change from Baseline to Month 6 in MOS Sleep Short of Breath or Headache(SOBHA) individual score as compared with Placebo. The MOS-Sleep Self Report Questionnaire is composed of 12 items that measure 6 dimensions of sleep over the past 4 weeks. Q1 is scored on a scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 is self-reported hours of sleep per night. Q3-Q12 are scored 1-6 ranging from 1=All of the time to 6=None of the time. SOBHA item is Q5. Scoring method: Answer to Q5 is reversed & rescaled to 0 to 100 such that 0="best possible" & 100="worst possible". MOS_n_new <- (6-MOS_n_old) x 20. Score range=0 to 100, where higher score means worse outcome.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 116 | 129 | 118 | 126 | 104
score on a scale | -9.7 (27.72) | -5.0 (27.50) | -11.0 (33.55) | -7.3 (26.96) | -2.1 (23.47)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.074, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.00, 95% CI 2-sided [-10.48 to 0.48], Standard Error of Mean 2.790
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.748, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-6.22 to 4.47], Standard Error of Mean 2.722
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.987, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-5.46 to 5.56], Standard Error of Mean 2.805
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.709, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -1.02, 95% CI 2-sided [-6.41 to 4.36], Standard Error of Mean 2.741

153. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Short of Breath or Headache - Month 12 - (MITT-VMS)
Description: Change from Baseline to Month 12 in MOS Sleep Short of Breath or Headache(SOBHA) individual score as compared with Placebo. The MOS-Sleep Self Report Questionnaire is composed of 12 items that measure 6 dimensions of sleep over the past 4 weeks. Q1 is scored on a scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 is self-reported hours of sleep per night. Q3-Q12 are scored 1-6 ranging from 1=All of the time to 6=None of the time. SOBHA item is Q5. Scoring method: Answer to Q5 is reversed & rescaled to 0 to 100 such that 0="best possible" & 100="worst possible". MOS_n_new <- (6-MOS_n_old) x 20. Score range=0 to 100, where higher score means worse outcome.
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 97 | 118 | 103 | 104 | 93
score on a scale | -8.9 (30.41) | -7.1 (24.60) | -12.4 (34.65) | -10.8 (27.15) | -2.8 (27.60)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.379, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -2.61, 95% CI 2-sided [-8.44 to 3.22], Standard Error of Mean 2.968
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.279, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -3.07, 95% CI 2-sided [-8.64 to 2.49], Standard Error of Mean 2.832
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.894, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-6.19 to 5.40], Standard Error of Mean 2.949
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.308, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -2.98, 95% CI 2-sided [-8.72 to 2.76], Standard Error of Mean 2.923

154. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Adequacy - Week 12 - (MITT-VMS)
Description: Change from Baseline to Wk 12 in MOS Sleep Adequacy individual score as compared with Placebo. The MOS-Sleep Self Report Questionnaire is composed of 12 items that measure 6 dimensions of sleep over the past 4 weeks. Q1 is scored on a scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 is self-reported hours of sleep per night. Q3-Q12 are scored 1-6 ranging from 1=All of the time to 6=None of the time. Sleep Adequacy includes items Q4, Q12. Scoring method: Answers for Q4 and Q12 are reversed and rescaled to 0-100 as follows: MOS_4_new = (6-MOS_4_old) x 20; MOS_12_new = (6-MOS_12_old) x 20. Score is the average of item scores; score range = 0 to 100, where higher score means better outcome.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 135 | 132 | 142 | 116
score on a scale | 12.8 (28.30) | 11.0 (26.57) | 17.3 (30.06) | 10.7 (28.33) | 11.3 (26.09)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.558, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = 1.81, 95% CI 2-sided [-4.24 to 7.86], Standard Error of Mean 3.081
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.233, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = 3.61, 95% CI 2-sided [-2.34 to 9.57], Standard Error of Mean 3.031
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.043, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = 6.16, 95% CI 2-sided [0.20 to 12.13], Standard Error of Mean 3.036
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.488, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = 2.07, 95% CI 2-sided [-3.80 to 7.95], Standard Error of Mean 2.990

155. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Adequacy - Month 6 - (MITT-VMS)
Description: Change from Baseline to Month 6 in MOS Sleep Adequacy individual score as compared with Placebo. The MOS-Sleep Self Report Questionnaire is composed of 12 items that measure 6 dimensions of sleep over the past 4 weeks. Q1 is scored on a scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 is self-reported hours of sleep per night. Q3-Q12 are scored 1-6 ranging from 1=All of the time to 6=None of the time. Sleep Adequacy includes items Q4, Q12. Scoring method: Answers for Q4 and Q12 are reversed and rescaled to 0-100 as follows: MOS_4_new = (6-MOS_4_old) x 20; MOS_12_new = (6-MOS_12_old) x 20. Score is the average of item scores; score range = 0 to 100, where higher score means better outcome.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 116 | 130 | 118 | 126 | 104
score on a scale | 13.2 (28.61) | 15.2 (26.89) | 14.7 (30.12) | 15.2 (28.75) | 9.5 (27.36)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.205, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = 4.07, 95% CI 2-sided [-2.23 to 10.37], Standard Error of Mean 3.206
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = 9.58, 95% CI 2-sided [3.43 to 15.74], Standard Error of Mean 3.133
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.115, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = 5.04, 95% CI 2-sided [-1.23 to 11.32], Standard Error of Mean 3.193
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.005, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = 8.94, 95% CI 2-sided [2.75 to 15.13], Standard Error of Mean 3.152

156. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Adequacy - Month 12 - (MITT-VMS)
Description: Change from Baseline to Month 12 in MOS Sleep Adequacy individual score as compared with Placebo. The MOS-Sleep Self Report Questionnaire is composed of 12 items that measure 6 dimensions of sleep over the past 4 weeks. Q1 is scored on a scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 is self-reported hours of sleep per night. Q3-Q12 are scored 1-6 ranging from 1=All of the time to 6=None of the time. Sleep Adequacy includes items Q4, Q12. Scoring method: Answers for Q4 and Q12 are reversed and rescaled to 0-100 as follows: MOS_4_new = (6-MOS_4_old) x 20; MOS_12_new = (6-MOS_12_old) x 20. Score is the average of item scores; score range = 0 to 100, where higher score means better outcome.
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 97 | 118 | 104 | 104 | 93
score on a scale | 10.4 (28.43) | 10.5 (31.07) | 17.6 (31.61) | 13.7 (27.70) | 10.0 (31.76)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.796, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = 0.96, 95% CI 2-sided [-6.34 to 8.27], Standard Error of Mean 3.719
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.150, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = 5.14, 95% CI 2-sided [-1.87 to 12.15], Standard Error of Mean 3.568
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.019, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = 8.58, 95% CI 2-sided [1.39 to 15.77], Standard Error of Mean 3.657
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.041, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = 7.51, 95% CI 2-sided [0.30 to 14.71], Standard Error of Mean 3.667

157. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Somnolence - Week 12 - (MITT-VMS)
Description: Change from Baseline to Wk 12 in MOS Sleep Somnolence individual score as compared with Placebo. The MOS-Sleep Self Report Questionnaire is composed of 12 items that measure 6 dimensions of sleep over the past 4 weeks. Q1 is scored on a scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 is self-reported hours of sleep per night. Q3-Q12 are scored 1-6 ranging from 1=All of the time to 6=None of the time. Sleep Somnolence items include Q6, Q9, Q11. Scoring method: Answers to Q6, Q 9 and Q11 are reversed & rescaled to 0 to 100 such that 0="best possible" & 100="worst possible". MOS_n_new <- (6-MOS_n_old) x 20. Score is the average of item scores; score range range=0 to 100, where higher score means worse outcome.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 135 | 132 | 142 | 116
score on a scale | -11.3 (20.70) | -9.2 (17.82) | -10.4 (22.61) | -10.8 (21.78) | -8.7 (20.62)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.221, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -2.69, 95% CI 2-sided [-7.00 to 1.62], Standard Error of Mean 2.197
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.511, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -1.42, 95% CI 2-sided [-5.65 to 2.81], Standard Error of Mean 2.154
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.761, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = 0.66, 95% CI 2-sided [-3.60 to 4.92], Standard Error of Mean 2.168
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.332, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -2.07, 95% CI 2-sided [-6.25 to 2.11], Standard Error of Mean 2.128

158. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Somnolence - Month 6 - (MITT-VMS)
Description: Change from Baseline to Month 6 in MOS Sleep Somnolence individual score as compared with Placebo. The MOS-Sleep Self Report Questionnaire is composed of 12 items that measure 6 dimensions of sleep over the past 4 weeks. Q1 is scored on a scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 is self-reported hours of sleep per night. Q3-Q12 are scored 1-6 ranging from 1=All of the time to 6=None of the time. Sleep Somnolence items include Q6, Q9, Q11. Scoring method: Answers to Q6, Q 9 and Q11 are reversed & rescaled to 0 to 100 such that 0="best possible" & 100="worst possible". MOS_n_new <- (6-MOS_n_old) x 20. Score is the average of item scores; score range range=0 to 100, where higher score means worse outcome.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 116 | 130 | 118 | 126 | 104
score on a scale | -10.1 (21.60) | -10.8 (21.46) | -12.4 (22.98) | -10.5 (23.69) | -9.6 (21.64)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.687, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -1.00, 95% CI 2-sided [-5.86 to 3.86], Standard Error of Mean 2.474
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.373, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -2.15, 95% CI 2-sided [-6.88 to 2.58], Standard Error of Mean 2.411
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.714, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.91, 95% CI 2-sided [-5.75 to 3.94], Standard Error of Mean 2.466
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.711, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.90, 95% CI 2-sided [-5.67 to 3.87], Standard Error of Mean 2.427

159. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Somnolence - Month 12 - (MITT-VMS)
Description: Change from Baseline to Month 12 in MOS Sleep Somnolence individual score as compared with Placebo. The MOS-Sleep Self Report Questionnaire is composed of 12 items that measure 6 dimensions of sleep over the past 4 weeks. Q1 is scored on a scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 is self-reported hours of sleep per night. Q3-Q12 are scored 1-6 ranging from 1=All of the time to 6=None of the time. Sleep Somnolence items include Q6, Q9, Q11. Scoring method: Answers to Q6, Q 9 and Q11 are reversed & rescaled to 0 to 100 such that 0="best possible" & 100="worst possible". MOS_n_new <- (6-MOS_n_old) x 20. Score is the average of item scores; score range range=0 to 100, where higher score means worse outcome.
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 97 | 118 | 104 | 104 | 93
score on a scale | -8.0 (22.93) | -11.1 (21.51) | -13.1 (20.03) | -13.4 (23.82) | -6.7 (25.95)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.415, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -2.19, 95% CI 2-sided [-7.46 to 3.08], Standard Error of Mean 2.682
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.019, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -6.01, 95% CI 2-sided [-11.04 to -0.97], Standard Error of Mean 2.564
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.074, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -4.72, 95% CI 2-sided [-9.90 to 0.46], Standard Error of Mean 2.639
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.030, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -5.75, 95% CI 2-sided [-10.94 to -0.57], Standard Error of Mean 2.637

160. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Problems Index I - Week 12 - (MITT-VMS)
Description: Change from Baseline to Wk 12 in MOS Sleep Problems Index I individual score as compared with Placebo. The MOS-Sleep Self Report Questionnaire is composed of 12 items that measure 6 dimensions of sleep over the past 4 weeks. Q1 is scored on a scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 is self-reported hours of sleep per night. Q3-12 scored 1-6 where 1=All of the time to 6=None of the time. Sleep Problems Index I includes items Q4, Q5, Q7, Q8, Q9, Q12. Scoring method: Answers to Q, 5, 7, 8, 9 are reversed & rescaled to realign to be same direction and range (0 to 100 with 0="best possible" & 100="worst possible" as follows: MOS_n_new = (6-MOS_n_old) x 20. Answers to Q4, & 12 are rescaled to 0-100 as follows: MOS_4_new =(MOS_4_old - 1) x 20; MOS_12_new=(MOS_12_old - 1) x 20. Score is the average of item scores; score range range=0 to 100, where higher score means worse outcome.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 135 | 132 | 142 | 116
score on a scale | -15.2 (17.45) | -11.3 (17.04) | -17.7 (19.47) | -13.5 (19.65) | -9.9 (20.50)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.059, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -3.99, 95% CI 2-sided [-8.13 to 0.16], Standard Error of Mean 2.109
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.215, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -2.57, 95% CI 2-sided [-6.63 to 1.49], Standard Error of Mean 2.067
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.015, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -5.10, 95% CI 2-sided [-9.19 to -1.00], Standard Error of Mean 2.084
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.122, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -3.16, 95% CI 2-sided [-7.17 to 0.85], Standard Error of Mean 2.042

161. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Problems Index I - Month 6 - (MITT-VMS)
Description: Change from Baseline to Month 6 in MOS Sleep Problems Index I individual score as compared with Placebo. The MOS-Sleep Self Report Questionnaire is composed of 12 items that measure 6 dimensions of sleep over the past 4 weeks. Q1 is scored on a scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 is self-reported hours of sleep per night. Q3-12 scored 1-6 where 1=All of the time to 6=None of the time. Sleep Problems Index I includes items Q4, Q5, Q7, Q8, Q9, Q12. Scoring method: Answers to Q, 5, 7, 8, 9 are reversed & rescaled to realign to be same direction and range (0 to 100 with 0="best possible" & 100="worst possible" as follows: MOS_n_new = (6-MOS_n_old) x 20. Answers to Q4, & 12 are rescaled to 0-100 as follows: MOS_4_new =(MOS_4_old - 1) x 20; MOS_12_new=(MOS_12_old - 1) x 20. Score is the average of item scores; score range range=0 to 100, where higher score means worse outcome.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 116 | 130 | 118 | 126 | 104
score on a scale | -16.1 (16.64) | -14.3 (16.56) | -18.0 (20.71) | -15.7 (19.34) | -9.8 (20.37)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.013, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.32, 95% CI 2-sided [-9.52 to -1.13], Standard Error of Mean 2.135
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.006, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.76, 95% CI 2-sided [-9.85 to -1.68], Standard Error of Mean 2.080
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.009, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.59, 95% CI 2-sided [-9.77 to -1.40], Standard Error of Mean 2.132
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.007, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.68, 95% CI 2-sided [-9.79 to -1.57], Standard Error of Mean 2.093

162. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Problems Index I - Month 12 - (MITT-VMS)
Description: Change from Baseline to Month 12 in MOS Sleep Problems Index I individual score as compared with Placebo. The MOS-Sleep Self Report Questionnaire is composed of 12 items that measure 6 dimensions of sleep over the past 4 weeks. Q1 is scored on a scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 is self-reported hours of sleep per night. Q3-12 scored 1-6 where 1=All of the time to 6=None of the time. Sleep Problems Index I includes items Q4, Q5, Q7, Q8, Q9, Q12. Scoring method: Answers to Q, 5, 7, 8, 9 are reversed & rescaled to realign to be same direction and range (0 to 100 with 0="best possible" & 100="worst possible" as follows: MOS_n_new = (6-MOS_n_old) x 20. Answers to Q4, & 12 are rescaled to 0-100 as follows: MOS_4_new =(MOS_4_old - 1) x 20; MOS_12_new=(MOS_12_old - 1) x 20. Score is the average of item scores; score range range=0 to 100, where higher score means worse outcome.
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 97 | 118 | 104 | 104 | 93
score on a scale | -13.3 (20.52) | -13.5 (18.04) | -18.9 (21.49) | -16.1 (20.01) | -9.1 (22.62)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.171, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -3.39, 95% CI 2-sided [-8.24 to 1.47], Standard Error of Mean 2.470
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.006, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -6.49, 95% CI 2-sided [-11.14 to -1.85], Standard Error of Mean 2.364
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.003, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -7.39, 95% CI 2-sided [-12.17 to -2.61], Standard Error of Mean 2.434
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.006, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -6.69, 95% CI 2-sided [-11.46 to -1.92], Standard Error of Mean 2.429

163. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Problems Index II - Week 12 - (MITT-VMS)
Description: Change from Baseline to Wk 12 in MOS Sleep Problems Index II individual score as compared with Placebo. The MOS-Sleep Self Report Questionnaire is composed of 12 items that measure 6 dimensions of sleep over the past 4 weeks. Q1 is scored on a scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 is self reported hours of sleep per night. Q3-12 scored 1-6 where 1=All of the time to 6=None of the time. Sleep Problems Index II items include Q1, Q3, Q4, Q5, Q6, Q7, Q8, Q9, Q12. Scoring method: Answers to Q3, 5, 6, 7, 8, & 9 are reversed & rescaled to realign to be same direction and range 0 to 100 with 0="best possible" & 100="worst possible" as follows: MOS_n_new = (6-MOS_n_old) x 20, for n=Q3, 5, 6, 7, 8, and 9. Answers to Q1, 4 & 12 are rescaled to 0-100 as follows: MOS_1_new =(MOS_1_old - 1) x 25; MOS_4_new =(MOS_4_old - 1) x 20; MOS_12_new=(MOS_12_old - 1) x 20. Score is the average of item scores; score range range=0 to 100, where higher score means worse outcome.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 124 | 135 | 132 | 142 | 116
score on a scale | -16.8 (17.14) | -13.1 (16.16) | -18.5 (19.34) | -14.4 (19.19) | -11.8 (19.56)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.039, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -4.21, 95% CI 2-sided [-8.21 to -0.21], Standard Error of Mean 2.037
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.232, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -2.39, 95% CI 2-sided [-6.31 to 1.53], Standard Error of Mean 1.997
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.030, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -4.37, 95% CI 2-sided [-8.32 to -0.42], Standard Error of Mean 2.012
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.262, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -2.22, 95% CI 2-sided [-6.09 to 1.66], Standard Error of Mean 1.973

164. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Problems Index II - Month 6 - (MITT-VMS)
Description: Change from Baseline to Month 6 in MOS Sleep Problems Index II individual score as compared with Placebo. The MOS-Sleep Self Report Questionnaire is composed of 12 items that measure 6 dimensions of sleep over the past 4 weeks. Q1 is scored on a scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 is self reported hours of sleep per night. Q3-12 scored 1-6 where 1=All of the time to 6=None of the time. Sleep Problems Index II items include Q1, Q3, Q4, Q5, Q6, Q7, Q8, Q9, Q12. Scoring method: Answers to Q3, 5, 6, 7, 8, & 9 are reversed & rescaled to realign to be same direction and range 0 to 100 with 0="best possible" & 100="worst possible" as follows: MOS_n_new = (6-MOS_n_old) x 20, for n=Q3, 5, 6, 7, 8, and 9. Answers to Q1, 4 & 12 are rescaled to 0-100 as follows: MOS_1_new =(MOS_1_old - 1) x 25; MOS_4_new =(MOS_4_old - 1) x 20; MOS_12_new=(MOS_12_old - 1) x 20. Score is the average of item scores; score range range=0 to 100, where higher score means worse outcome.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 116 | 130 | 118 | 126 | 104
score on a scale | -17.5 (17.40) | -16.0 (16.69) | -19.8 (21.18) | -17.0 (19.02) | -11.6 (19.31)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.011, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.41, 95% CI 2-sided [-9.57 to -1.25], Standard Error of Mean 2.119
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.008, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.54, 95% CI 2-sided [-9.60 to -1.48], Standard Error of Mean 2.065
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.007, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.74, 95% CI 2-sided [-9.90 to -1.59], Standard Error of Mean 2.115
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.011, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.32, 95% CI 2-sided [-9.40 to -1.24], Standard Error of Mean 2.078

165. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Problems Index II - Month 12 - (MITT-VMS)
Description: Change from Baseline to Month 12 in MOS Sleep Problems Index II individual score as compared with Placebo. The MOS-Sleep Self Report Questionnaire is composed of 12 items that measure 6 dimensions of sleep over the past 4 weeks. Q1 is scored on a scale 1-5: 1=0-15 min, 2=16-30 min...5=>60 mins. Q2 is self reported hours of sleep per night. Q3-12 scored 1-6 where 1=All of the time to 6=None of the time. Sleep Problems Index II items include Q1, Q3, Q4, Q5, Q6, Q7, Q8, Q9, Q12. Scoring method: Answers to Q3, 5, 6, 7, 8, & 9 are reversed & rescaled to realign to be same direction and range 0 to 100 with 0="best possible" & 100="worst possible" as follows: MOS_n_new = (6-MOS_n_old) x 20, for n=Q3, 5, 6, 7, 8, and 9. Answers to Q1, 4 & 12 are rescaled to 0-100 as follows: MOS_1_new =(MOS_1_old - 1) x 25; MOS_4_new =(MOS_4_old - 1) x 20; MOS_12_new=(MOS_12_old - 1) x 20. Score is the average of item scores; score range range=0 to 100, where higher score means worse outcome.
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 97 | 118 | 104 | 104 | 93
score on a scale | -14.7 (21.13) | -15.7 (17.65) | -20.5 (21.49) | -17.4 (19.48) | -10.5 (21.71)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.083, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -4.21, 95% CI 2-sided [-8.96 to 0.55], Standard Error of Mean 2.421
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -7.36, 95% CI 2-sided [-11.91 to -2.81], Standard Error of Mean 2.317
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -7.92, 95% CI 2-sided [-12.60 to -3.23], Standard Error of Mean 2.384
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.005, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -6.78, 95% CI 2-sided [-11.46 to -2.10], Standard Error of Mean 2.381

166. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Optimal Sleep - Week 12 - (MITT-VMS)
Description: Change from Baseline (BL) to Week 12 in MOS Optimal Sleep Score as compared with Placebo. The MOS-Sleep Self Report Questionnaire is composed of 12 items measuring 6 dimensions of sleep over the past 4 wks. Optimal sleep is based on Q2 (self-reported average hrs sleep per night in past 4 wks). Scoring method: hrs of sleep coded 0 (non-optimal) or 1 (optimal) where 1-6 hrs & 9-23 hrs = 0, 7-8 hrs = 1. Change from BL: subject sleeps 7-8 hrs at BL & 1-6 or 9-23 hrs at follow-up, change = -1; subject sleeps 1-6 or 9-23 hrs at BL & 7-8 hrs at follow-up, change = +1; subject sleeps 1-6 or 9-23 hrs at BL & 1-6 or 9-23 hrs at follow-up, change = 0. Mean change from BL: changes are summed to give the Net Total (equivalent to the number subjects w/ improved sleep hrs minus the number subjects w/ worsened sleep hrs), which is divided by the number of subjects to give the mean proportion of net change, where >0 = overall improvement and <0 = overall worsening in the study arm.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Proportion of Net Change
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 123 | 134 | 132 | 142 | 115
Proportion of Net Change | 0.2 (0.55) | 0.2 (0.54) | 0.2 (0.45) | 0.2 (0.53) | 0.2 (0.58)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.938, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.12 to 0.11], Standard Error of Mean 0.060
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.779, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.10 to 0.13], Standard Error of Mean 0.059
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.646, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.14 to 0.09], Standard Error of Mean 0.059
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.421, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.07 to 0.16], Standard Error of Mean 0.058

167. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Optimal Sleep - Month 6 - (MITT-VMS)
Description: Change from Baseline (BL) to Month 6 in MOS Optimal Sleep Score as compared with Placebo. The MOS-Sleep Self Report Questionnaire is composed of 12 items measuring 6 dimensions of sleep over the past 4 wks. Optimal sleep is based on Q2 (self-reported average hrs sleep per night in past 4 wks). Scoring method: hrs of sleep coded 0 (non-optimal) or 1 (optimal) where 1-6 hrs & 9-23 hrs = 0, 7-8 hrs = 1. Change from BL: subject sleeps 7-8 hrs at BL & 1-6 or 9-23 hrs at follow-up, change = -1; subject sleeps 1-6 or 9-23 hrs at BL & 7-8 hrs at follow-up, change = +1; subject sleeps 1-6 or 9-23 hrs at BL & 1-6 or 9-23 hrs at follow-up, change = 0. Mean change from BL: changes are summed to give the Net Total (equivalent to the number subjects w/ improved sleep hrs minus the number subjects w/ worsened sleep hrs), which is divided by the number of subjects to give the mean proportion of net change, where >0 = overall improvement and <0 = overall worsening in the study arm.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Proportion of Net Change
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 115 | 129 | 118 | 125 | 104
Proportion of Net Change | 0.3 (0.52) | 0.2 (0.52) | 0.2 (0.57) | 0.1 (0.57) | 0.2 (0.52)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.075, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.01 to 0.24], Standard Error of Mean 0.063
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.074, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.01 to 0.23], Standard Error of Mean 0.062
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.370, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.07 to 0.18], Standard Error of Mean 0.063
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.851, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.11 to 0.13], Standard Error of Mean 0.062

168. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Optimal Sleep - Month 12 - (MITT-VMS)
Description: Change from Baseline (BL) to Month 12 in MOS Optimal Sleep Score as compared with Placebo. The MOS-Sleep Self Report Questionnaire is composed of 12 items measuring 6 dimensions of sleep over the past 4 wks. Optimal sleep is based on Q2 (self-reported average hrs sleep per night in past 4 wks). Scoring method: hrs of sleep coded 0 (non-optimal) or 1 (optimal) where 1-6 hrs & 9-23 hrs = 0, 7-8 hrs = 1. Change from BL: subject sleeps 7-8 hrs at BL & 1-6 or 9-23 hrs at follow-up, change = -1; subject sleeps 1-6 or 9-23 hrs at BL & 7-8 hrs at follow-up, change = +1; subject sleeps 1-6 or 9-23 hrs at BL & 1-6 or 9-23 hrs at follow-up, change = 0. Mean change from BL: changes are summed to give the Net Total (equivalent to the number subjects w/ improved sleep hrs minus the number subjects w/ worsened sleep hrs), which is divided by the number of subjects to give the mean proportion of net change, where >0 = overall improvement and <0 = overall worsening in the study arm.
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Proportion of Net Change
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 96 | 117 | 104 | 104 | 93
Proportion of Net Change | 0.2 (0.47) | 0.3 (0.58) | 0.1 (0.57) | 0.1 (0.51) | 0.2 (0.47)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.452, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.18 to 0.08], Standard Error of Mean 0.067
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.244, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.05 to 0.20], Standard Error of Mean 0.064
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.354, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.19 to 0.07], Standard Error of Mean 0.065
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.527, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.17 to 0.09], Standard Error of Mean 0.065

169. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Vasomotor Domain Score - Week 12 (MITT)
Description: as for outcome 127
Time Frame: Baseline and Week 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 354 | 364 | 375 | 376 | 117
score on a scale | -3.5 (2.02) | -3.1 (2.00) | -3.1 (2.01) | -2.9 (1.94) | -2.2 (1.84)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -1.92, 95% CI 2-sided [-2.29 to -1.55], Standard Error of Mean 0.190
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -1.44, 95% CI 2-sided [-1.81 to -1.07], Standard Error of Mean 0.189
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -1.44, 95% CI 2-sided [-1.81 to -1.07], Standard Error of Mean 0.189
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -1.25, 95% CI 2-sided [-1.62 to -0.88], Standard Error of Mean 0.188

170. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Vasomotor Domain Score - Month 6 (MITT)
Description: as for outcome 128
Time Frame: Baseline and Month 6
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 316 | 333 | 342 | 324 | 104
score on a scale | -4.0 (1.95) | -3.7 (2.02) | -3.5 (2.15) | -3.3 (1.94) | -3.0 (2.26)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -1.73, 95% CI 2-sided [-2.12 to -1.34], Standard Error of Mean 0.199
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -1.29, 95% CI 2-sided [-1.68 to -0.91], Standard Error of Mean 0.197
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -1.20, 95% CI 2-sided [-1.58 to -0.81], Standard Error of Mean 0.197
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-1.34 to -0.57], Standard Error of Mean 0.198

171. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Vasomotor Domain Score - Month 12 (MITT)
Description: as for outcome 129
Time Frame: Baseline and Month 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 283 | 304 | 312 | 280 | 93
score on a scale | -3.8 (2.05) | -3.7 (1.89) | -3.4 (2.06) | -3.3 (1.80) | -2.8 (2.26)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -1.65, 95% CI 2-sided [-2.06 to -1.25], Standard Error of Mean 0.207
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -1.47, 95% CI 2-sided [-1.87 to -1.07], Standard Error of Mean 0.204
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -1.30, 95% CI 2-sided [-1.70 to -0.90], Standard Error of Mean 0.205
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -1.08, 95% CI 2-sided [-1.48 to -0.67], Standard Error of Mean 0.207

172. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Psychosocial Domain Score - Week 12 (MITT)
Description: as for outcome 130
Time Frame: Baseline and Week 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 354 | 363 | 373 | 376 | 117
score on a scale | -1.1 (1.52) | -1.0 (1.66) | -1.1 (1.58) | -1.0 (1.49) | -1.0 (1.68)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.126, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.46 to 0.06], Standard Error of Mean 0.131
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.200, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.42 to 0.09], Standard Error of Mean 0.130
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.222, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.41 to 0.10], Standard Error of Mean 0.130
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.358, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.37 to 0.14], Standard Error of Mean 0.130

173. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Psychosocial Domain Score - Month 6 (MITT)
Description: as for outcome 131
Time Frame: Baseline and Month 6
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 316 | 330 | 343 | 324 | 104
score on a scale | -1.3 (1.68) | -1.1 (1.65) | -1.1 (1.65) | -1.0 (1.55) | -1.0 (1.61)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.023, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.59 to -0.04], Standard Error of Mean 0.138
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.045, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.55 to -0.01], Standard Error of Mean 0.138
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.384, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.39 to 0.15], Standard Error of Mean 0.137
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.424, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.38 to 0.16], Standard Error of Mean 0.138

174. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Psychosocial Domain Score - Month 12 (MITT)
Description: as for outcome 132
Time Frame: Baseline and Month 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 282 | 303 | 312 | 280 | 93
score on a scale | -1.1 (1.65) | -1.1 (1.74) | -1.1 (1.66) | -1.0 (1.64) | -1.0 (1.61)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.153, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.52 to 0.08], Standard Error of Mean 0.152
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.058, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.58 to 0.01], Standard Error of Mean 0.151
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.550, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.39 to 0.21], Standard Error of Mean 0.151
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.854, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.33 to 0.27], Standard Error of Mean 0.153

175. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Physical Domain Score - Week 12 (MITT)
Description: as for outcome 133
Time Frame: Baseline and Week 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 354 | 364 | 374 | 376 | 117
score on a scale | -1.1 (1.41) | -1.1 (1.44) | -1.3 (1.40) | -1.1 (1.39) | -1.0 (1.38)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.181, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.38 to 0.07], Standard Error of Mean 0.116
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.108, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.41 to 0.04], Standard Error of Mean 0.116
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.014, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.51 to -0.06], Standard Error of Mean 0.115
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.323, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.34 to 0.11], Standard Error of Mean 0.115

176. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Physical Domain Score - Month 6 (MITT)
Description: as for outcome 134
Time Frame: Baseline and Month 6
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 316 | 332 | 343 | 324 | 104
score on a scale | -1.2 (1.42) | -1.1 (1.46) | -1.2 (1.46) | -1.0 (1.39) | -1.1 (1.40)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.056, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.48 to 0.01], Standard Error of Mean 0.124
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.279, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.38 to 0.11], Standard Error of Mean 0.124
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.435, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.34 to 0.15], Standard Error of Mean 0.123
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.607, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.31 to 0.18], Standard Error of Mean 0.124

177. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Physical Domain Score - Month 12 (MITT)
Description: as for outcome 135
Time Frame: Baseline and Month 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 282 | 304 | 312 | 280 | 93
score on a scale | -1.1 (1.52) | -1.1 (1.48) | -1.2 (1.43) | -1.1 (1.50) | -0.9 (1.39)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.060, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.53 to 0.01], Standard Error of Mean 0.138
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.026, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.57 to -0.04], Standard Error of Mean 0.137
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.097, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.49 to 0.04], Standard Error of Mean 0.136
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.230, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.44 to 0.10], Standard Error of Mean 0.138

178. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Sexual Domain Score - Week 12 (MITT)
Description: as for outcome 136
Time Frame: Baseline and Week 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 352 | 364 | 371 | 375 | 117
score on a scale | -1.4 (2.06) | -1.3 (2.21) | -1.5 (2.02) | -1.5 (2.15) | -1.3 (2.21)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.107, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.61 to 0.06], Standard Error of Mean 0.170
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.302, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.51 to 0.16], Standard Error of Mean 0.169
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.106, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.60 to 0.06], Standard Error of Mean 0.169
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.156, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.57 to 0.09], Standard Error of Mean 0.169

179. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Sexual Domain Score - Month 6 (MITT)
Description: as for outcome 137
Time Frame: Baseline and Month 6
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 315 | 332 | 342 | 322 | 104
score on a scale | -1.4 (2.11) | -1.4 (2.12) | -1.4 (2.05) | -1.3 (2.10) | -1.3 (1.93)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.081, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.65 to 0.04], Standard Error of Mean 0.177
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.212, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.56 to 0.12], Standard Error of Mean 0.175
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.345, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.51 to 0.18], Standard Error of Mean 0.175
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.829, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.38 to 0.31], Standard Error of Mean 0.176

180. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Sexual Domain Score - Month 12 (MITT)
Description: as for outcome 138
Time Frame: Baseline and Month 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 281 | 304 | 310 | 278 | 93
score on a scale | -1.3 (2.26) | -1.4 (2.32) | -1.3 (2.10) | -1.2 (2.25) | -1.1 (2.29)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.029, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-0.84 to -0.05], Standard Error of Mean 0.201
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.026, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-0.84 to -0.05], Standard Error of Mean 0.199
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.093, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-0.72 to 0.06], Standard Error of Mean 0.199
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.223, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.64 to 0.15], Standard Error of Mean 0.202

181. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Overall Scores - Week 12 (MITT)
Description: Change in Overall Scores from Baseline to Week 12. The MENQOL is self-administered questionnaire which assessed changes in quality of life over a one-month period. It is composed of 29 questions indicating if subject experienced the problem (Yes/No) and if Yes, rating scale ranged from 0=Not bothered at all to 6=Extremely bothered. The scale contains four domains: vasomotor, psychosocial, physical and sexual. For analysis, the original scores were converted to the analysis score ranging from 1-8 where No=1, 0=2, 1=3...and 6=8. The Overall Score is the mean of the 4 domain scores with 1 being "not at all bothered" and 8 being "extremely bothered".
Time Frame: Baseline and Week 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 354 | 364 | 375 | 376 | 117
score on a scale | -1.8 (1.31) | -1.6 (1.38) | -1.7 (1.35) | -1.6 (1.35) | -1.4 (1.36)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-0.85 to -0.40], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-0.71 to -0.26], Standard Error of Mean 0.11
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-0.75 to -0.30], Standard Error of Mean 0.11
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.64 to -0.20], Standard Error of Mean 0.11

182. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Overall Scores - Month 6 (MITT)
Description: Change in Overall Scores from Baseline to Month 6. The MENQOL is self-administered questionnaire which assessed changes in quality of life over a one-month period. It is composed of 29 questions indicating if subject experienced the problem (Yes/No) and if Yes, rating scale ranged from 0=Not bothered at all to 6=Extremely bothered. The scale contains four domains: vasomotor, psychosocial, physical and sexual. For analysis, the original scores were converted to the analysis score ranging from 1-8 where No=1, 0=2, 1=3...and 6=8. The Overall Score is the mean of the 4 domain scores with 1 being "not at all bothered" and 8 being "extremely bothered".
Time Frame: Baseline and Month 6
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 316 | 333 | 343 | 324 | 104
score on a scale | -2.0 (1.32) | -1.8 (1.38) | -1.8 (1.39) | -1.7 (1.29) | -1.6 (1.31)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-0.85 to -0.38], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-0.69 to -0.22], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.003, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.59 to -0.12], Standard Error of Mean 0.12
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.030, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.50 to -0.03], Standard Error of Mean 0.12

183. Secondary Outcome: Menopause-specific Quality of Life Questionnaire (MENQOL) - Overall Scores - Month 12 (MITT)
Description: Change in Overall Scores from Baseline to Month 12. The MENQOL is self-administered questionnaire which assessed changes in quality of life over a one-month period. It is composed of 29 questions indicating if subject experienced the problem (Yes/No) and if Yes, rating scale ranged from 0=Not bothered at all to 6=Extremely bothered. The scale contains four domains: vasomotor, psychosocial, physical and sexual. For analysis, the original scores were converted to the analysis score ranging from 1-8 where No=1, 0=2, 1=3...and 6=8. The Overall Score is the mean of the 4 domain scores with 1 being "not at all bothered" and 8 being "extremely bothered".
Time Frame: Baseline and Month 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 283 | 304 | 312 | 280 | 93
score on a scale | -1.8 (1.43) | -1.8 (1.45) | -1.7 (1.38) | -1.6 (1.38) | -1.5 (1.50)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-0.89 to -0.36], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-0.88 to -0.36], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.73 to -0.21], Standard Error of Mean 0.13
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.006, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.63 to -0.10], Standard Error of Mean 0.13

184. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Sleep Scale - Total Sleep Score - Week 12 (MITT)
Description: as for outcome 142
Time Frame: Baseline and Week 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 350 | 358 | 370 | 365 | 112
score on a scale | -15.1 (17.64) | -13.0 (17.42) | -13.9 (17.40) | -13.3 (18.22) | -11.5 (19.60)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.003, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -4.88, 95% CI 2-sided [-8.08 to -1.69], Standard Error of Mean 1.629
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.027, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -3.61, 95% CI 2-sided [-6.80 to -0.42], Standard Error of Mean 1.626
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.034, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -3.44, 95% CI 2-sided [-6.61 to -0.26], Standard Error of Mean 1.618
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.119, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -2.53, 95% CI 2-sided [-5.71 to 0.65], Standard Error of Mean 1.621

185. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Sleep Scale - Total Sleep Score - Month 6 (MITT)
Description: as for outcome 143
Time Frame: Baseline and Month 6
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 313 | 321 | 339 | 317 | 101
score on a scale | -15.6 (18.13) | -14.8 (16.10) | -14.7 (18.95) | -14.6 (18.93) | -11.7 (19.40)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.39, 95% CI 2-sided [-8.73 to -2.05], Standard Error of Mean 1.700
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.39, 95% CI 2-sided [-8.72 to -2.06], Standard Error of Mean 1.696
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.004, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -4.88, 95% CI 2-sided [-8.19 to -1.58], Standard Error of Mean 1.685
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.009, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -4.42, 95% CI 2-sided [-7.75 to -1.09], Standard Error of Mean 1.698

186. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Sleep Scale - Total Sleep Score - Month 12 (MITT)
Description: as for outcome 144
Time Frame: Baseline and Month 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 281 | 300 | 308 | 270 | 92
score on a scale | -14.4 (18.36) | -14.5 (17.85) | -15.3 (18.78) | -15.3 (19.28) | -10.3 (21.78)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -6.54, 95% CI 2-sided [-10.18 to -2.90], Standard Error of Mean 1.855
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -7.61, 95% CI 2-sided [-11.23 to -4.00], Standard Error of Mean 1.843
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -7.44, 95% CI 2-sided [-11.04 to -3.84], Standard Error of Mean 1.835
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -6.76, 95% CI 2-sided [-10.41 to -3.10], Standard Error of Mean 1.863

187. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Disturbance - Week 12 - (MITT)
Description: as for outcome 145
Time Frame: Baseline and Week 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 354 | 365 | 374 | 376 | 117
score on a scale | -21.0 (23.74) | -18.1 (24.62) | -18.7 (23.11) | -17.3 (24.88) | -14.9 (26.57)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -7.34, 95% CI 2-sided [-11.55 to -3.13], Standard Error of Mean 2.146
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.009, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -5.60, 95% CI 2-sided [-9.80 to -1.40], Standard Error of Mean 2.139
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.016, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -5.13, 95% CI 2-sided [-9.31 to -0.95], Standard Error of Mean 2.132
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.154, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -3.04, 95% CI 2-sided [-7.22 to 1.14], Standard Error of Mean 2.130

188. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Disturbance - Month 6 - (MITT)
Description: as for outcome 146
Time Frame: Baseline and Month 6
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 317 | 333 | 343 | 324 | 104
score on a scale | -22.3 (25.24) | -20.2 (22.46) | -20.1 (25.12) | -19.4 (24.85) | -15.4 (27.57)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -8.38, 95% CI 2-sided [-12.72 to -4.04], Standard Error of Mean 2.213
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -7.52, 95% CI 2-sided [-11.83 to -3.20], Standard Error of Mean 2.201
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -7.32, 95% CI 2-sided [-11.63 to -3.02], Standard Error of Mean 2.193
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.011, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.60, 95% CI 2-sided [-9.93 to -1.27], Standard Error of Mean 2.207

189. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Disturbance - Month 12 - (MITT)
Description: as for outcome 147
Time Frame: Baseline and Month 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 283 | 305 | 312 | 280 | 93
score on a scale | -20.2 (25.27) | -19.9 (24.90) | -19.9 (25.01) | -19.7 (24.13) | -14.1 (28.67)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -8.97, 95% CI 2-sided [-13.76 to -4.19], Standard Error of Mean 2.439
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -9.60, 95% CI 2-sided [-14.34 to -4.85], Standard Error of Mean 2.420
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -9.30, 95% CI 2-sided [-14.03 to -4.56], Standard Error of Mean 2.412
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -7.72, 95% CI 2-sided [-12.51 to -2.93], Standard Error of Mean 2.442

190. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Snoring - Week 12 - (MITT)
Description: as for outcome 148
Time Frame: Baseline and Week 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 351 | 364 | 371 | 375 | 117
score on a scale | -2.6 (25.30) | -4.7 (26.08) | -4.5 (28.93) | -3.4 (26.94) | -5.6 (25.03)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.434, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = 2.02, 95% CI 2-sided [-3.03 to 7.07], Standard Error of Mean 2.576
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.442, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = 1.97, 95% CI 2-sided [-3.06 to 7.00], Standard Error of Mean 2.564
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.558, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = 1.50, 95% CI 2-sided [-3.52 to 6.51], Standard Error of Mean 2.558
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.534, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = 1.59, 95% CI 2-sided [-3.42 to 6.60], Standard Error of Mean 2.555

191. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Snoring - Month 6 - (MITT)
Description: as for outcome 149
Time Frame: Baseline and Month 6
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 312 | 332 | 340 | 323 | 104
score on a scale | -2.4 (28.00) | -6.0 (25.73) | -6.8 (27.32) | -3.7 (28.98) | -3.5 (27.08)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.927, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-5.08 to 5.58], Standard Error of Mean 2.719
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.541, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -1.65, 95% CI 2-sided [-6.95 to 3.64], Standard Error of Mean 2.699
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.171, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -3.68, 95% CI 2-sided [-8.96 to 1.60], Standard Error of Mean 2.691
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.667, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -1.17, 95% CI 2-sided [-6.48 to 4.15], Standard Error of Mean 2.708

192. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Snoring - Month 12 - (MITT)
Description: as for outcome 150
Time Frame: Baseline and Month 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 280 | 305 | 311 | 277 | 93
score on a scale | -3.4 (29.62) | -7.5 (27.71) | -5.0 (28.57) | -4.5 (24.79) | -4.5 (26.23)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.662, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = 1.25, 95% CI 2-sided [-4.36 to 6.87], Standard Error of Mean 2.863
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.635, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -1.35, 95% CI 2-sided [-6.91 to 4.21], Standard Error of Mean 2.834
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.877, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-5.98 to 5.11], Standard Error of Mean 2.827
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.893, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-6.01 to 5.24], Standard Error of Mean 2.867

193. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Short of Breath or Headache - Week 12 - (MITT)
Description: as for outcome 151
Time Frame: Baseline and Week 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 354 | 364 | 374 | 376 | 117
score on a scale | -6.0 (24.56) | -6.0 (23.67) | -7.1 (27.97) | -6.3 (27.03) | -3.4 (25.50)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.830, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-4.48 to 3.59], Standard Error of Mean 2.058
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.755, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-4.66 to 3.38], Standard Error of Mean 2.050
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.802, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [-3.50 to 4.53], Standard Error of Mean 2.046
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.823, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-4.46 to 3.55], Standard Error of Mean 2.043

194. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Short of Breath or Headache - Month 6 - (MITT)
Description: as for outcome 152
Time Frame: Baseline and Month 6
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 317 | 332 | 343 | 324 | 104
score on a scale | -6.2 (28.14) | -5.9 (24.36) | -7.5 (27.19) | -5.7 (26.34) | -2.1 (23.47)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.255, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -2.46, 95% CI 2-sided [-6.71 to 1.78], Standard Error of Mean 2.166
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.293, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -2.27, 95% CI 2-sided [-6.49 to 1.96], Standard Error of Mean 2.154
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.502, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -1.44, 95% CI 2-sided [-5.66 to 2.77], Standard Error of Mean 2.148
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.495, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -1.47, 95% CI 2-sided [-5.71 to 2.76], Standard Error of Mean 2.161

195. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Short of Breath or Headache - Month 12 - (MITT)
Description: as for outcome 153
Time Frame: Baseline and Month 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 283 | 305 | 311 | 280 | 93
score on a scale | -6.6 (27.64) | -6.4 (23.58) | -7.9 (28.34) | -6.5 (28.07) | -2.8 (27.60)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.389, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -1.96, 95% CI 2-sided [-6.42 to 2.50], Standard Error of Mean 2.274
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.281, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -2.43, 95% CI 2-sided [-6.85 to 1.99], Standard Error of Mean 2.253
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.504, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -1.51, 95% CI 2-sided [-5.92 to 2.91], Standard Error of Mean 2.250
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.460, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -1.68, 95% CI 2-sided [-6.15 to 2.78], Standard Error of Mean 2.277

196. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Adequacy - Week 12 - (MITT)
Description: as for outcome 154
Time Frame: Baseline and Week 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 354 | 365 | 374 | 376 | 117
score on a scale | 11.9 (29.12) | 9.0 (27.40) | 11.4 (27.54) | 11.9 (27.30) | 11.3 (25.98)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.084, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = 4.35, 95% CI 2-sided [-0.58 to 9.28], Standard Error of Mean 2.513
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.298, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = 2.61, 95% CI 2-sided [-2.30 to 7.53], Standard Error of Mean 2.506
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.136, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = 3.72, 95% CI 2-sided [-1.17 to 8.62], Standard Error of Mean 2.496
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.163, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = 3.48, 95% CI 2-sided [-1.41 to 8.37], Standard Error of Mean 2.492

197. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Adequacy - Month 6 - (MITT)
Description: as for outcome 155
Time Frame: Baseline and Month 6
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 317 | 333 | 343 | 324 | 104
score on a scale | 10.5 (26.86) | 11.7 (28.11) | 11.0 (28.85) | 14.5 (27.92) | 9.5 (27.36)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.054, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = 5.11, 95% CI 2-sided [-0.08 to 10.31], Standard Error of Mean 2.647
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.007, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = 7.10, 95% CI 2-sided [1.93 to 12.26], Standard Error of Mean 2.634
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.025, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = 5.90, 95% CI 2-sided [0.75 to 11.04], Standard Error of Mean 2.623
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = 8.38, 95% CI 2-sided [3.20 to 13.55], Standard Error of Mean 2.638

198. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Adequacy - Month 12 - (MITT)
Description: as for outcome 156
Time Frame: Baseline and Month 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 283 | 305 | 312 | 280 | 93
score on a scale | 9.8 (27.33) | 12.0 (29.86) | 12.6 (27.71) | 14.1 (28.81) | 10.0 (31.76)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.089, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = 5.02, 95% CI 2-sided [-0.76 to 10.80], Standard Error of Mean 2.945
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.010, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = 7.56, 95% CI 2-sided [1.83 to 13.29], Standard Error of Mean 2.920
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.009, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = 7.65, 95% CI 2-sided [1.94 to 13.36], Standard Error of Mean 2.911
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.007, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = 7.89, 95% CI 2-sided [2.11 to 13.67], Standard Error of Mean 2.944

199. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Somnolence - Week 12 - (MITT)
Description: as for outcome 157
Time Frame: Baseline and Week 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 354 | 365 | 374 | 376 | 117
score on a scale | -9.2 (20.49) | -8.1 (18.67) | -7.6 (19.57) | -8.9 (21.09) | -8.7 (20.54)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.349, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -1.64, 95% CI 2-sided [-5.07 to 1.79], Standard Error of Mean 1.749
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.499, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -1.18, 95% CI 2-sided [-4.60 to 2.24], Standard Error of Mean 1.743
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.936, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-3.27 to 3.55], Standard Error of Mean 1.737
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.696, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-4.08 to 2.72], Standard Error of Mean 1.736

200. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Somnolence - Month 6 - (MITT)
Description: as for outcome 158
Time Frame: Baseline and Month 6
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 317 | 333 | 343 | 324 | 104
score on a scale | -9.4 (22.40) | -8.4 (19.88) | -9.6 (20.04) | -8.7 (21.65) | -9.6 (21.64)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.572, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -1.09, 95% CI 2-sided [-4.86 to 2.69], Standard Error of Mean 1.924
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.553, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -1.14, 95% CI 2-sided [-4.89 to 2.62], Standard Error of Mean 1.914
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.456, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -1.42, 95% CI 2-sided [-5.16 to 2.32], Standard Error of Mean 1.907
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.949, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-3.89 to 3.64], Standard Error of Mean 1.919

201. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Somnolence - Month 12 - (MITT)
Description: as for outcome 159
Time Frame: Baseline and Month 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 283 | 305 | 312 | 280 | 93
score on a scale | -8.5 (22.79) | -9.2 (19.17) | -9.9 (19.33) | -9.4 (23.06) | -6.7 (25.95)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.097, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -3.36, 95% CI 2-sided [-7.34 to 0.61], Standard Error of Mean 2.026
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.008, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -5.34, 95% CI 2-sided [-9.28 to -1.40], Standard Error of Mean 2.010
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.014, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -4.94, 95% CI 2-sided [-8.87 to -1.01], Standard Error of Mean 2.003
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.056, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -3.88, 95% CI 2-sided [-7.86 to 0.10], Standard Error of Mean 2.029

202. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Problems Index I - Week 12 - (MITT)
Description: as for outcome 160
Time Frame: Baseline and Week 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 354 | 365 | 374 | 376 | 117
score on a scale | -13.5 (17.90) | -11.4 (18.02) | -12.2 (18.29) | -12.8 (19.33) | -9.8 (20.47)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.003, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -4.92, 95% CI 2-sided [-8.18 to -1.65], Standard Error of Mean 1.665
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.023, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -3.79, 95% CI 2-sided [-7.05 to -0.53], Standard Error of Mean 1.660
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.047, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -3.28, 95% CI 2-sided [-6.52 to -0.04], Standard Error of Mean 1.653
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.039, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -3.41, 95% CI 2-sided [-6.65 to -0.17], Standard Error of Mean 1.652

203. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Problems Index I - Month 6 - (MITT)
Description: as for outcome 161
Time Frame: Baseline and Month 6
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 317 | 333 | 343 | 324 | 104
score on a scale | -14.0 (17.60) | -12.9 (16.76) | -13.2 (19.16) | -13.8 (19.77) | -9.8 (20.37)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.69, 95% CI 2-sided [-9.05 to -2.33], Standard Error of Mean 1.713
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.58, 95% CI 2-sided [-8.93 to -2.24], Standard Error of Mean 1.704
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.003, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.12, 95% CI 2-sided [-8.45 to -1.79], Standard Error of Mean 1.697
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.003, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.11, 95% CI 2-sided [-8.46 to -1.76], Standard Error of Mean 1.708

204. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Problems Index I - Month 12 - (MITT)
Description: as for outcome 162
Time Frame: Baseline and Month 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 283 | 305 | 312 | 280 | 93
score on a scale | -12.8 (18.19) | -13.0 (18.36) | -13.7 (19.02) | -14.0 (20.14) | -9.1 (22.62)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -6.01, 95% CI 2-sided [-9.71 to -2.32], Standard Error of Mean 1.885
Statistical Analysis 2: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -7.22, 95% CI 2-sided [-10.89 to -3.55], Standard Error of Mean 1.871
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -6.92, 95% CI 2-sided [-10.58 to -3.27], Standard Error of Mean 1.863
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -6.42, 95% CI 2-sided [-10.12 to -2.72], Standard Error of Mean 1.886

205. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Problems Index II - Week 12 - (MITT)
Description: as for outcome 163
Time Frame: Baseline and Week 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 354 | 365 | 374 | 376 | 117
score on a scale | -15.1 (17.64) | -13.0 (17.38) | -13.9 (17.40) | -13.4 (18.47) | -11.8 (19.48)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.004, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -4.60, 95% CI 2-sided [-7.75 to -1.44], Standard Error of Mean 1.609
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.030, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = -3.49, 95% CI 2-sided [-6.64 to -0.34], Standard Error of Mean 1.605
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.049, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -3.15, 95% CI 2-sided [-6.29 to -0.02], Standard Error of Mean 1.598
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.121, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -2.48, 95% CI 2-sided [-5.61 to 0.65], Standard Error of Mean 1.597

206. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Sleep Problems Index II - Month 6 - (MITT)
Description: as for outcome 164
Time Frame: Baseline and Month 6
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 317 | 333 | 343 | 324 | 104
score on a scale | -15.5 (18.15) | -14.6 (16.41) | -14.9 (18.95) | -14.8 (18.87) | -11.6 (19.31)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.44, 95% CI 2-sided [-8.74 to -2.14], Standard Error of Mean 1.682
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.53, 95% CI 2-sided [-8.81 to -2.25], Standard Error of Mean 1.674
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -5.12, 95% CI 2-sided [-8.39 to -1.85], Standard Error of Mean 1.667
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.006, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = -4.64, 95% CI 2-sided [-7.93 to -1.35], Standard Error of Mean 1.677

207. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Individual Score for Sleep Problems Index II - Month 12 - (MITT)
Description: as for outcome 165
Time Frame: Baseline and Month 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 283 | 305 | 312 | 280 | 93
score on a scale | -14.3 (18.35) | -14.6 (17.95) | -15.4 (18.74) | -15.1 (19.43) | -10.5 (21.71)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -6.28, 95% CI 2-sided [-9.91 to -2.65], Standard Error of Mean 1.849
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -7.58, 95% CI 2-sided [-11.18 to -3.98], Standard Error of Mean 1.835
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -7.43, 95% CI 2-sided [-11.02 to -3.84], Standard Error of Mean 1.828
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -6.54, 95% CI 2-sided [-10.17 to -2.91], Standard Error of Mean 1.851

208. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Optimal Sleep - Week 12 - (MITT)
Description: Change from Baseline (BL) to Wk 12 in MOS Optimal Sleep Score as compared with Placebo.The MOS-Sleep Self Report Questionnaire is composed of 12 items measuring 6 dimensions of sleep over the past 4 wks. Optimal sleep is based on Q2 (self-reported average hrs sleep per night in past 4 wks). Scoring method: hrs of sleep coded 0 (non-optimal) or 1 (optimal) where 1-6 hrs & 9-23 hrs = 0, 7-8 hrs = 1. Change from BL: subject sleeps 7-8 hrs at BL & 1-6 or 9-23 hrs at follow-up, change = -1; subject sleeps 1-6 or 9-23 hrs at BL & 7-8 hrs at follow-up, change = +1; subject sleeps 1-6 or 9-23 hrs at BL & 1-6 or 9-23 hrs at follow-up, change = 0. Mean change from BL: changes are summed to give the Net Total (equivalent to the number subjects w/ improved sleep hrs minus the number subjects w/ worsened sleep hrs), which is divided by the number of subjects to give the mean proportion of net change, where >0 = overall improvement and <0 = overall worsening in the study arm.
Time Frame: Baseline and Week 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: Proportion of Net Change
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 353 | 364 | 372 | 376 | 116
Proportion of Net Change | 0.2 (0.53) | 0.1 (0.56) | 0.2 (0.49) | 0.1 (0.52) | 0.2 (0.59)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.225, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.04 to 0.16], Standard Error of Mean 0.049
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.741, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Week 12; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.08 to 0.11], Standard Error of Mean 0.049
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.414, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.06 to 0.14], Standard Error of Mean 0.049
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.690, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Week 12; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.11 to 0.08], Standard Error of Mean 0.049

209. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Optimal Sleep - Month 6 - (MITT)
Description: Change from Baseline (BL) to Month 6 in MOS Optimal Sleep Score as compared with Placebo.The MOS-Sleep Self Report Questionnaire is composed of 12 items measuring 6 dimensions of sleep over the past 4 wks. Optimal sleep is based on Q2 (self-reported average hrs sleep per night in past 4 wks). Scoring method: hrs of sleep coded 0 (non-optimal) or 1 (optimal) where 1-6 hrs & 9-23 hrs = 0, 7-8 hrs = 1. Change from BL: subject sleeps 7-8 hrs at BL & 1-6 or 9-23 hrs at follow-up, change = -1; subject sleeps 1-6 or 9-23 hrs at BL & 7-8 hrs at follow-up, change = +1; subject sleeps 1-6 or 9-23 hrs at BL & 1-6 or 9-23 hrs at follow-up, change = 0. Mean change from BL: changes are summed to give the Net Total (equivalent to the number subjects w/ improved sleep hrs minus the number subjects w/ worsened sleep hrs), which is divided by the number of subjects to give the mean proportion of net change, where >0 = overall improvement and <0 = overall worsening in the study arm.
Time Frame: Baseline and Month 6
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: Proportion of Net Change
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 316 | 331 | 339 | 323 | 104
Proportion of Net Change | 0.2 (0.56) | 0.2 (0.55) | 0.2 (0.53) | 0.1 (0.56) | 0.2 (0.52)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.045, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [0.00 to 0.21], Standard Error of Mean 0.052
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.069, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 6; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.01 to 0.20], Standard Error of Mean 0.052
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.126, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.02 to 0.18], Standard Error of Mean 0.052
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.907, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 6; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.10 to 0.11], Standard Error of Mean 0.052

210. Secondary Outcome: Medical Outcomes Sleep Study (MOS) Optimal Sleep - Month 12 - (MITT)
Description: Change from Baseline (BL) to Month 12 in MOS Optimal Sleep Score as compared with Placebo.The MOS-Sleep Self Report Questionnaire is composed of 12 items measuring 6 dimensions of sleep over the past 4 wks. Optimal sleep is based on Q2 (self-reported average hrs sleep per night in past 4 wks). Scoring method: hrs of sleep coded 0 (non-optimal) or 1 (optimal) where 1-6 hrs & 9-23 hrs = 0, 7-8 hrs = 1. Change from BL: subject sleeps 7-8 hrs at BL & 1-6 or 9-23 hrs at follow-up, change = -1; subject sleeps 1-6 or 9-23 hrs at BL & 7-8 hrs at follow-up, change = +1; subject sleeps 1-6 or 9-23 hrs at BL & 1-6 or 9-23 hrs at follow-up, change = 0. Mean change from BL: changes are summed to give the Net Total (equivalent to the number subjects w/ improved sleep hrs minus the number subjects w/ worsened sleep hrs), which is divided by the number of subjects to give the mean proportion of net change, where >0 = overall improvement and <0 = overall worsening in the study arm.
Time Frame: Baseline and Month 12
Population: All randomized subjects who took at least one dose (2 capsules) of IP.
Measure: Mean (Standard Deviation); unit: Proportion of Net Change
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
Number analyzed (Participants) | 282 | 303 | 311 | 280 | 93
Proportion of Net Change | 0.1 (0.51) | 0.2 (0.56) | 0.1 (0.55) | 0.1 (0.52) | 0.2 (0.47)
Statistical Analysis 1: Comparison: Combined Estradiol 1 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.992, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 1 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.11 to 0.11], Standard Error of Mean 0.055
Statistical Analysis 2: Comparison: Combined Estradiol 0.5 mg / Progesterone 100 mg vs Placebo; Test type: Superiority; p = 0.450, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 100 mg against Placebo at Month 12; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.07 to 0.15], Standard Error of Mean 0.054
Statistical Analysis 3: Comparison: Combined Estradiol 0.5 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.663, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.5 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.13 to 0.08], Standard Error of Mean 0.054
Statistical Analysis 4: Comparison: Combined Estradiol 0.25 mg / Progesterone 50 mg vs Placebo; Test type: Superiority; p = 0.309, Mixed Models Analysis — p-value is derived from comparison between Combined Estradiol 0.25 mg / Progesterone 50 mg against Placebo at Month 12; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.16 to 0.05], Standard Error of Mean 0.055

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected on or after the subject signed Informed Consent through fifteen days following the last dose of Investigational Product. Treatment Emergent Adverse Event data were collected on or after the first dose of IP through fifteen days following the last dose of IP.
Arm/Group | Combined Estradiol 1 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 100 mg | Combined Estradiol 0.5 mg / Progesterone 50 mg | Combined Estradiol 0.25 mg / Progesterone 50 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/415 | 0/424 | 1/421 | 0/424 | 0/151
Serious Adverse Events (participants affected / at risk) | 9/415 | 15/424 | 9/421 | 11/424 | 2/151
Other Adverse Events (participants affected / at risk) | 324/415 | 277/424 | 291/421 | 232/424 | 41/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Estradiol 1 mg / Progesterone 100 mg (N=415) | Combined Estradiol 0.5 mg / Progesterone 100 mg (N=424) | Combined Estradiol 0.5 mg / Progesterone 50 mg (N=421) | Combined Estradiol 0.25 mg / Progesterone 50 mg (N=424) | Placebo (N=151)
Cardiac Tamponade (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Stress Cardiomyopothy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Colitis Ischaemic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastroduodenal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Angioedema (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cholecystitis Infective (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Clostridium Difficile Colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infectious Mononucleosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Jaw Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Chondrocalcinosis Pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Breast Cancer Female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0 | 0
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Non-Small Cell Lung Cancer Stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Balance Disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cerebellar Infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Uterine Leiomyoma (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Uterine Prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Aortic Aneurysm (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Aortic Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Estradiol 1 mg / Progesterone 100 mg (N=415) | Combined Estradiol 0.5 mg / Progesterone 100 mg (N=424) | Combined Estradiol 0.5 mg / Progesterone 50 mg (N=421) | Combined Estradiol 0.25 mg / Progesterone 50 mg (N=424) | Placebo (N=151)
Headache (Nervous system disorders) | 31 | 24 | 45 | 43 | 4
Nasopharyngitis (Infections and infestations) | 25 | 41 | 37 | 24 | 4
Breast Tenderness (Reproductive system and breast disorders) | 45 | 19 | 25 | 10 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 22 | 26 | 34 | 15 | 6
Nausea (Gastrointestinal disorders) | 20 | 25 | 19 | 16 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 22 | 11 | 15 | 15 | 1
Abdominal Pain (Gastrointestinal disorders) | 22 | 10 | 14 | 15 | 4
Sinusitis (Infections and infestations) | 20 | 15 | 13 | 13 | 3
Dizziness (Nervous system disorders) | 17 | 15 | 10 | 8 | 3
Pelvic Pain (Reproductive system and breast disorders) | 17 | 15 | 10 | 7 | 0
Diarrhoea (Gastrointestinal disorders) | 13 | 13 | 11 | 11 | 2
Vulvovaginal Mycotic Infection (Infections and infestations) | 14 | 15 | 14 | 5 | 4
Abdominal Distension (Gastrointestinal disorders) | 15 | 6 | 11 | 11 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 16 | 13 | 7 | 7 | 1
Hypertension (Vascular disorders) | 7 | 13 | 9 | 12 | 2
Influenza (Infections and infestations) | 4 | 6 | 14 | 12 | 2
Vaginal Haemorrhage (Reproductive system and breast disorders) | 14 | 10 | 3 | 8 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days